# **Statistical Analysis Plan**

SAP Text Version Number: Final Version 1.0 SAP Text Date: 20-May-2022

Sponsor Name: Galderma S.A./Galderma R&D, LLC

Protocol Number: RD.06.SPR.203065

**Protocol Title:** A Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy and Safety of Nemolizumab (CD14152) in Subjects with Prurigo Nodularis

## **Protocol Version and Date:**

V1.0, 21-Feb-2020; V3.0, 25-Jun-2020; V4.0, 22-Dec-2020 V5.0, 19-Nov-2021

Syneos Health Project Code: 7009814

Author: , Biostatistician II

#### **Notice of Confidential and Proprietary Information:**

The information contained in this document is confidential belonging to Galderma S.A./Galderma R&D, LLC. Acceptance of this document constitutes agreement by the recipient that no information contained herein will be published or disclosed without prior written authorization from an official of Galderma S.A./Galderma R&D, LLC. However, this document may be disclosed to appropriate Institutional Review Board and Ethics Committees or duly authorized representatives of a national regulatory authority under the condition that they are requested to keep it confidential. In the event of an actual or suspected breach of this obligation, Syneos Health should be notified promptly.

# **Revision History**

| Version # | Date<br>(DD-Mmm-YYYY) | Document Owner | Revision Summary |
|---|---|---|---|
| Final<br>Version 1.0 | 20-May-2022 | | Final Version |

I confirm that I have reviewed this document and agree with the content.

| Approvals | | |
|---|---|---|
| Syneos | Health Approval | |
| | | May 20, 2022 |
| Name, Title Developing Biostatistician | Signature | Date (DD-Mmm-<br>YYYY) |
| | | May 20, 2022 |
| Name, Title | Signature | Date (DD-Mmm-<br>YYYY) |
| Senior Reviewing Biostatistician | | , |
| Galderma S.A./Ga | alderma R&D, LLC Approval | |
| | = | May 20, 2022 |
| Name, Title<br>Sponsor Contact | Signature | Date (DD-Mmm-<br>YYYY) |

# **Table of Contents**

| Rev | rision Hi | istory | 2 |
|-----|-----------|-------------------------------------|----|
| App | orovals | | 3 |
| 1. | Gloss | ary of Abbreviations | 8 |
| 2. | Purpo | ose | 12 |
| | 2.1. | Responsibilities | 12 |
| | 2.2. | Timings of Analyses | 12 |
| 3. | Study | Objectives | 13 |
| | 3.1. | Primary Objective | 13 |
| | 3.2. | Secondary Objectives | 13 |
| 4. | Study | Details/Design | 14 |
| | 4.1. | Brief Description | 14 |
| | 4.2. | Subject Selection | 16 |
| | | 4.2.1. Inclusion Criteria | 16 |
| | | 4.2.2. Exclusion Criteria | 16 |
| | 4.3. | Determination of Sample Size | 16 |
| | 4.4. | Treatment Assignment and Blinding | 17 |
| | 4.5. | Administration of Study Medication | 18 |
| | 4.6. | Study Procedures and Flowchart | 19 |
| 5. | Endpo | oints | 24 |
| | 5.1. | Primary Efficacy Endpoints | 24 |
| | 5.2. | Key Secondary Efficacy Endpoints | 24 |
| | 5.3. | Secondary Efficacy Endpoints | 24 |
| | 5.4. | Pharmacokinetic Endpoints | 25 |
| | 5.5. | Immunogenicity Endpoints | 25 |
| | 5.6. | Safety Endpoints | 25 |
| 6. | Analy | sis Sets | 26 |
| | 6.1. | Screened Population | 26 |
| | 6.2. | Intent-to-Treat Population | 26 |
| | 6.3. | Per-Protocol Population | 26 |
| | 6.4. | Safety Population | 26 |
| | 6.5. | Pharmacokinetic Analysis Population | 26 |

| | 6.6. | Protoco | ol Deviations | 26 |
|---|---|---|---|---|
| 7. | Estima | ands | | 28 |
| 8. | Gener | al Aspec | ts for Statistical Analysis | 31 |
| | 8.1. | Genera | l Methods | 31 |
| | 8.2. | Key De | finitions | 31 |
| | 8.3. | Missing | Data | 32 |
| | 8.4. | Visit Wi | indows | 33 |
| | 8.5. | Pooling | of Centers | 34 |
| | 8.6. | Subgro | ups | 35 |
| 9. | Demo | graphic, | Other Baseline Characteristics and Medication | 36 |
| | 9.1. | Subject | Disposition and Withdrawals | 36 |
| | 9.2. | Demog | raphic and Baseline Disease Characteristics | 36 |
| | 9.3. | Medical | l History | 37 |
| | 9.4. | Medical | I and Surgical Procedure | 37 |
| | 9.5. | Medicat | tion | 38 |
| | 9.6. | Extent of | of Exposure | 39 |
| | 9.7. | Treatme | ent Compliance | 39 |
| 10. | Effica | cy | | 40 |
| | 10.1. | Primary | / Efficacy Endpoints | 40 |
| | | 10.1.1. | Primary Analysis of Primary Efficacy Endpoint | 40 |
| | | 10.1.2. | Sensitivity Analyses of Primary Efficacy Endpoint | 41 |
| | | 10.1.3. | Subgroup Analyses of Primary Efficacy Endpoints | 41 |
| | 10.2. | Key Se | condary Efficacy Endpoints | 42 |
| | 10.3. | Second | lary Efficacy Endpoints | 42 |
| | | 10.3.1. | Investigator's Global Assessment (IGA) | 45 |
| | | 10.3.2. | Prurigo Activity Score (PAS) | 46 |
| | | 10.3.3. | Pruritus Numeric Rating Scale (NRS) | 46 |
| | | 10.3.4. | Sleep Disturbance Numeric Rating Scale (SD NRS) | 48 |
| | | 10.3.5. | Subject Sleep Diary | 49 |
| | | 10.3.6. | PN Associated Pain Intensity and Frequency | 50 |
| | | 10.3.7. | Patient Global Assessment of Disease (PGAD) | |
| | | 10.3.8. | Patient Global Assessment of Treatment (PGAT) | 51 |

| | | 10.3.9. | Dermatology Life Quality Index | 51 |
|---|---|---|---|---|
| | | 10.3.10. | Hospital Anxiety and Depression Scale (HADS) | 51 |
| | | 10.3.11. | EuroQoL 5 Dimension Instrument | 52 |
| | | 10.3.12. | Rescue Therapy Used | 52 |
| 11. | Pharm | nacokineti | ics | 53 |
| | 11.1. | Pharma | cokinetic Concentration Presentation | 53 |
| | 11.2. | Pharma | cokinetic and Pharmacodynamics Parameters Estimation | 53 |
| | 11.3. | Biomark | (ers | 53 |
| 12. | Immui | nogenicity | / | 54 |
| 13. | Safety | ′ | | 55 |
| | 13.1. | Adverse | e Events | 55 |
| | 13.2. | Laborate | ory Evaluations | 57 |
| | | 13.2.1. | Clinical Laboratory Evaluations | 57 |
| | | 13.2.2. | Pregnancy Testing | 59 |
| | | 13.2.3. | Virology and TB Testing | 59 |
| | 13.3. | Vital Sig | ıns | 59 |
| | 13.4. | ECG | | 60 |
| | 13.5. | Physical | I Examination | 60 |
| | 13.6. | Respirat | tory Assessments | 61 |
| | | 13.6.1. | Respiratory Examination | 61 |
| | | 13.6.2. | Peak Expiratory Flow | 61 |
| | | 13.6.3. | Asthma Control Test | 61 |
| 14. | Chang | ges from A | Analysis Planned in Protocol | 63 |
| 15. | Refere | ence List. | | 64 |
| 16. | Progra | amming C | Considerations | 65 |
| | 16.1. | General | Considerations | 65 |
| | 16.2. | Table, F | Figure, and Listing Format | 65 |
| | | 16.2.1. | General | 65 |
| | | 16.2.2. | Headers | 66 |
| | | 16.2.3. | Display Titles | 66 |
| | | 16.2.4. | Column Headers | 66 |
| | | 16.2.5. | Body of the Data Display | 66 |

| | | 16.2.6. | Footnotes | 68 |
|-----|---------|------------|---------------------------------------|----|
| 17. | Quality | y Control | | 70 |
| 18. | Index | of Tables | · | 71 |
| 19. | Index | of Figures | S | 87 |
| 20. | Index | of Listing | s | 89 |
| 21. | Appen | dices | | 91 |
| | 21.1. | Tipping | Point Analysis | 91 |
| | 21.2. | Multiple | Imputation | 91 |
| | | 21.2.1. | Imputation Phase | 91 |
| | | 21.2.2. | Analysis Phase | 91 |
| | | 21.2.3. | Pooling Phase | 91 |
| | 21.3. | Example | e SAS Code | 92 |
| | 21.4. | Potentia | ally Clinically Significant Ranges | 94 |

#### 1. **Glossary of Abbreviations**

| Abbreviation | Description |
|--------------|-----------------------------------|
| Α | Anxiety |
| ACT | Asthma Control Test |
| ADA | Anti-Drug Antibodies |
| ADaM | Analysis Dataset Model |
| AE | Adverse Event |
| AESI | Adverse Event of Special Interest |
| ALP | Alkaline Phosphatase |
| ALT | Alanine Aminotransferase |
| ANCOVA | Analysis of Covariance |
| AP | Average Pruritus |
| AST | Aspartate Aminotransferase |
| ATC | Anatomical Therapeutic Chemical |
| BDRM | Blind Data Review Meeting |
| BLQ | Below the Limit of Quantification |
| ВМІ | Body Mass Index |
| CHMP | Committee for Medicinal Products |
| CI | Confidence Interval |
| СМН | Cochran-Mantel-Haenszel |
| COVID-19 | Coronavirus Disease-19 |
| CRA | Clinical Research Associate |
| CRF | Case Report Form |
| CRO | Contract Research Organization |
| CS | Clinical Significant |
| CSR | Clinical Study Report |
| CTMS | Clinical Trial Management System |
| CV | Coefficient of Variation |
| D | Depression |
| DBL | Data Base Lock |
| DCS | Dual-Chamber Syringe |

| Abbreviation | Description |
|--------------|-------------------------------------------|
| DD | Drug Dictionary |
| DLQI | Dermatology Life Quality Index |
| ECG | Electrocardiogram |
| eCRF | Electronic Case Report Form |
| ePRO | Electronic Patient Reported Outcome |
| EQ-5D | EuroQoL 5-Dimension |
| ET | Early Termination |
| FSH | Follicle-Stimulating Hormone |
| HADS | Hospital Anxiety and Depression Scale |
| HBcAb | Hepatitis B core Antibody |
| HBsAg | Hepatitis B surface Antigen |
| HCV | Hepatitis C Virus |
| HDL | High-Density Lipoproteins |
| HIV | Human Immunodeficiency Virus |
| IAC | Independent Adjudication Committee |
| ICF | Informed Consent Form |
| ICH | International Conference on Harmonization |
| ID | Identifier |
| IDMC | Independent Data Monitoring Committee |
| IGA | Investigator Global Assessment |
| IL | Interleukin |
| IRT | Interactive Response Technology |
| ITT | Intent-to-Treat |
| IVRS | Interactive Voice Response System |
| IWRS | Interactive Web Response System |
| LDL | Low-Density Lipoproteins |
| LLN | Lower Limit of Normal |
| LLT | Lowest Level Term |
| LOCF | Last Observation Carried Forward |
| LTE | Long-Term Extension |
| LSMeans | Least Squares Means |

| Abbreviation | Description |
|--------------|-----------------------------------------------------------|
| MAR | Missing at Random |
| MCMC | Markov Chain Monte Carlo |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MI | Multiple Imputation |
| min | Minutes |
| MMRM | Mixed-Effect Models for Repeated Measures |
| MNAR | Missing Not at Random |
| MSD | Morning Sleep Diary |
| N/A | Not Applicable |
| NAb | Neutralizing Antibodies |
| NCS | Not Clinical Significant |
| NRS | Numeric Rating Scale |
| ос | Observed Case |
| PAS | Prurigo Activity Score |
| PD | Pharmacodynamics |
| PDF | Portable Document Format |
| PEF | Peak Expiratory Flow |
| PGx | Pharmacogenomic |
| PGAD | Patient Global Assessment of Disease |
| PGAT | Patient Global Assessment of Treatment |
| PGIC-P | Patient Global Impression of Change – Pruritus |
| PGIC-SD | Patient Global Impression of Change – Sleep Disturbance |
| PGIS-P | Patient Global Impression of Severity – Pruritus |
| PGIS-SD | Patient Global Impression of Severity – Sleep Disturbance |
| рН | Potential of Hydrogen |
| PK | Pharmacokinetic |
| PN | Prurigo Nodularis |
| PopPK | Population Pharmacokinetic |
| PP NRS | Peak Pruritus Numeric Rating Scale |
| PP | Per-Protocol |
| PPS | Per-Protocol Set |

| Abbreviation | Description |
|--------------|-------------------------------------------|
| PRO | Patient-Reported Outcome |
| PT | Preferred Term |
| Q1 | 1st Quartile |
| Q3 | 3d Quartile |
| Q4W | Every 4 Weeks |
| QC | Quality Control |
| QoL | Quality of Life |
| RNA | Ribonucleic Acid |
| RTSM | Randomization and Trial Supply Management |
| SAE | Serious Adverse Event |
| SAF | Safety Population |
| SAP | Statistical Analysis Plan |
| SAS | Statistical Analysis System |
| SC | Subcutaneous |
| SD | Standard Deviation |
| SD NRS | Sleep Disturbance Numeric Rating Scale |
| SDTM | Study Data Tabulation Model |
| SOC | System Organ Class |
| SOP | Standard Operating Procedure |
| ТВ | Tuberculosis |
| TEAE | Treatment-Emergent Adverse Event |
| TFL | Table, Figure and Listing |
| TMF | Trial Master File |
| ULN | Upper Limit of Normal |
| UPT | Urine Pregnancy Test |
| USA | United States of America |
| VAS | Visual Analogue Scale |
| W | Week |
| WASO | Wakefulness after Sleep Onset |
| WHO | World Health Organization |

# 2. Purpose

The purpose of this statistical analysis plan (SAP) is to ensure that the data listings, summary tables and figures which will be produced, and the statistical methodologies that will be used, are complete and appropriate to allow valid conclusions regarding the study objectives. The planned analyses identified in this SAP will be included in regulatory submissions and/or future manuscripts. Exploratory analyses not identified or defined in this SAP may be performed to support the clinical development program. Any post-hoc or unplanned analyses performed and not identified in this SAP will be documented in the respective clinical study report (CSR).

# 2.1. Responsibilities

Syneos Health will perform the statistical analyses and is responsible for the production and quality control of all tables, figures and listings.

Descriptive summary and listing will be provided for pharmacokinetic concentration. Definition of the Pharmacokinetic analysis population and derivation of Pharmacokinetic parameters will be performed by a designated CRO. This designated CRO will be responsible for the ad-hoc Modeling / Simulation Plan and the Modeling & Simulation Report. Any analysis of pharmacokinetic parameters will not be included in the CSR final TFLs but in the dedicated Modeling & Simulation Report. For further details see Section 11.

# 2.2. Timings of Analyses

A primary analysis will be carried out once all subjects have completed the final study visit or terminate early from the study. No personnel directly involved with the conduct of the study shall have access to the unblinded data before the completion of the trial in order to avoid introducing bias to the remaining study data.

The final analysis will be performed after all subjects completed the study.

An independent data monitoring committee (IDMC) will review and monitor subject safety throughout the study, and an independent adjudication committee (IAC) will review all asthma-related adverse events throughout the study. Details on the IDMC and IAC, including the plan of analysis for outputs; the composition of the committees; and the procedures, roles, responsibilities, and communications are provided in the respective IDMC (v2.0, dated 01-Nov-2021) and Appendix 2 of IAC charters (v2.0, dated 13-Jan-2022).

#### **Study Objectives** 3.

#### 3.1. **Primary Objective**

The primary objective is to assess the efficacy of Nemolizumab (CD14152) compared to placebo in subjects ≥ 18 years of age with prurigo nodularis (PN) after a 16-week treatment period.

#### 3.2. **Secondary Objectives**

The secondary objectives are to assess safety, pharmacokinetics, and immunogenicity of Nemolizumab (CD14152) compared to placebo.

# 4. Study Details/Design

## 4.1. Brief Description

This phase 3, multicenter, double-blind, placebo-controlled, randomized, parallel group study is designed to evaluate the efficacy and safety of Nemolizumab in subjects with PN.

Subjects' participation in the study will be up to 28 weeks. The study consists of a screening period (up to 4 weeks), a 16-week treatment period, and an 8-week follow up period (12 weeks after the last study drug injection). Refer to Figure 4-1 for an overview of study design.

Figure 4-1: Study Design



(R): Kandomization

🕽 : Nemolizumab 30 mg administration 😛 : Placebo administration

- \* Applicable for subjects who do not participate in the LTE study only
- \*\* Loading dose (two injections) administered at baseline visit for subjects weighing < 90 kg</p>
- \*\*\* Two injections administered at all applicable visits for subjects weighing ≥ 90 kg at the baseline visit

Abbreviations: BL = baseline; W = week.

Following provision of written informed consent, subjects with PN will be screened for enrolment in the study. Eligible subjects will return for a baseline visit where, following randomization, they will be administered either 60 mg of Nemolizumab or placebo via 2 SC injections. Thereafter, study drug will be administered Q4W at Weeks 4, 8, and 12 by a single SC injection of either Nemolizumab 30 mg or placebo

for subjects weighing < 90 kg at baseline or by two SC injections of either Nemolizumab 30 mg or placebo for subjects weighing ≥ 90 kg at baseline. Efficacy and safety assessments will be performed at visits throughout the screening and treatment period, as outlined in the Schedule of Assessments (Table 4-2).

At the end of the 16-week treatment period, consenting subjects may be eligible to enter an active treatment/long-term extension (LTE) study (RD.06.SPR.202699). Subjects who participate in the LTE are not required to complete the follow-up visit. Subjects who do not participate in the LTE will return for a follow-up visit at Week 24 (12 weeks after the last study drug injection).

Subjects who prematurely discontinue the study drug will be asked to continue participation in the study and return for all remaining visits and assessments (including daily assessment of pruritus and sleep disturbance). Subjects who discontinue study drug due to required rescue therapy may be eligible to participate in the LTE study following completion of study visits through Week 16. Subjects who discontinue the study prematurely should complete an early termination (ET) visit and a follow-up visit 12 weeks after the last study drug injection.

As no approved medicine for PN exists with which to compare Nemolizumab, a placebo-controlled design was implemented in this study to allow blinding, randomization, and identical administration procedures to control for human bias or other influences on the disease (e.g., natural disease course), while enabling demonstration of differences in clinical effect and safety profile of investigational treatment, if present. All subjects will have access to rescue medication to minimize risk and for ethical considerations. It is the position of the Committee for Medicinal Products for Human Use (CHMP) that, where ethical and feasible, a placebo control arm should be included in the pivotal trial(s) used to support marketing authorization application.

A 16-week treatment period is considered adequate to evaluate the efficacy and safety of Nemolizumab based on the results of the phase 2a study (RD.03.SPR.115828) in subjects with PN. All subjects who complete the treatment period (Week 16 visit) can be considered for LTE study eligibility. A 2-to-1 randomization is selected to minimize the number of subjects exposed to placebo for an extended period of time.

Although the pathophysiology of PN is still not fully understood, the efficacy endpoints selected for the phase 3 trial are relevant to the underlying manifestations associated with the disease under study (i.e., skin lesions, chronic itch, sleep disturbance, and quality of life impairment). The selected endpoints for assessing the safety and PK of Nemolizumab (CD14152) are in accordance with current standards. Blinding subjects and the designated study team to the treatment assignment(s) helps ensure objectivity and minimize bias. Randomization through the Interactive Response Technology (IRT) guards against selection bias.

The study includes an 8-week follow-up period (i.e., 12 weeks after the last study drug injection) for subjects who decline or are not eligible to enroll in the LTE study. The duration of the follow-up period from the final Nemolizumab dose (12 weeks) corresponds to approximately 5 half-lives of Nemolizumab, which is considered adequate to ensure subject safety. The follow-up visit is not required for subjects who participate in the LTE, where the primary objective is long-term evaluation of safety.

Differences may be detectable during the study drug reconstitution process between active study drug and placebo but appear similar after reconstitution is complete (approximately 10 minutes). Throughout the study, a pharmacist (or other qualified personnel) will prepare study drug for injection, including confirmation

of complete reconstitution, prior to delivery of study drug for injection. The pharmacist (or other qualified personnel) preparing study drug should not be involved with any study assessments and should not discuss any aspects of study drug reconstitution with the subject or study staff involved in subject interviews or study assessments.

The placebo-controlled design includes a provision for rescue therapy for pruritus, based on the investigator's clinical judgment. Subjects requiring rescue therapy may be eligible for the LTE study but will be required to continue scheduled study visits until the Week 16 visit before LTE eligibility will be assessed.

To avoid bias and to ensure the integrity of the blind, personnel directly involved with the ongoing conduct of the study from the Sponsor, blinded statistical team at Syneos Health, or other investigational study centers will not have access to any information that may lead to unblinding.

A subject will have fulfilled the requirements for study completion if/when the subject has completed all study periods, including Week 16 or the last scheduled visit as indicated in the Schedule of Assessments (Table 4-2).

The end of the study will be the last subject's last visit or the last subject's scheduled visit as indicated in the Schedule of Assessments (Table 4-2).

### 4.2. Subject Selection

Eligible subjects for this clinical study will be adults with a clinical diagnosis of PN for at least 6 months, manifested by pruriginous nodular lesions on the trunk and/or limbs, and at least 20 nodules on the entire body bilaterally distributed. The inclusion criterion for IGA is consistent with the disease severity targeted in the study: An IGA of 3 or 4 corresponds to moderate or severe PN, respectively. Severe pruritus will be defined by PP NRS scores  $\geq 7.0$  within the past 24 hours at screening and the mean PP NRS score  $\geq 7.0$  during the previous week at baseline. Subjects with chronic pruritus due to other active conditions or unilateral pruriginous lesions are ineligible. Further, subjects must undergo specific required washout periods from restricted topical and systemic treatments before enrolling in the study. The study population is selected based on the current unmet need in the management of PN, the mode of action of Nemolizumab (CD14152), and the need to understand the efficacy and safety of Nemolizumab (CD14152) in the adult population with PN.

#### 4.2.1. Inclusion Criteria

For a detailed description of subject's inclusion criteria see protocol Section 8.1.

#### 4.2.2. Exclusion Criteria

For a detailed description of subject's exclusion criteria see protocol Section 8.2.

#### 4.3. Determination of Sample Size

In order to achieve at least 90% power for both primary endpoints at 5% significance level, 270 (180 Nemolizumab, 90 placebo) subjects will be randomized to detect the following differences in both primary endpoints between treatment groups with 2:1 randomization, assuming a 15% dropout rate during treatment period.

NRS responders (≥ 4 point reduction from baseline): Based on phase 2a data, it is expected that the NRS response at Week 16 would be 50% in Nemolizumab and 20% in placebo.

IGA response (0/1): It is expected that the IGA response at Week 16 would be 30% in Nemolizumab and 10% in placebo.

Table 4-1 provides the resulting power with 270 subjects (180 Nemolizumab, 90 placebo) for different responses in primary endpoints.

Table 4-1: Results of Power Analysis

| Endpoint | Placebo | Nemolizumab | Power at 5% significance<br>level (N= 270 [180<br>Nemolizumab, 90 placebo]) |
|---|---|---|---|
| IGA responder | 10% | 30% | 90% |
| | 10% | 27% | 83% |
| | 10% | 25% | 77% |
| PP-NRS Responder | 20% | 50% | > 90% |
| | 20% | 45% | > 90% |
| | 20% | 40% | 84% |
| Assuming 15% attrition rate during treatment period. Based on continuity corrected Chi-square test. | | | |

# 4.4. Treatment Assignment and Blinding

Upon confirmation of eligibility for a given subject to participate in the study, a unique randomization number will be assigned to that subject via Interactive Response Technology (IRT).

The randomization number for a given subject will be used to identify the treatment arm the subject will be assigned to.

Subjects will be randomized in a 2:1 ratio to receive treatment of either Nemolizumab (CD14152) or placebo. The randomization scheme will be stratified by the study site and body weight at randomization (< 90 kg and ≥ 90 kg) using the IRT system.

All attempts will be made to keep the study center staff and subjects blinded throughout the study. Members of the study center staff, including those responsible for dual-chamber syringe (DCS) preparation, will not have access to the randomized treatment assignment.

To ensure double-blind administration of study drug, the study center pharmacist(s) or other qualified personnel will prepare all Nemolizumab (CD14152) or placebo treatments, according to the current version of the pharmacy manual and assigned DCS provided by the IRT system.

As there may be detectable differences between active and placebo during the reconstitution process, the DCS is delivered for injection after the reconstitution is complete. The pharmacist (or other qualified personnel) preparing study drug should not be involved with any study assessments and should not discuss any aspects of study drug reconstitution with the subject or study staff involved in subject interviews or study assessments.

To maintain the integrity of the study blinding, the bioanalytical laboratory staff who process/analyze the PK/anti-drug antibody (ADA)/pharmacodynamic (PD)/ pharmacogenomic (PGx) samples will not provide any information to the Sponsor, CRO, or investigational study center personnel directly involved with the ongoing conduct of the study that may lead to unblinding during the ongoing study. PK and ADA results will released by the bioanalytical laboratory after data base lock (DBL).

Unblinding of a subject's individual treatment code should occur only in case of a medical emergency or in the event of a serious medical condition that necessitates identification of the study drug for the welfare of that subject, as judged by the investigator. The emergency unblinding process utilizes IRT to allow the investigator to have unrestricted, immediate, and direct access to the subject's individual study treatment. When possible (i.e., when the health of the subject is not immediately at risk), the investigator or sub-investigator is encouraged to consult with the medical monitor and the Sponsor before breaking the blind.

If emergency unblinding is required:

- Only the investigator will make the decision to unblind the treatment assignment.
- Only the affected subject will be unblinded.
- The IRT system will provide the treatment assignment to the investigator.

Refer to the Randomization and Trial Supply Management (RTSM) User Guide for information on the steps for breaking the blind in the IRT system.

When the blinding code is broken, the reason must be fully documented. If the code is broken by the investigator, the subject must be withdrawn from the study and must also be appropriately followed for a minimum of 12 weeks after the last dose of study drug.

The reporting requirements for unblinding are the same for reporting an SAE. See also Section 12.7.4 of protocol.

The randomization code will remain blinded to all study sites and study team members until completion of the study and after the study database has been locked.

The IDMC will review data at periodic intervals throughout the study as defined in the IDMC charter. The IDMC charter will specify the procedures for unblinding to ensure treatment assignment remains undisclosed to all individuals involved in the direct execution and management of the study until the final database is locked.

# 4.5. Administration of Study Medication

All study drug injections will occur at the study center, following instructions provided in the instructions for use and the current version of the pharmacy manual. After confirming that the study drug is fully reconstituted, the pharmacist (or other qualified personnel) will deliver the DCS to the investigator or other qualified personnel, for SC injection in the subject's abdomen or an alternative injection site. A different injection site should be selected for each injection. Refer to the current version of the pharmacy manual and the instructions for use for further details. The site of injection should be recorded in the subject's treatment record as well as the eCRF at each time point.

For subjects willing and able to self-inject, study center staff will provide training on study drug injections. Subjects will be allowed to inject medication following appropriate training and under supervision by study center clinic staff (with DCS preparation including reconstitution performed by the pharmacist or other qualified personnel and delivered for injection after reconstitution is complete). Study center/clinic staff can perform all injections if the subject does not wish to perform injections. The eCRF will record who performed study drug injection at each visit.

Sponsor: Galderma S.A./Galderma R&D, LLC; Protocol No.: RD.06.SPR.203065

After study drug administration, subjects will be monitored closely for any signs or symptoms of hypersensitivity reaction before being discharged. For the first 2 visits where study drug is administered, subjects should remain at the study center for at least 30 minutes following study drug administration.

# 4.6. Study Procedures and Flowchart

See Table 4-2 for study procedures.

Table 4-2: Schedule of Assessments

| Study period | Screening<br>period<br>(Day -28 to<br>Day-1) | period Treatment period | | | | | | Follow-<br>up ° | Early<br>Termination | Unscheduled visit |
|---|---|---|---|---|---|---|---|---|---|---|
| Visit | V1 | V2 | No visit <sup>b</sup> | V3 | V4 | V5 | V6 | V7 | 4 | |
| Week | Screening <sup>a</sup> | Baseline | W1 | W4<br>Day 29 | W8<br>Day 57 | W12<br>Day 85 | W16<br>Day 113 | W24 | (if applicable) | (if applicable) |
| Day | | 2 | Day 8 | | | | | Day 169 | | |
| Visit window | D-28 to D-8 | Day 1 | ±0 days | ±2 days | ±2 days | ±5 days | ±5 days | ±7 days | 1 | |
| Informed consent form | X | | | | | | | | | |
| Photography, skin biopsy, and PGx consent form(s) (if applicable) | X | | | | | | | | | (X) |
| Inclusion/exclusion criteria | X | Х | | | | | | | | |
| Demographics | X | | | | | 2 | | | | i i |
| Medical history, previous therapies and procedures, smoking status | х | | | | | | | | | (X) |
| | | PAT | ENT-REPOR | TED OUTC | OME ASSE | SSMENTS | | | 200 | |
| PP NRS/AP NRS/SD NRS/<br>subject sleep diary <sup>e,f</sup> | х | ( | | | | Х | | | х | (X) |
| PGIS-P/PGIS-SD <sup>e,f</sup> | | X | ХÞ | | | 4 | X | | X | (X) |
| PGIC-P/PGIC-SD <sup>e,f</sup> | p. | | ХÞ | | | | X | | X | (X) |
| PGAD <sup>g</sup> | | Х | ХÞ | | | | X | | Х | (X) |
| PGAT 9 | | | | | | | Х | | X | (X) |
| PN-associated pain frequency and intensity <sup>g</sup> | | X | | X | X | х | х | | х | (X) |
| DLQI <sup>g</sup> | 6 | Х | | X | | 0% | X | | X | (X) |
| EQ-5D/HADS <sup>g</sup> | | X | | | | | X | | X | (X) |
| | | | CLINI | CAL PHOTO | OGRAPHS | 26 | | | -04- | |
| Full body clinical photographs (optional) | 3 | Х | | | | 2 | X | | х | (X) |
| | | | CLINICAL E | FFICACY | ASSESSME | NTS | | | | |
| IGA | X | Х | | Х | Х | Х | Х | | X | (X) |
| PAS | X | X | | X | X | Х | Х | | Х | (X) |

This document is confidential.

SAP Version: Final Version 1.0, 20-May-2022 Controlled Document ID: **3903A.02**, Effective Date 31-Aug-2020 Filing requirements: TMF

| Study period | Screening<br>period<br>(Day -28 to<br>Day-1) | | | Treatmen | t period | | | Follow-<br>up ° | Early<br>Termination | Unscheduled visit |
|---|---|---|---|---|---|---|---|---|---|---|
| Visit | V1 | V2 | No visit <sup>b</sup> | V3 | V4 | V5 | V6 | V7 | 4) | |
| Week | Screening <sup>a</sup> | Baseline | W1 | W4 | W8 | W12 | W16 | W24 | (if applicable) | (if applicable) |
| Day | D 004- D 0 | Down | Day 8 | Day 29 | Day 57 | Day 85 | Day 113 | Day 169 | | |
| Visit window | D-28 to D-8 | Day 1 | ±0 days | ±2 days | ±2 days | ±5 days | ±5 days | ±7 days | | |
| | | <i>ii</i> . | SAFI | ETY ASSES | SMENTS | | ž | | ************************************** | |
| ACT <sup>g, i</sup> | X | X | | X | X | X | X | X | X | (X) |
| Respiratory exam | X | X | | Х | Х | X | X | X | X | (X) |
| PEF testing <sup>j</sup> | X | X | | Χj | X | Χj | Х | X | X | (X) |
| Vital signs | Х | Х | | Х | X | Х | Х | X | X | (X) |
| Full physical examination | X | X | | | X | | Х | X | X | (X) |
| Height | X | | | | | . X | ×. | | 5%<br>5m | (X) |
| Weight | Х | Х | | | | | Х | | X | (X) |
| 12-lead ECG k | X | X | | | | 4 | X | | X | (X) |
| Contraceptive counseling | Χ | | | | | 03 | | | 176 | (X) |
| Adverse Events <sup>g</sup> | Х | Х | | Х | Х | Х | X | X | Х | (X) |
| Concomitant therapies and procedures <sup>a</sup> | X | Х | | X | X | X | Х | X | Х | (X) |
| | | | LABOR | ATORY AS | SESSMENT | S | | | | |
| Blood sample for virology (HIV,<br>Hepatitis B, and C test) | X | | | | | | | | | (X) |
| Blood samples for TB test <sup>1</sup> | Х | | | | | s. | | | 5 | (X) |
| Blood samples for hematology and biochemistry m.n | х | Х | ž | X | X | 25 | X | X | х | (X) |
| Urinalysis <sup>n</sup> | X | X | | | X | | X | X | X | (X) |
| Pregnancy test <sup>o</sup> | Serum | Urine | | Urine | Urine | Urine | Urine | Urine | Urine | (Urine) |
| FSHP | X | | 2 | | | 30 | | | n) | |
| | | | PK, ADA, PI | D AND PGX | ASSESSM | ENTS | | | | |
| Blood sample for PK d. n. q | | X | | X | X | X | X | X | X | (X) |
| Blood sample for ADA <sup>d, n</sup> | | Х | | | X | | X | | Х | (X) |
| Blood sample for PD <sup>r</sup> | | X | | | X | | X | | | (X) |

This document is confidential.

SAP Version: Final Version 1.0, 20-May-2022 Controlled Document ID: **3903A.02**, Effective Date 31-Aug-2020 Filing requirements: TMF

| Study period | Screening<br>period<br>(Day -28 to<br>Day-1) | | | Treatmen | t period | | | Follow-<br>up ° | Early<br>Termination | Unscheduled visit |
|---|---|---|---|---|---|---|---|---|---|---|
| Visit | V1 | V2 | No visit <sup>b</sup> | V3 | V4 | V5 | V6 | V7 | | |
| Week | Screening <sup>a</sup> | Baseline | W1 | W4 | W8 | W12 | W16 | W24 | (if applicable) | (if applicable) |
| Day | D-28 to D-8 | Day 1 | Day 8 | Day 29 | Day 57 | Day 85 | Day 113 | Day 169 | (ii applicable) | |
| Visit window | | Day 1 | ±0 days | ±2 days | ±2 days | ±5 days | ±5 days | ±7 days | | |
| Stratum corneum sample for PD r | | X | | | | C03 | X | | | (X) |
| Skin biopsy for PD (optional) <sup>r</sup> | | X | | | | | X | | | (X) |
| PGx sample (optional) <sup>s</sup> | | X | | | | 66 | | | | (X) |
| | | | STUDY | ORUG ADM | INISTRATIO | ON | | | | |
| Randomization | | X | | | | i i | | | D) | (X) |
| Study drug injection t. u. v. w | | X <sup>t</sup> | | X | X | X | | | | (X) |

Abbreviations: ACT, asthma control test; ADA, anti-drug antibodies; AP NRS, Average Pruritus Numeric Rating Scale; DLQI, Dermatology Life Quality Index; ECG, electrocardiogram; EQ-5D, EuroQoL 5-Dimension; FSH, follicle-stimulating hormone; HADS, Hospital Anxiety and Depression Scale; HIV, human immunodeficiency virus; IGA, Investigator Global Assessment; NRS, numeric rating scale; PAS, prurigo activity score; PD, pharmacodynamics; PEF, peak expiratory flow; PGAD, Patient Global Assessment of Disease; PGAT, Patient Global Assessment of Treatment; PGIC-P, Patient Global Impression of Change – Pruritus; PGIC-SD, Patient Global Impression of Severity – Pruritus; PGIS-SD, Patient Global Impression of Severity – Pruritus; PGIS-SD, Patient Global Impression of Severity – Sleep Disturbance; PGX, pharmacogenomic; PK, pharmacokinetic; PP NRS, Peak Pruritus Numeric Rating Scale; SD NRS, Sleep Disturbance Numeric Rating Scale; TB, tuberculosis; UPT, urine pregnancy test.

- Screening visit must be performed at least 7 days prior to Day 1 visit. Subjects deemed eliq ble will be provided with electronic handheld devices.
- b) Subjects will complete PGIS-P, PGIC-P, PGIS-SD, PGIC-SD, and PGAD assessments at Week 1 (i.e., 7 days after the Day 1/Baseline visit) for test-retest validation of itch and sleep PRO measures.
- c) The follow-up visit will be conducted for subjects who decline or are not eligible to enter the LTE study (including early termination) and should be conducted 12 weeks after the last study drug injection. (The follow-up visit is not required for subjects who will rollover to the LTE study.)
- d) Assessments to be conducted at the unscheduled visit depend on the reason for the visit. PK and ADA analyses are required only at unscheduled visits that are conducted for safety reasons. Subjects requiring rescue therapy between scheduled visits should return to the clinic for an unscheduled visit for investigator assessments of efficacy before starting rescue therapy. See Section 10.2.1 of protocol for details.
- e) SD NRS and sleep diary questions to be recorded by subjects once daily in the morning and if possible, within 1 hour of getting out of bed (Visit 1/Screening through Visit 6/Week 16). PP NRS and AP NRS to be recorded by subjects once daily in the evening (Visit 1/Screening through Visit 6/Week 16), beginning after the screening visit. On designated visits, PGIS-SD and PGIC-SD should be recorded after the SD NRS and sleep diary in the morning; PGIS-P and PGIC-P should be recorded after the PP NRS and AP NRS in the evening.
- f) Pruritus assessments scheduled for clinic visit days that are recorded by subjects in the evening (i.e., PP NRS, AP NRS, PGIS-P, PGIC-P) will be recorded the evening before the clinic visit.
- g) Patient-reported outcome assessments and designated safety measurements should occur before investigator assessments, laboratory sample collections, and study drug administration.
- Optional for consenting subjects and only for selected equipped sites; see Section 11.8 of protocol for details on clinical photographs.
- i) Subjects with a medical history of asthma will complete the ACT testing at each scheduled visit. Subjects with de novo asthma will complete the ACT testing beginning from de novo diagnosis and at all subsequent scheduled visits.
- j) PEF testing will be performed for all subjects at screening, baseline, Week 8, Week 16, and follow-up visits. For subjects reporting a medical history of asthma, PEF testing will be performed at all visits during the clinical study. For subjects diagnosed with de novo asthma. PEF testing will be performed at all visits, starting with the visit in which the

This document is confidential

SAP Version: Final Version 1.0, 20-May-2022

Controlled Document ID: 3903A.02, Effective Date 31-Aug-2020

diagnosis was confirmed. Subjects should be asked to withhold asthma medication on study visit days until after PEF testing is complete, to the extent it does not pose an undue risk to the subject. See Section 12.6.3 of protocol for details.

- k) 12-lead ECGs should be performed in the supine position, before any scheduled vital sign measurements and blood draws. See Section 12.4 of protocol.
- I) In case of indeterminate result for TB test, the test should be repeated (only 1 retest is allowed). If the test is still indeterminate, the subject must not be included in the study, unless subject has a documented history of completion of an appropriate TB treatment regimen with no history of re-exposure to TB since their treatment was completed.
- m) Subjects should be well hydrated and fast for at least 8 hours before the visit(s) when blood chemistry testing is planned, except for the screening visit.
- n) At scheduled visits with laboratory, PK, and ADA assessments, samples are to be collected before study drug injection(s).
- o) Only for females of childbearing potential. Serum pregnancy test to be performed at screening visit and UPT for all other visits. If UPT is positive, it must be confirmed with a serum pregnancy test. See Section 12.5.4 of protocol for details.
- p) For postmenopausal subjects (i.e., no menses for 12 consecutive months), confirm status with a high FSH level in the postmenopausal range.
- q) As a guideline, PK samples should be collected at approximately the same time of day throughout the study, to the extent possible, before study drug injection (pre-dose samples). See Section 13.1 of protocol for details on PK assessments.
- r) Blood, stratum coreum, and biopsy samples for PD assessments are only collected at selected sites. Biopsy samples are optional and only for subjects who provide additional consent. See Section 14.3 of protocol for details.
- s) Optional PGx sample collection is only for subjects who provide additional consent. See Section 14.1 of protocol for details.
- t) Subjects weighing < 90 kg at baseline will receive a loading dose on Day 1 (i.e., 2 injections of Nemolizumab 30 mg or placebo) then single injections of either 30 mg Nemolizumab or placebo Q4W. Subjects weighing ≥ 90 kg at baseline will receive either 60 mg Nemolizumab or placebo via 2 injections Q4W at all study visits.
- u) Study drug reconstitution will be performed by the pharmacist (or other qualified personnel) throughout the study, and complete reconstitution confirmed, prior to delivery for injection. Study center staff will provide study drug injection training for subjects willing and able to self-inject study drug. Based on the subject's preference, study center staff can also perform all injections.
- v) After study drug administration, subjects will be monitored closely for any signs or symptoms of hypersensitivity reaction before being discharged. For the first 2 visits where study drug is administered, subjects should remain at the study center for at least 30 minutes following study drug administration.
- w) If a study visit occurs outside the visit window, study drug injection(s) can still be administered provided there is a minimum of 3 weeks but not more than 5 weeks since the last injection. If beyond 5 weeks, the next study drug injection should then occur at the next planned visit. Future visits should be scheduled as soon as possible and within the required windows based on the baseline/Day 1 visit date, while maintaining the minimum 3-week interval between 2 injections.

# 5. Endpoints

# 5.1. Primary Efficacy Endpoints

- Proportion of subjects with an improvement of ≥ 4 from baseline in PP NRS at Week 16
- Proportion of subjects with an IGA success (defined as an IGA of 0 [Clear] or 1 [Almost clear] and a ≥ 2-point improvement from baseline) at Week 16

# 5.2. Key Secondary Efficacy Endpoints

The key secondary efficacy endpoints are as follows:

- Proportion of subjects with an improvement of ≥ 4 from baseline in PP NRS at Week 4
- Proportion of subjects with PP NRS < 2 at Week 16</li>
- Proportion of subjects with an improvement of ≥ 4 from baseline in SD NRS at Week 16
- Proportion of subjects with an improvement of ≥ 4 from baseline in SD NRS at Week 4
- Proportion of subjects with PP NRS < 2 at Week 4</li>

# 5.3. Secondary Efficacy Endpoints

The secondary efficacy endpoints are as follows:

- IGA success rate at each visit through Week 16
- Percentage of pruriginous lesions with excoriations/crusts (Prurigo Activity Score [PAS] item 5a) at each visit through Week 16
- Percentage of healed prurigo lesions (PAS item 5b) at each visit through Week 16
- Change from baseline in number of lesions in representative area (PAS item 4) at each visit through Week 16
- Proportion of subjects with an improvement of ≥ 4 from baseline in PP NRS through Week 16
- Proportion of subjects with PP NRS < 2 from baseline through Week 16
- Proportion of subjects with PP NRS < 3 from baseline through Week 16</li>
- Absolute change from baseline in PP NRS through Week 16
- Percent change from baseline in PP NRS through Week 16
- Proportion of subjects with an improvement of ≥ 4 from baseline in Average Pruritus (AP) NRS through Week 16
- Proportion of subjects with PP NRS improvement ≥ 4 from baseline and IGA success at Week 16
- Proportion of subjects with AP NRS < 2 from baseline through Week 16</li>
- Absolute change from baseline in AP NRS through Week 16
- Percent change from baseline in AP NRS through Week 16
- Proportion of subjects with an improvement of ≥ 4 from baseline in SD NRS through Week 16

This document is confidential.

- Absolute change from baseline in SD NRS through Week 16
- Percent change from baseline in SD NRS through Week 16
- Change from baseline in sleep diary endpoints (sleep onset latency, wakefulness after sleep onset [WASO], total awake time, total sleep time, sleep efficiency) based on recordings from subject sleep diary through Week 16
- Change from baseline in PN-associated pain frequency through Week 16
- Change from baseline in PN-associated pain intensity through Week 16
- Proportion of subjects reporting low disease activity (clear, almost clear, or mild) based on Patient Global Assessment of Disease (PGAD) at Week 16
- Proportion of subjects satisfied with study treatment (good, very good, or excellent) based on Patient Global Assessment of Treatment (PGAT) at Week 16
- Proportion of subjects with an improvement of ≥ 4 in Dermatology Life Quality Index (DLQI) through Week 16
- Change from baseline in DLQI through Week 16
- Change from baseline in Hospital Anxiety and Depression Scale (HADS) for each subscale (i.e., depression and anxiety) at Week 16
- Change from baseline in EuroQoL 5-Dimension (EQ-5D) at Week 16

# 5.4. Pharmacokinetic Endpoints

• Nemolizumab (CD14152) serum concentrations

# 5.5. Immunogenicity Endpoints

ADA assay (screening, confirmatory, titer, NAb)

# 5.6. Safety Endpoints

- Incidence and severity of AEs, including TEAEs, AESIs, SAEs and Adjudicated AEs
- Clinical laboratory tests
- Vital signs
- Electrocardiogram
- Physical examination
- Respiratory assessment including respiratory examination, Peak expiratory flow, and Asthma Control Test (ACT)

# 6. Analysis Sets

## 6.1. Screened Population

The Screened population comprises all subjects who signed the ICF and have screening data entered into the database. This population includes screen failures and randomized subjects. Screen failed subjects are defined as those subjects who fail to meet inclusion criteria or meet exclusion criteria and discontinue the study prior to randomization. Subjects that are re-screened will only be counted once, under the subject ID assigned for the repeat screening.

Unless specified otherwise, this set will be used for subject listings and summaries of subject disposition.

# 6.2. Intent-to-Treat Population

The Intent-to-Treat (ITT) population will consist of all randomized subjects. The ITT population will be the primary population for efficacy analyses. All analyses under the ITT population will be analyzed under the treatment group as randomized.

#### 6.3. Per-Protocol Population

The Per-Protocol (PP) population will consist of all subjects in the ITT population and have no major protocol deviations that would have a significant effect on the efficacy of the study treatment (see Section 6.6). Only primary and key secondary endpoints will be analyzed using the PP population, under the treatment group as randomized.

#### 6.4. Safety Population

The Safety (SAF) population will consist of all randomized subjects who received at least 1 administration of study drug. The treatment group assignment in this population will be defined by the treatment actually received. This population will be used for the analyses of safety.

#### 6.5. Pharmacokinetic Analysis Population

The PK analysis population will consist of all subjects included in the SAF, with at least one measurable post-baseline PK assessment. Similar to SAF, the treatment group assignment in this population will be defined by the treatment actually received. This population will be used for the descriptive analyses of PK concentrations.

#### 6.6. Protocol Deviations

Protocol deviations will be recorded by the Clinical Research Associate (CRA) in the Clinical Trial Management System (CTMS). All protocol deviations will be categorized by the associated deviation type and will be assessed individually on a regular basis on whether they are major or minor. Details can be found in the Protocol Deviation and Non-compliance Management Plan.

Major protocol deviations that are analysis relevant lead to an exclusion of the subject from the per-protocol population. A case by case decision regarding exclusions of subjects from the per-protocol analysis will be made in a blind data review meeting (BDRM) which will take place prior to unblinding the study. The criteria for exclusion from the PP population will be specified in the BDRM Preparation Plan. Only major protocol deviation which have a significant effect on the primary efficacy will result in exclusion from the PP population.

A summary table for number and percentage of subjects with major protocol deviation will be generated by type of deviation and treatment group for the ITT population.


Protocol deviations incurred as a direct result of the COVID-19 pandemic should be specifically recorded and presented as a COVID-19 deviation. The number and percentage of subjects with major (including major COVID-19) deviation will be provided by type of deviation and treatment group for the ITT population and additionally provided by Site.

All protocol deviations and the protocol deviations related to COVID-19 will be listed for the ITT population.

# 7. Estimands

The primary and key secondary efficacy endpoints will be evaluated and assigned to treatment at the time of randomization based on ITT population. The estimand is defined to address the scientific question relevant to subjects who are able to complete treatment with a response assessment without further medication being required, other than the allowed rescue medication.

An intercurrent event is an event which occurs after start of treatment and thus complicates the description and interpretation of treatment effects. Table 7-1 below lists potential intercurrent events and the strategy to deal with them for the estimand. The estimands for endpoints are defined in Table 7-2 and Table 7-3.

Table 7-1: List of Intercurrent Events

| Intercurrent Event | Strategy to Deal With<br>Intercurrent Event Within<br>Analysis | Assessment of Subject |
|---|---|---|
| Treatment discontinuation | Treatment-policy strategy | Use observed response; Non-<br>responder if missing. |
| Rescue therapy | Composite strategy | Consider the subjects who take rescue therapy as non-responder. |

Table 7-2: Estimands for Co-primary Endpoints (2 endpoints)

| Endpoints | Estimands |
|---|---|
| Proportion of subjects | Population: ITT population |
| with an improvement of<br>≥ 4 from baseline in PP<br>NRS at Week 16 | Endpoint: a binary response indicates if subjects have a change from Baseline of ≥ 4 at Week 16 |
| | Intercurrent events: use of rescue therapies on or prior to Week 16 is considered as non-responder; the observed response at Week 16 after treatment discontinuation will be used in the analysis. Missing Week 16 response after treatment discontinuation is treated as non-responder |
| | Summary measure: treatment difference of Nemolizumab and placebo in response rate |
| Proportion of subjects | Population: ITT population |
| with an IGA success<br>(defined as an IGA of 0<br>[Clear] or 1 [Almost | Endpoint: a binary response indicates if subjects have IGA of 0 [clear] or 1 [almost clear] and a ≥ 2-point reduction from Baseline at Week 16 |
| clear] and a ≥ 2-point improvement from baseline) at Week 16 | Intercurrent events: use of rescue therapies on or prior to Week 16 is considered as non-responder; the observed response at Week 16 after treatment discontinuation will be used in the analysis. Missing Week 16 response after treatment discontinuation is treated as non-responder |

| Endpoints | Estimands |
|---|---|
| | Summary measure: treatment difference of Nemolizumab and placebo in response rate |

Table 7-3: Estimands for Key Secondary Endpoints (5 endpoints)

| Endpoints | Estimands |
|---|---|
| Proportion of subjects with an improvement of | Population: ITT population |
| ≥ 4 from baseline in PP<br>NRS at Week 4 | <b>Endpoint:</b> a binary response indicates if subjects with an improvement of PP NRS ≥ 4 at Week 4 |
| | Intercurrent events: use of rescue therapies on or prior to Week 4 is considered as non-responder; the observed response at Week 4 after treatment discontinuation will be used in the analysis. Missing Week 4 response after treatment discontinuation is treated as non-responder |
| | Summary measure: treatment difference of Nemolizumab and placebo in response rate |
| Proportion of subjects | Population: ITT population |
| with PP NRS < 2 at<br>Week 16 | Endpoint: a binary response indicates if subjects with PP NRS < 2 at Week 16 |
| | Intercurrent events: use of rescue therapies on or prior to Week 16 is considered as non-responder; the observed response at Week 16 after treatment discontinuation will be used in the analysis. Missing Week 16 response after treatment discontinuation is treated as non-responder |
| | Summary measure: treatment difference of Nemolizumab and placebo in response rate |
| Proportion of subjects | Population: ITT population |
| with an improvement of<br>≥ 4 from baseline in SD<br>NRS at Week 16 | Endpoint: a binary response indicates if subjects with an improvement of SD NRS ≥ 4 at Week 16 |
| | Intercurrent events: use of rescue therapies on or prior to Week 16 is considered as non-responder; the observed response at Week 16 after treatment discontinuation will be used in the analysis. Missing Week 16 response after treatment discontinuation is treated as non-responder |
| | Summary measure: treatment difference of Nemolizumab and placebo in response rate |
| Proportion of subjects | Population: ITT population |
| with an improvement of | Endpoint: a binary response indicates if subjects with an improvement of SD NRS ≥ 4 at Week 4 |

| Endpoints | Estimands |
|---|---|
| ≥ 4 from baseline in SD<br>NRS at Week 4 | Intercurrent events: use of rescue therapies on or prior to Week 4 is considered as non-responder; the observed response at Week 4 after treatment discontinuation will be used in the analysis. Missing Week 4 response after treatment discontinuation is treated as non-responder |
| | Summary measure: treatment difference of Nemolizumab and placebo in response rate |
| Proportion of subjects<br>with PP NRS < 2 at<br>Week 4 | Population: ITT population Endpoint: a binary response indicates if subjects with PP NRS < 2 at |
| | Week 4 |
| | Intercurrent events: use of rescue therapies on or prior to Week 4 is considered as non-responder; the observed response at Week 4 after treatment discontinuation will be used in the analysis. Missing Week 4 response after treatment discontinuation is treated as non-responder |
| | Summary measure: treatment difference of Nemolizumab and placebo in response rate |

# 8. General Aspects for Statistical Analysis

#### 8.1. General Methods

- All data will be listed, and summary tables will be provided.
- Unless otherwise specified, summaries will be presented for each treatment and overall, if indicated, by visit.
- Continuous variables will be summarized using the number of observations (n), mean, standard deviation (SD), median, 1<sup>st</sup> Quartile (Q1), 3<sup>rd</sup> Quartile (Q3), minimum, and maximum. Categorical variables will be summarized using number of observations (n), frequency and percentages of subjects
- Unless otherwise stated, all statistical tests will be two-sided and conducted at the 5% level; all presented confidence intervals (CIs) will be two-sided 95% CIs.

### 8.2. Key Definitions

**Screening period** is a period of up to 4 weeks before Baseline/Day 1 during which subject eligibility is evaluated. Subjects receiving rescue therapies during the screening period are not eligible to participate in the study.

The 16-week **treatment period** is defined as Baseline/Day 1 to Week 16. If early discontinued during treatment period, it is defined as the period until 4 weeks (<=28 days) after last dosing date or early termination date whichever is earlier.

**Follow-up period** is defined as the post end of treatment period to follow-up visit in respective treatment period.

The **Baseline value** is defined as the last non-missing value before the first dose of study drug. In case that the date of first injection is not available, the date of randomization is considered.

For diary data (PP NRS, SD NRS), the Baseline values will be derived from data collected during the 7 days prior to the first administration of study drug, if subject is treated. Otherwise, the data collected during 7 days prior to randomization will be used. Baseline score will be the weekly prorated average of non-missing subject diary scores reported during the 7 days. A minimum of 4 daily scores out of the 7 days is required to calculate the weekly prorated average score. If there are less than 4 non-missing assessments in the baseline diary window, the interval lower bound can be extended up to 7 additional days, one day at a time, to obtain the most recent 4 non-missing values. For sensitivity analysis, a minimum of 2 or 3 daily scores out of the 7 days will be used to calculate the weekly prorated average score for primary and key secondary endpoints and the interval will not be extended with additional days.

The date of first treatment is defined as the date of first injection of study drug.

The date of last treatment is defined as the date of last injection of study drug.

**Study day** is defined as the number of days from the date of first treatment (randomization date if not treated) and will be calculated as follows:

• If the event date ≥ date of first treatment, then study day = event date - date of first treatment + 1.

Treatment Day 1 is therefore defined as the day of first treatment.

- If the event date < date of first treatment, then study day = event date date of first treatment.
- If subject is randomized, but not treated, then study day = event date date of randomization.

A subject's **date of last participation** in the trial is the last date of contact and is recorded as the date of completion or date of withdrawal on the completion page of the case report form (CRF).

Only the **subjects infected by COVID-19** during study participation will be considered subjects with COVID-19 infection.

#### 8.3. Missing Data

The primary method to impute the missing values will be as follows:

**Continuous Endpoints:** For continuous secondary endpoints (except EQ-5D, HADS) during treatment period, the MI under MAR assumption approach and the MMRM approach will be used to handle the missing data.

**Binary Endpoints:** All missing values will be treated as a non-responder for the binary endpoints for primary, key secondary and secondary endpoints. To assess the robustness of non-responder analysis for primary and key secondary endpoints, a tipping point analysis will be performed. The MI under MAR assumption, last observation carried forward (LOCF) approach, and observed case (OC) approach will be used as sensitivity analysis to impute the missing values for the primary and key secondary endpoints. If applicable, the continuous response will be imputed first, and the response will then be categorized.

**Use of rescue therapy:** All efficacy data, except OC, will be treated as treatment failure and considered as non-responder on or after rescue therapy is used. In OC analysis, no observed data after subject has received rescue treatment will be excluded. There will be no imputations for missing data.

Adverse events and concomitant medications/procedures: Missing assessment times will have imputed times for the purposes of assessing treatment emergence for AEs or classifying medications/procedures into prior/concomitant. However, the assessment date and time (start date, stop date, and time if collected from CRF) without imputation will be presented in the listings.

For the start of a concomitant medication/procedure or AE:

- Only the year is reported: If the subject received the first study drug dose in the year reported, then
  the date of the first dose of study drug will be used as the start date; otherwise, January 1 of the
  year reported will be used as the start date.
- The month and year are reported: If the subject received the first study drug in the month and year reported, then the date of the first dose of study drug will be used as the start date; otherwise, the first day of the month and year will be used as the start date.
- The time is collected but missing: If the start date is the same as the date the subject started
  receiving study drug, then the time of the first dose of study drug will be used as the start time;
  otherwise, 00:00 will be used as the start time.

For the end of a concomitant medication/procedure or AE:

- Only the year is reported: The earlier between December 31 of the year reported and the date of the last study contact with the subject will be used as the stop date.
- The month and year are reported: The earlier between the last date of the month and year reported and the date of the final contact with the subject will be used as the stop date.
- The time is collected but missing: 23:59 (or 23:59:59 if collected up to seconds) will be used as the stop time.

If an AE has the start date completely missing and the stop date on/after the first dose date of study drug, this AE will be considered as treatment emergent (TEAE).

If a medication/procedure has the stop date completely missing, this medication/procedure will be considered as ongoing and concomitant. If the start date of a medication/procedure is completely missing and impossible to identify different by stop date, this medication will be considered as concomitant.

## 8.4. Visit Windows

Efficacy by-visit summaries will use the analysis visit. Unscheduled and early termination visits will be windowed based on the analysis visit window in Table 8-1 which is based on study day. If multiple measurements are taken within the same window, the one taken closest to the target study day will be used for the analysis. If there are multiple measurements with same difference from target day, the later assessment should be used for the analysis.

Table 8-1: Analysis Visit Window

| Analysis Visit | Target Study<br>Day | Visit Window for<br>IGA, PAS, PN<br>associated Pain<br>frequency and<br>intensity | Visit Window for<br>PGIS-P, PGIS-SD,<br>PGIC-P, PGIC-SD,<br>PGAD, PGAT, EQ-<br>5D, HADS | Visit Window for DLQI |
|---|---|---|---|---|
| Baseline | 1 | ≤1 | ≤1 | <=1 |
| Week 1 | 8 | NA | 2 to 60 | NA |
| Week 4 | 29 | 2 to 42 | NA | 2 to 60 |
| Week 8 | 57 | 43 to 70 | NA | NA |
| Week 12 | 85 | 71 to 98 | NA | NA |
| Week 16 | 113 | 99 to 154 | 61 to 154 | 61 to 154 |
| Week 24 Follow-<br>up | 169 | 155 to 182 | NA | NA |

All daily diary efficacy data will be classified into analysis visits as described in Table 8-2 considering the data during the 7 days immediately preceding the target day of analysis visit.

Analysis visit of diary (ePRO) data will be defined depending on the data collection as below.

Diary data assessed within the extended timeframe below will be considered for analysis. The following rule will be applayed for post-treatment assessments only.

- Evening assessment (PP/AP NRS) recorded from 17:00:00 to 00:59:59
- Morning assessment (SD NRS, morning sleep diary) recorded from 5:00:00 to 17:59:59

#### Consecutive daily assessment:

For the evening assessments (PP NRS, AP NRS), the daily data collected up to Week 16 will be classified into analysis visits considering the data during the 7 days immediately preceding the target study day of analysis visit. Similarly, for the morning assessment (SD NRS, morning sleep diary), the 7 days data up to the target study day will be classified into analysis visit. Details of the analysis visit window are in Table 8-2 below.

Table 8-2: Analysis Visit Window for Evening and Morning Assessments

| Analysis Visit | Target Study Day | Visit Window for evening | Visit Window for morning |
|---|---|---|---|
| | of Analysis Visit | assessment (PP NRS, AP | assessment (SD NRS, |
| | | NRS) | morning sleep diary) |
| Baseline <sup>a</sup> | 1 | -7 to -1 | -6 to 1 before dosing |
| Week 1 | 8 | 1 to 7 | 2 to 8 |
| Week 2 | 15 | 8 to 14 | 9 to 15 |
| Week 3 | 22 | 15 to 21 | 16 to 22 |
| Week 4 | 29 | 22 to 28 | 23 to 29 |
| Week 5 | 36 | 29 to 35 | 30 to 36 |
| Week 6 | 43 | 36 to 42 | 37 to 43 |
| Week 7 | 50 | 43 to 49 | 44 to 50 |
| Week 8 | 57 | 50 to 56 | 51 to 57 |
| Week 9 | 64 | 57 to 63 | 58 to 64 |
| Week 10 | 71 | 64 to 70 | 65 to 71 |
| Week 11 | 78 | 71 to 77 | 72 to 78 |
| Week 12 | 85 | 78 to 84 | 79 to 85 |
| Week 13 | 92 | 85 to 91 | 86 to 92 |
| Week 14 | 99 | 92 to 98 | 93 to 99 |
| Week 15 | 106 | 99 to 105 | 100 to 106 |
| Week 16 <sup>b</sup> | 113 | 106 to 112 | 107 to 113 |

<sup>&</sup>lt;sup>a</sup> If there are less than 4 non-missing assessments within last 7 days prior to the first dose, the interval lower bound will be extended up to 7 additional days, one day at a time, to obtain the most recent 4 non-missing values. The extention will not be applied for the sensitivity analysis by using a minimum of 2 (or 3) daily scores out of the 7 days.

Safety and pharmacokinetics data will not be windowed for by-visit summary. i.e., scheduled visit data will be used for analysis.

### 8.5. Pooling of Centers

A small center is defined as a center with less than 12 randomized subjects. Small centers will be pooled prior to analyses.

First, centers will be sorted by country, number of randomized subjects (descending order) and center number (ascending order). Pooling will start with combining the largest of the set of small centers with the

<sup>&</sup>lt;sup>b</sup> If there are less than 4 assessments during Week 16 visit window, upper bound of the visit window (106 - 112) or (107 - 113) will be extended for 5 additional days. If there are still less than 4 assessments after extending upper bound of the visit window, lower bound of the visit window will be extended for another 5 days until 4 assessments are reached.

smallest center within that country. If there is a further need to combine data (the size of the pooled centers includes less than 12 subjects), the next smallest center will be combined with the next largest of the small centers, until the criterion of a minimum of 12 subjects is met.

The process will continue until all pooled centers have a minimum of 12 subjects within the country. Any remaining centers will be pooled with the last pooled center within the country. The pooled centers will be referred to 'analysis centers' in the statistical analyses.

## 8.6. Subgroups

Descriptive summary and analysis for primary and key secondary endpoints will be produced for the following subgroups:

- Region (Europe, North America, Asia Pacific)
- Age groups (18-65, and > 65)
- Sex (Male, Female)
- Race (White, Black or African American, Asian, American Indian or Alaska Native, Native Hawaiian or Pacific Islander, Other (including Multiple))
- Weight at randomization (< 90 kg, ≥ 90 kg)</li>
- Baseline IGA score (Moderate [3], Severe [4]).

# 9. Demographic, Other Baseline Characteristics and Medication

#### 9.1. Subject Disposition and Withdrawals

All subjects of the Screened population will be accounted for in this study.

Subject accounting will summarize subjects screened, re-screened, screen failed, randomized and randomized but not treated for all subjects by overall, country and site.

Subject accounting by visit will be summarized by treatment group and overall at each visit (scheduled visits only).

Subject disposition will be summarized based on the ITT population by treatment and overall. Summaries will include subjects randomized, subjects randomized but not treated, subjects treated, subjects completed treatment, subjects discontinued treatment, primary reason for discontinuation of treatment (including summary of subjects who stopped treatment due to COVID-19), subjects completed the study, subjects discontinued from the study, primary reason for discontinuation from the study (including summary of subjects who discontinued due to COVID-19), subjects rolled over to long term extension (LTE), and subjects completed Follow-up. Subjects who stopped treatment or discontinued study due to COVID-19 will be identified using other specify field in CRF.

Subject disposition will also be summarized by site on the ITT population.

Screen failure will be summarized for all screened subjects. Number of subjects screened and failed will be presented. Number and percentage of reason for screen failure (including summary of subjects who failed due to COVID-19) will be summarized.

Subjects in each analysis population (ITT, SAF, PP, PK analysis population) will be summarized by treatment group on the ITT population.

In addition, time (days since the first dose of study drug) to permanent discontinuation of study drug by reason for discontinuation will be displayed graphically in subjects having permanently discontinued from the study drug.

Randomization, study completion, drug completion, visit dates will be listed for the ITT population. Screen failure reason will also be listed. Additional listing of missed assessment for subjects who discontinued due to COVID-19 will be presented for the ITT population.

Analysis populations will be summarized and listed on the ITT population.

All inclusion and exclusion criteria not met will be listed on the Screened population.

#### 9.2. Demographic and Baseline Disease Characteristics

Summary statistics for demographic and other Baseline disease characteristics will be presented for the ITT, SAF, PP and PK analysis population.

Age (years), height (cm), weight (kg), and BMI (kg/m²) will be summarized using summary statistics for continuous variables. Age groups (18-65, and > 65), sex, region (Europe, North America, and Asia Pacific),
race, ethnicity, and smoking status will be summarized using the summary statistics for categorical variables. Weight will additionally be presented for each subgroup < 90 kg and ≥ 90 kg.

The Baseline disease characteristics IGA, weekly average PP NRS, weekly average AP NRS, weekly average SD NRS, pain frequency and intensity, PAS item 4 (number of lesion in representative area), item 5a (excoriation/crusts), item 5b (healed lesion stages), and baseline DLQI will be summarized. IGA, pain frequency, PAS item 5a and 5b will be summarized as a categorical variable.

A summary table for the stratification factor weight at randomization will be provided to show any discrepancies between what was reported through Interactive Voice Response System (IVRS)/Interactive Web Response System (IWRS) versus eCRF data (at baseline visit).

All demographic and baseline disease characteristics data will be listed on the ITT population.

### 9.3. Medical History

Medical history will be collected only at screening and will be coded using Medical Dictionary for Regulatory Activities (MedDRA), Version 25.0.

Medical history will be summarized by treatment group. The summary will include number and percentage of subjects reporting each system organ class (SOC), preferred term (PT) and lowest level term (LLT) and will be sorted alphabetically by SOC and descending frequency of PT within SOC and descending frequency of LLT within PT in the Nemolizumab treatment group. Summary tables will be presented for the ITT population.

Medical history data listings will be presented by subject number for the ITT population.

## 9.4. Medical and Surgical Procedure

Medical and surgical procedures will be coded using MedDRA, Version 25.0.

Prior medical and surgical procedures are defined as those which have been stopped before first treatment.

- Procedure before informed consent signed is defined as those stopped before the date of informed consent signed to the study.
- Procedure during screening period is defined as those stopped on or after the date of informed consent signed until before first treatment date.

Concomitant medical and surgical procedures will be defined as those started or stopped on or after the first treatment, or were ongoing during the study. If a procedure is started before the first treatment but is ongoing or stopped on or after the first treatment, it will be considered concomitant.

- Procedures during treatment period will be defined from start of treatment till 4 weeks (<= 28 days)</li>
   after the last treatment or early discontinuation date whichever is earlier.
- Procedures during follow-up period is defined from post treatment period (4 weeks (> 28 days) after the last treatment or early discontinuation date, whichever is earlier) to follow-up visit date.

If the stop date and 'ongoing' are missing then the procedure will be considered concomitant.

The following medical and surgical procedures (prior, concomitant and rescue procedures) will be summarized by treatment group using the number and percent of subjects reporting each SOC and PT and sorted alphabetically by SOC and descending frequency of PT within SOC in the Nemolizumab treatment group. Summary tables will be presented for the ITT population.

- Prior procedure before screening (before informed consent date)
- Prior procedure before first dosing (from screening [informed consent date] before the first treatment)
- Concomitant procedure during treatment period
- Concomitant procedure during follow-up period
- Rescue procedure during treatment period
- Rescue procedure during follow-up period

Medical and surgical procedures listings and rescue procedure listing will be presented by treatment group on the ITT population and sorted by subject number, start date, stop date, SOC, and PT.

#### 9.5. Medication

Medications will be classified and summarized on the ITT population as follows:

Prior medications are defined as those which stop before the first injection of study drug during the study.

- Prior medication before informed consent signed is defined as those stopped before the date of informed consent signed to the study.
- Prior medication during screening period is defined as those stopped during screening period (on or after the informed consent date, until before the first treatment date).

Concomitant medications are defined as those started, stopped, or ongoing on or after the first injection of study drug.

- *Medication during treatment period* is defined from start of treatment till 4 weeks (<= 28 days) after the last treatment or early discontinuation date whichever is earlier.
- *Medication during follow-up period* is defined from post treatment period (4 weeks (> 28 days) after the last treatment or early discontinuation date, whichever is earlier) to follow-up visit date

If the stop date and 'ongoing' are missing then the medication will be considered as concomitant medication.

Medications (prior, concomitant and rescue medications) will be coded using Version Global B3, March 2022 of the World Health Organization's Drug Dictionary (WHO DD). Preferred Anatomical Therapeutic Chemical (ATC) coding will be performed.

The following summaries by ATC level 2, ATC level 4 and preferred term (PT) will be produced on the ITT population. Subjects with more than one medication in a given ATC level and preferred name will be counted only once in that category. It will be sorted ATC level alphabetically and descending frequency in PT within ATC level term.

• Prior medication before screening (before informed consent date)


 Prior medication before first dosing (from screening [informed consent date] before the first treatment)

Concomitant medication during treatment period

Concomitant medication during follow-up period

Rescue medication during treatment period

Rescue medication during follow-up period

All medications (prior and concomitant medications, rescue medications) will be listed for the ITT population.

### 9.6. Extent of Exposure

Following parameters will be summarized:

 Treatment duration (in days) is calculated as follows, where date of first treatment is defined as the first day: [(date of last treatment – date of first treatment) + 1].

• Total dose administered (mg) will be calculated as the sum of all doses of study drug administered.

 Total dose planned (mg) will be calculated as the sum of all doses of study drug planned (dispensed) according to the treatment schedule of the treatment group.

The number of subjects who missed at least one dose

• The number of subjects who missed at least one dose due to COVID-19

The number of doses missed

The number of doses missed due to COVID-19

Treatment Compliance as described in Section 9.7.

Note: The missed dose due to COVID-19 are captured as other-reason reported in CRF.

#### 9.7. Treatment Compliance

Treatment compliance will be assessed through the treatment records and drug dispensation logs. As study drug is administered in the clinic, treatment compliance will be overseen and documented by the investigator and study staff (using the treatment records and drug accountability records).

Treatment compliance (%) is calculated as the total number of actual injections / the total number of expected injections \* 100. The total number of actual injections is counted based on collected study drug administration data. The total number of expected injections is counted based on the dosage schedule and dispensed as per protocol.

Filing requirements: TMF

# 10. Efficacy

Unless otherwise stated, all efficacy analyses will be performed on the ITT population.

All efficacy variables will be summarized by treatment group at each analysis visit. The primary comparison of interest is Nemolizumab compared to placebo.

To control the type I error at 5%, a fixed sequential testing approach will be implemented. For testing purposes, both primary endpoints will be tested first in a predefined order as listed in Section 5.1 at 5% significance level, and testing of key secondary endpoints will start only if both primary endpoints are successful at 5% level of significance. Key secondary endpoints will be tested in an order listed in Section 5.2, stopping when non-significant result (p > 0.05) is found.

## 10.1. Primary Efficacy Endpoints

10.1.1. Primary Analysis of Primary Efficacy Endpoint

The primary endpoints include the following endpoints:

- The proportion of subjects with an improvement of ≥ 4 from baseline in PP NRS at Week 16.
- The proportion of subjects reporting success on the IGA at Week 16, defined as an IGA response
  of 0 [Clear] or 1 [Almost clear] and a ≥ 2-point reduction from baseline;

For both primary endpoints, any subjects with missing data at Week 16 will be considered as a non-responder for the respective endpoint. If a subject is in receipt of rescue medication at any point on or prior to Week 16, data on or after receipt of rescue medication will be regarded as a non-responder.

The statistical hypotheses associated with the primary analysis of improvement in PP NRS ≥ 4 from baseline at Week 16 using treatment difference is, similarly:

Null hypothesis H0:  $P_{PP NRS\_nemolizumab} - P_{PP NRS\_placebo} = 0;$  Alternative hypothesis H1:  $P_{PP NRS\_nemolizumab} - P_{PP NRS\_placebo} \neq 0,$ 

where  $P_{PP\ NRS\_nemolizumab}$  and  $P_{PP\ NRS\_placebo}$  are the proportion of subjects categorized as having a PP NRS improvement from baseline to Week 16 of  $\geq$  4, for Nemolizumab and placebo, respectively.

The statistical hypotheses associated with the primary analysis of IGA success at Week 16 using treatment difference is:

Null hypothesis H0:  $P_{IGA\_nemolizumab} - P_{IGA\_placebo} = 0;$ Alternative hypothesis H1:  $P_{IGA\_nemolizumab} - P_{IGA\_placebo} \neq 0,$ 

where P<sub>IGA\_nemolizumab</sub> and P<sub>IGA\_placebo</sub> are the proportion of subjects categorized as success under IGA at Week 16 for Nemolizumab and Placebo, respectively.

Both primary endpoints will be analyzed using a Cochran-Mantel-Haenszel (CMH) test adjusted for the randomization strata analysis center and body weight at randomization (< 90 kg,  $\geq$  90 kg), in order to test the difference between Nemolizumab and placebo for the proportion of subjects achieving success in each endpoint. The estimate of the treatment difference and corresponding two-sided 95% CI and p-values will be presented. The confidence intervals will be based on Wald statistic controlling for stratification variables. Strata-adjusted proportion differences will be obtained using weighted average of stratum-specific proportion using CMH.

In addition an unadjusted CMH test will be performed.

Bar charts for the proportions of subjects with an improvement of ≥ 4 from baseline in PP NRS and IGA success at Week 16 will be presented.

## 10.1.2. Sensitivity Analyses of Primary Efficacy Endpoint

Sensitivity analyses for both primary endpoints will be conducted in order to test for the robustness of the primary analyses. The following sensitivity analyses will be conducted:

- Same analysis on PP population (including the bar charts for the proportion of subjects with an improvement of ≥ 4 from baseline in PP NRS and IGA success at Week 16).
- Tipping point analysis: To assess the robustness of non-responder analysis, a tipping point analysis will be performed by converting non-responders due to missing data to responders in successive increments (Δ) for both treatment groups. The value of Δ that overturns (i.e., non-significant) the primary results will represent the tipping point (see Appendix 21.1). A graphic display of all possible combinations of the number of responders among both treatment groups will be presented.
- Multiple Imputation (MI) method for missing data (or where rescue medication is received), assuming all missing data are Missing at Random (MAR) (see Appendix 21.2).
- Pattern-mixture model under assumption Missing Not at Random (MNAR) controlled-based pattern
  imputation. MI-based imputation will be applied as described above. Under MNAR assumption, a
  controlled based pattern imputation where only observation in placebo treatment group will be used
  to impute.
- Last Observation Carried Forward (LOCF) imputation method for missing data (or where rescue
  medication is received). Missing post-baseline values will be carried forward from the last non-missing
  post-baseline value. Baseline value will not be carried forward to post-baseline value.
- Observed Case (OC) no data will be imputed. For this analysis, if any rescue medication is received, data on or post rescue therapy will be analyzed as observed (i.e., not treated as non-responders).
- Removal of COVID-19 affected visits (i.e. exclusion of subjects from visit, if visit was missed due to COVID-19).
- 'Actual stratum' instead of 'stratum at the randomization' for subjects stratified incorrectly.
- Using at least 2 assessments for calculation of weekly average PP NRS instead of 4.
- Using at least 3 assessments for calculation of weekly average PP NRS instead of 4.

Tipping point analysis, multiple imputation methods, LOCF and OC analysis, analysis without COVID-19 affected visits and analysis with actual stratum will be performed on the ITT population. Except for OC analyses, assessments on or after rescue therapy used will be considered as non-responders.

# 10.1.3. Subgroup Analyses of Primary Efficacy Endpoints

In addition, the same analyses as described in Section 10.1.1 will be performed for the following subgroups:

- Region (Europe, North America, Asia-Pacific)
- Age groups (18-65, and > 65)
- Sex (Male, Female)
- Race (White, Black or African American, Asian, American Indian or Alaska Native, Native Hawaiian or Pacific Islander, Other (including Multiple))
- Weight at randomization (< 90 kg, ≥ 90 kg)</li>
- Baseline IGA Score (Moderate (3), Severe (4))

The subgroup analyses will be performed on the ITT population. Forest plot will be presented along with subgroup analysis results.

# 10.2. Key Secondary Efficacy Endpoints

The following key secondary endpoints are to be analyzed, in order:

- Proportion of subjects with an improvement of ≥ 4 from baseline to Week 4 in PP NRS;
- 2. Proportion of subjects with PP NRS < 2 at Week 16
- 3. Proportion of subjects with an improvement of ≥ 4 from baseline in SD NRS at Week 16
- 4. Proportion of subjects with an improvement of ≥ 4 from baseline in SD NRS at Week 4
- 5. Proportion of subjects with PP NRS < 2 at Week 4

All key secondary endpoints will be analyzed on the ITT population as primary endpoints (Section 10.1.1) including graphical presentation.

Additionally, the same sensitivity analyses as for the primary endpoints will be performed (Section 10.1.2), including bar charts for the key secondary endpoints or PP population.

Analysis of key secondary endpoints will be produced for the subgroups, too (Section 10.1.3).

# 10.3. Secondary Efficacy Endpoints

The following secondary endpoints are to be analyzed at the scheduled visits (Table 10-1):

Filing requirements: TMF

Table 10-1: Secondary Efficacy Endpoints

| Endpoint | Analysis Visit | Analysis to be done on which Population | Statistical Tests |
|---|---|---|---|
| IGA success rate at each visit | Baseline, W4, W8, W12,<br>W16 | On the ITT and PP population | СМН |
| Percentage of pruriginous lesions with excoriations/crusts (PAS items 5a) at each visit | Baseline, W4, W8, W12,<br>W16 | On the ITT and PP population | СМН |
| Percentage of healed lesion stages (PAS items 5b) at each visit | Baseline, W4, W8, W12,<br>W16 | On the ITT and PP population | СМН |
| Change from baseline in PAS item 4 (number of lesions in representative area) at each visit | Baseline, W4, W8, W12,<br>W16 | On the ITT and PP population | ANCOVA |
| Proportion of subjects with PP NRS at each visit: a) Improvement ≥ 4 from baseline; b) < 2 at visit c) < 3 at visit | Baseline, W4, W8, W12,<br>W16 | On the ITT and PP<br>Population | СМН |
| Absolute and Percent change from baseline in PP NRS at each visit | Baseline, W4, W8, W12,<br>W16 | On the ITT and PP<br>Population | ANCOVA |
| Proportion of subjects with PP NRS improvement ≥ 4 from baseline and IGA success | Baseline, W16 | On the ITT and PP<br>Population | CMH |
| Proportion of subjects with AP NRS at each visit: a) Improvement ≥ 4 in change from baseline; b) < 2 at visit | Baseline, W4, W8, W12,<br>W16 | On the ITT Population | СМН |
| Absolute and Percent change from baseline in AP NRS at each visit | Baseline, W4, W8, W12,<br>W16 | On the ITT Population | ANCOVA |
| Proportion of subjects with change from baseline improvement ≥ 4 in SD NRS at each visit | Baseline, W4, W8, W12,<br>W16 | On the ITT Population | СМН |
| Absolute and Percent change from baseline in SD NRS at each visit | Baseline, W4, W8, W12,<br>W16 | On the ITT Population | ANCOVA |

| Endpoint | Analysis Visit | Analysis to be done on which Population | Statistical Tests |
|---|---|---|---|
| Change from baseline in sleep diary<br>endpoints at each visit (sleep onset latency,<br>WASO, total awake time, total sleep time,<br>sleep efficiency) | Baseline, W4, W8, W12,<br>W16 | On the ITT Population | No hypothesis testing |
| Change from baseline in PN-Associated Pain Frequency and Intensity at each visit | Baseline, W4, W8, W12,<br>W16 | On the ITT Population | СМН |
| Proportion of subjects reporting low disease activity (clear, almost clear, mild) based on Patient Global Assessment of Disease (PGAD) at each visit | Baseline, W16 | On the ITT Population | СМН |
| Proportion of subjects satisfied with study treatment (good, very good, excellent) based on Patient Global Assessment of Treatment (PGAT) at each visit | W16 | On the ITT Population | СМН |
| Proportion of subjects with an improvement of ≥ 4 in DLQI at each visit | Baseline, W4, W16 | On the ITT Population | СМН |
| Change from baseline in DLQI at each visit | Baseline, W4, W16 | On the ITT Population | ANCOVA |
| Change from baseline in HADS for each subscale at each visit | Baseline, W16 | On the ITT Population | ANCOVA |
| Change from baseline in EQ-5D for each subscale at each visit | Baseline, W16 | On the ITT Population | ANCOVA |

Abbreviations: AP=Average Pruritus; DLQI=Dermatology Life Quality Index; EQ-5D=EuroQoL 5-Dimension; HADS=Hospital Anxiety and Depression Scale; IGA=Investigator Global Assessment; NRS=Numeric Rating Scale; PAS=Prurigo Activity Score; PGAD=Patient Global Assessment of Disease; PGAT=Patient Global Assessment of Treatment; PP=Peak Pruritus; SD=Sleep Disturbance; W=Week.

Binary secondary endpoints will be analyzed as described in Section 10.1.1. if not specified otherwise. Missing values will be imputed as non-responder except for OC analysis. If a subject is in receipt of rescue medication at any point, data on or after receipt of rescue medication will be regarded as a non-responder.

Continuous secondary endpoints (except EQ-5D, HADS) will be analyzed using multiple-imputation (MI) assuming MAR and using mixed effect model for repeated measure (MMRM) approach, including analysis center and body weight at randomization cut-off (< 90 kg and  $\geq$  90 kg) as factor and baseline as covariate where applies. The estimated treatment difference for each endpoint at each visit will be displayed in the summary of statistical analysis together with the 95% CI and associated p-value. EQ-5D and HADS endpoints will be analyzed using ANCOVA including analysis center and body weight at randomization cut-off (< 90 kg and  $\geq$  90 kg) as factor and baseline as covariate. All secondary endpoints will be presented descriptively using OC.

#### 10.3.1. Investigator's Global Assessment (IGA)

The IGA is a 5-point scale ranging from 0 (clear) to 4 (severe) used by the investigator or trained designee to evaluate the global severity of PN and the clinical response to a treatment (see Table 10-2).

Table 10-2: Investigator Global Assessment Scale

| 0 | Clear | No nodules |
|---|--------------|---------------------------------------|
| 1 | Almost Clear | Rare palpable pruriginous nodules |
| 2 | Mild | Few palpable pruriginous nodules |
| 3 | Moderate | Many palpable pruriginous nodules |
| 4 | Severe | Abundant palpable pruriginous nodules |

IGA treatment success is defined as 0 (clear) or 1 (almost clear) on the IGA scale and a  $\geq$  2-point reduction from Baseline.

IGA will be collected at Baseline/Day 1, Week 4, Week 8, Week 12, Week 16 and Early Termination. In case of missing assessment at Baseline, the last available assessment prior study drug administration will be considered as Baseline.

IGA will be summarized as a categorical and continuous variable at each analysis visit. Absolute change from Baseline for the IGA score will also be presented in the summary on the ITT and PP population.

The proportion of subjects with IGA success (OC, non-responder, LOCF) will be summarized on the ITT and PP Population. It will also be analyzed using non-responder imputation and a Cochran-Mantel-Haenszel (CMH) test adjusted for the randomization strata analysis center and body weight at randomization (< 90 kg,  $\geq$  90 kg). The estimate of treatment unadjusted and strata-adjusted differences with the corresponding two-sided 95% confidence intervals, and p-values from the CMH test will be presented.

Line plots for proportion of subject with IGA success using non-responder imputation will be generated for the ITT and PP population.

## 10.3.2. Prurigo Activity Score (PAS)

The Investigator or designee will use the PAS as an evaluation of the disease. This includes a count of the number of lesions in a representative area and a calculated staging (stage 0 to stage 4) based on the percentage of lesions with excoriations/crusts and healed lesions compared to all lesions.

Following items will be summarized at Baseline, Week 4, Week 8, Week 12, Week 16:

- PAS item 1a/1b: Type of prurigo
- PAS item 2: Number of pruriginous lesions
- PAS item 3: Affected area(s)
- PAS item 4: Number of lesions in representative area.
- PAS item 5a: Pruriginous lesions with excoriations/crusts
- PAS item 5b: Healed prurigo lesions

PAS items will be summarized as a categorical or continuous variable at each analysis visit, respectively. Absolute change from Baseline for continuous parameter PAS item 4 will also be presented in the summary on the ITT and PP population.

The proportion of subjects with pruriginous lesions with excoriation/crusts (PAS item 5a = 76-100%) and of subjects with healed lesion stages (PAS item 5b = 0-25%) will be presented using non-responder approach. The estimate of treatment unadjusted and strata-adjusted proportion differences with the corresponding two-sided 95% CI, and p-values from the CMH test will be presented.

Absolute and percentage change from Baseline in PAS item 4 will be analyzed using ANCOVA with MI assuming MAR approach, including analysis center and body weight at randomization cut-off (< 90 kg and ≥ 90 kg) as factor and baseline as covariate. The least squares means (LSMeans), standard error of LSMeans, and 95% CI for change from baseline, as well as the difference in LSMeans between the treatment groups, the two-sided 95% CI, and associated p-value will be presented for ITT and PP population.

# 10.3.3. Pruritus Numeric Rating Scale (NRS)

The Pruritus NRS is a scale to be used by the subjects to report the intensity of their pruritus (itch) during the last 24 hours. Peak pruritus (PP NRS) is an assessment of the maximum itch intensity in that period while average pruritus (AP NRS) provides a measure of overall pruritus intensity.

Subjects will be asked the following question:

- For maximum itch intensity (PP NRS): "On a scale of 0 to 10, with 0 being 'no itch' and 10 being the 'worst itch imaginable', how would you rate your itch at the worst moment during the previous 24 hours?"
- For average itch intensity (AP NRS): "On a scale of 0 to 10, with 0 being 'no itch' and 10 being the 'worst itch imaginable', how would you rate your itch overall during the previous 24 hours?"

The screening PP/AP NRS will be determined by a single assessment using the PP/AP NRS (score ranging from 0 to 10) for the 24-hour period immediately preceding the screening visit.


The Baseline PP/AP NRS will be determined based on the average of daily PP/AP NRS (score ranging from 0 to 10) respectively during the 7 days immediately preceding Baseline (rounding to nearest whole number is not permitted). A minimum of 4 daily scores out of the 7 days immediately preceding Baseline (up to one day before date of first treatment) is required for this calculation. If there are less than 4 non-missing assessments in the baseline diary window, the interval lower bound can be extended up to 7 additional days, one day at a time, to obtain the most recent 4 non-missing values.

PP/AP NRS at all follow-up visits will be determined in the same manner. Subjects will receive instructions on how to record their PP/AP NRS scores and will complete the assessment once daily in the evening throughout the clinical study (including the run-in and the follow-up period).

PP NRS will be determined by an average as described above at every week from Baseline to Week 16 as a continuous variable.

Descriptive summary of PP NRS will be provided on the ITT and PP populations using observed cases. Absolute change and percentage change from Baseline for the PP NRS will also be included in the summary on the ITT and PP populations.

AP NRS will be determined by an average as described above at every week from Baseline to Week 16 as a continuous variable. Descriptive summary of AP NRS will be provided on the ITT population. Absolute change and percent change from Baseline for the AP NRS score will also be included in the summary.

Absolute and percentage change from Baseline in PP/AP NRS will be analyzed using ANCOVA with MI assuming MAR and using MMRM approach, including analysis center and body weight at randomization cut-off (< 90 kg and ≥ 90 kg) as factor and baseline as covariate on ITT population. The least squares means (LSMeans), standard error of LSMeans, and 95% CI for change from baseline, as well as the difference in LSMeans between the treatment groups, the two-sided 95% CI, and associated p-value will be presented.

Proportion of subjects with PP NRS at each analysis visit will be summarized:

- Improvement ≥ 4 from baseline
- < 2 at visit</li>
- < 3 at visit</li>

Proportion of subjects with AP NRS at each visit will be summarized:

- Improvement ≥ 4 in change from baseline
- < 2 at visit</li>

The proportions of subjects will be presented on the ITT population using OC and non-responder for AP NRS and using OC, non-responder and LOCF for PP NRS. The estimate of treatment unadjusted and strata-adjusted proportion differences with the corresponding two-sided 95% CI, and p-values from the CMH test will be presented using non-responder.

Line plots for proportion of subjects with PP NRS improvement ≥ 4 and proportion of subjects with PP NRS < 2 using non-responder imputation will be presented on the ITT and PP population.

Additionally the weekly average PP NRS will be recalculated by using at least 2 assessments, or 3 assessments, instead of at least 4 assessments and without extending the visit window for sensitivity analysis.

The proportion of subjects with the weekly average PP NRS using 2, or 3 assessments, will be summarized at each analysis visit:

- PP NRS Improvement ≥ 4 from baseline
- PP NRS < 2</li>

In addition, proportion of subjects with PP NRS improvement ≥ 4 from baseline and IGA success (see Section 10.3.1) at Week 16 will be summarized on the ITT and PP population. The proportion of subjects will be presented using OC, non-responder and LOCF. The estimate of treatment unadjusted and strata-adjusted proportion differences with the corresponding two-sided 95% CI, and p-values from the CMH test will be presented.

Line plots for the change and percentage change from Baseline in PP NRS using OC on the ITT population will also be presented.

10.3.4. Sleep Disturbance Numeric Rating Scale (SD NRS)

The SD NRS is a scale to be used by the subjects to report the degree of their sleep loss related to PN.

The Baseline SD NRS will be determined based on the average of daily SD NRS (score ranging from 0 to 10) during the 7 days up to the treatment start (including until treatment start time) (rounding to nearest whole number is not permitted). A minimum of 4 daily scores out of the 7 days up to Baseline study day is required for this calculation. SD NRS at all following visits will be determined following the rules described in Table 8-2. If there are less than 4 non-missing assessments in the baseline diary window, the interval lower bound can be extended up to 7 additional days, one day at a time, to obtain the most recent 4 non-missing values.

Subjects will be asked the following question:

• "On a scale of 0 to 10, with 0 being 'no sleep loss related to the symptoms of my skin disease (prurigo nodularis)' and 10 being 'I did not sleep at all due to the symptoms of prurigo nodularis', how would you rate your sleep last night?"

Summary using OC will be provided on the ITT population. Absolute change and percentage change from Baseline will also be included in the summary.

Absolute and percentage change from Baseline at each analysis visits will be analyzed using ANCOVA with MI assuming MAR and using MMRM approach, including analysis center and body weight at randomization cut-off (< 90 kg and ≥ 90 kg) as factor and baseline as covariate on ITT population. The LSMeans, standard error of LSMeans, and 95% CI for change from baseline, as well as the difference in LSMeans between the treatment groups, the two-sided 95% CI, and associated p-value will be presented. Improvement in SD NRS will be calculated using Baseline as the reference point for change in SD NRS score.

The proportion of subjects with an improvement of SD NRS ≥ 4 will be summarized using OC and non-responder imputation on ITT population. The estimate of treatment unadjusted and strata-adjusted differences with the corresponding two-sided 95% confidence intervals, and p-values from the CMH test will be presented using non-responder imputation on ITT population.

Line plot for proportion of subjects with SD NRS improvement ≥ 4 using non-responder imputation will be presented on the ITT population.

Additionally the proportions of subjects with an improvement of SD NRS ≥ 4 from Baseline will be summarized by using at least 2 assessments, or 3 assessments, for calculation of weekly average SD NRS for sensitivity analysis. Proportions are summarized using non-responder imputation on ITT population.

### 10.3.5. Subject Sleep Diary

Subjects will be given a morning sleep diary (MSD) to record the quality of their sleep. The subject sleep diary is a modification of the consensus sleep diary and is designed to gather information about the subject's sleep pattern and how symptoms related to PN (e.g., itching, burning) affect their sleep.

Subjects will be instructed to complete the sleep diary (Questions 1 to 11) once daily in the morning (i.e., within 1 hour of getting out of bed), with the daily SD NRS. If a subject does not complete the sleep diary in the morning before a scheduled visit, the subject will be allowed to complete the assessment at the clinic visit.

The Baseline sleep diary metrics will be determined based on the average of daily sleep diary metrics respectively during the 7 days data up to the Baseline study day [including until treatment start time] (rounding to nearest whole number is not permitted). A minimum of 4 daily scores out of the 7 days up to Baseline study day is required for this calculation. If there are less than 4 non-missing assessments in the baseline diary window, the interval lower bound can be extended up to 7 additional days, one day at a time, to obtain the most recent 4 non-missing values. Sleep diary metrics at all other visits will be determined following the rules described in Table 8-2.

The sleep diary metrics will be derived as below (see Table 10-3) using questions in the morning based on morning sleep diary.

Table 10-3: Sleep Diary Metrics

| Sleep Parameter | SSD Items Used to Derive the Sleep Parameter |
|---|---|
| Sleep onset latency (SOL) | Q3 |
| Wakefulness after sleep onset (WASO) | Q5 + Q7 |
| Terminal WASO (TWASO) | Q9 – Q8 |
| Total awake time (TWT) | SOL+ WASO + TWASO |
| Time in bed (TIB) | Q9 – Q1 |
| Total sleep time (TST) | TIB – TWT |
| Sleep efficiency (SE) | (TST/TIB)*100 |
| WASO related to PN (WASO-PN) | Q5 |
| Number of WASO related to PN (NWASO-PN) | Q4 |

Sleep diary metrics will be summarized as continuous variables on observed cases on the ITT population. Change from Baseline in sleep diary metrics will also be summarized.

If Q8 (wake up time) is after Q9 (get out of bed), then Terminal WASO (Q9-Q8) will be set to 0.


If Q8 (wake up time) is before Q1 (get into bed), the time on the next day will be considered for Q9 as only time is collected.

If the duration between Q1 and Q9 is >24 hours, this data will be considered as uncalculable and the derived parameters (total awake time and total sleep time) are set to missing.

If total sleep time is negative, it will be considered as missing (not zero) for analysis. The same applies for total awake time.

No hypothesis testing will be performed.

10.3.6. PN Associated Pain Intensity and Frequency

Subjects will be asked to report the intensity and frequency of pain they endure related to their PN. Pain intensity is captured using a NRS.

Subjects will rate the frequency of their pain on a 6-point scale (0 = Never, 1 = Less than once a week, 2 = 1-2 Days a week, 3 = 3-4 Days a week, 4 = 5-6 Days a week, 5 = Everyday) in response to the following question:

"How often would you say that you experience pain from your skin disease (prurigo nodularis)?"

Subjects will rate the intensity of their pain using an 11-point NRS (0-10) in response to the following question:

"On a scale of 0 to 10, with 0 being "no pain" and 10 being "the worst unbearable pain", how would you rate the pain associated with your skin disease (prurigo nodularis) at the worst moment during the past week?"

Summaries using OC will be generated for PN associated pain frequency and intensity at Baseline, Week 4, Week 8, Week 12, and Week 16 on ITT population. Pain frequency will be summarized as a categorical variable. Pain intensity will be summarized as a continuous variable. Absolute change from Baseline in PN associated pain intensity from Baseline will also be summarized.

No hypothesis testing will be performed.

10.3.7. Patient Global Assessment of Disease (PGAD)

For the PGAD, subjects will be asked to rate their overall impression of their skin disease (prurigo nodularis) severity using a 5-point scale (0 = clear, 1 = almost clear, 2 = mild, 3 = moderate, 4 = severe). Subjects will be asked the following question:

"Overall, how would you describe your skin disease (prurigo nodularis) right now?"

PGAD will be collected at Baseline/Day 1, Week 1, Week 16 and Early Termination and be summarized for Baseline, Week 1 and Week 16 as a categorical variable using OC on the ITT population.

The proportion of subjects reporting low disease activity (clear, almost clear, or mild) based on PGAD will be summarized using OC on the ITT population. The estimate of treatment unadjusted and strata-adjusted differences with the corresponding two-sided 95% CI, and p-values from the CMH test will be presented.

#### 10.3.8. Patient Global Assessment of Treatment (PGAT)

The PGAT utilizes a 5-point Likert scale (0 = poor, 1 = fair, 2 = good, 3 = very good, 4 = excellent) or subjects to rate the way they feel their skin disease (prurigo nodularis) is responding to the study treatment. Subjects will be asked the following question at Week 16 and Early Termination:

"How would you rate the way your skin disease (prurigo nodularis) responded to the study medication?"

PGAT will be summarized as a categorical variable for Week 16 using OC on the ITT population.

The proportion of subjects satisfied with study treatment (good, very good, or excellent) based on PGAT will be summarized using OC on the ITT population. The estimate of treatment unadjusted and strata-adjusted differences with the corresponding two-sided 95% CI, and p-values from the CMH test will be presented.

#### 10.3.9. Dermatology Life Quality Index

The DLQI is a validated 10-item questionnaire covering domains including symptoms/feelings, daily activities, leisure, work/school, personal relationships, and treatment.

The subject will rate each question ranging from 0 (not at all) to 3 (very much). The DLQI total score is calculated by summing each questionnaire. Total score will have a maximum score of 30 and a minimum of 0. The higher the score, the more quality of life is impaired.

DLQI will be collected at Baseline/Day 1, Week 4, Week 16 and Early Termination. DLQI total score will be summarized as a continuous variable using OC on the ITT population for Baseline, Week 4 and Week 16. Absolute change from Baseline in DLQI total score will also be summarized.

Absolute change from Baseline in DLQI total score at Week 4 and Week 16 will be analyzed using ANCOVA with MI assuming MAR and using MMRM approach, including analysis center and body weight at randomization cut-off (< 90 kg and ≥ 90 kg) as factor and baseline as covariate. The LSMeans, standard error of LSMeans, and 95% CI for change from baseline, as well as the difference in LSMeans between the treatment groups, the two-sided 95% CI, and associated p-value will be presented on ITT population.

Improvement of  $\geq 4$  in DLQI will be calculated using Baseline as the reference point for change in DLQI total score. The proportion of subjects with an improvement of  $\geq 4$  will be summarized on the ITT population using OC and non-responder imputation. The estimate of treatment unadjusted and strata-adjusted differences with the corresponding two-sided 95% CI, and p-values from the Cochran-Mantel-Haenszel test using non-responder will be presented for ITT population.

A line plot for proportion of subjects with DLQI improvement ≥4 using non-responder imputation will be presented on the ITT population.

#### 10.3.10. Hospital Anxiety and Depression Scale (HADS)

HADS is a 14-question validated questionnaire completed by the subject. Each question has a multiple choice answer which is scored between 0 and 3. Questions are identified as relating to anxiety (A) or depression (D) and a summation for each area is performed leading to a total score of 0 to 21 for each area. Scores of 0 to 7 are considered normal, 8 to 10 are borderline, and  $\geq$  11 indicate clinical effects.

HADS will be collected at Baseline/Day 1, Week 16 and Early Termination and subscales will be summarized separately for each subscale (Total Score Anxiety and Total Score Depression) as continuous

variable using OC for Baseline and Week 16. on the ITT Population. Absolute change from Baseline in HADS subscale scores will also be summarized.

Absolute change from Baseline in HADS subscale scores will be analyzed for Week 16 using ANCOVA using observed case, including analysis center and body weight at randomization cut-off (< 90 kg and ≥ 90 kg) as factor and baseline as covariate. The LSMeans, standard error of LSMeans, and 95% CI for change from baseline, as well as the difference in LSMeans between the treatment groups, the two-sided 95% CI, and associated p-value will be presented.

#### 10.3.11. EuroQoL 5 Dimension Instrument

The EQ-5D instrument is a validated questionnaire, completed by the subject and consists of 2 parts. The first part consists of 5 multiple choice QoL questions and the second is a 100 point VAS scale with 0 being "Worst imaginable health state" and 100 being "Best imaginable health state".

EQ-5D VAS will be collected at Baseline/Day 1, Week 16 and Early Termination and be summarized as a continuous variable using OC for Baseline and Week 16 on the ITT Population. Absolute change from Baseline in EQ-5D VAS will also be summarized using OC.

Absolute change from Baseline in EQ-5D VAS at Week 16 will be analyzed using ANCOVA using observed case, including analysis center and body weight at randomization cut-off (< 90 kg and ≥ 90 kg) as factor and baseline as covariate. The LSMeans, standard error of LSMeans, and 95% CI for change from baseline, as well as the difference in LSMeans between the treatment groups, the two-sided 95% CI, and associated p-value will be presented.

Five dimensions of EQ-5D (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) will be summarized as a categorical variable using OC.

#### 10.3.12. Rescue Therapy Used

Subjects who used either medication or procedure as rescue therapy will be summarized using OC.

The number and percentage of subjects receiving any prior or concomitant rescue therapy will be summarized by rescue treatment type (topical, phototherapy, systemic, intralesional corticosteroids, and corresponding subgroups), preferred term within treatment type and overall.

If a subject used multiple rescue therapies (e.g., use a rescue therapy again after completing to use the previous one), count both therapies into each duration.

In addition, the time to first rescue therapy use will be calculated. The data will be analyzed using Kaplan-Meier methodology by presenting the point estimates of the quartiles estimates with the corresponding 95% CI. Kaplan-Meier estimates of time to first rescue therapy use will be summarized by visit. Subjects who do not use any rescue therapy will be censored for the analysis and date of last visit will be used as the censoring date. Subjects who discontinued without intake of rescue therapy will also be censored as described above. A Kaplan-Meier curve will also be provided.

Filing requirements: TMF

# 11. Pharmacokinetics

The serum concentration of Nemolizumab will be assessed at Baseline, Week 4, Week 8, Week 12, Week 16, Week 24 Follow-up and Early Termination visit. PK analyses are required during any unscheduled visit conducted for safety reasons. As a guideline, PK samples should be collected at approximately the same time of day throughout the study, to the extent possible, before study drug injection (pre-dose samples).

#### 11.1. Pharmacokinetic Concentration Presentation

Serum concentration data (unit: ng/mL) will be summarized on the PK analysis population by visit and by body weight at randomization cut-off (< 90 kg or ≥ 90 kg) from Baseline to Week 24, using the following statistics: arithmetic mean, SD, coefficient of variation (CV), geometric mean, geometric CV, median, minimum, maximum, 95% CI of the arithmetic mean, and number below the limit of quantification (BLQ).

Mean and individual (spaghetti plot) serum concentration(s) will be plotted by visit and by body weight at randomization cut-off (< 90 kg or ≥ 90 kg) on both a linear and semi-logarithmic scale on the PK analysis population (2 plots).

Individual serum concentrations will be listed on the PK analysis population.

# 11.2. Pharmacokinetic and Pharmacodynamics Parameters Estimation

PopPK and PK/PD analyses will be conducted by a designated CRO using pre-specified models based on existing information from previous studies in adults. For efficacy, PD endpoints are defined as the 2 primary clinical efficacy endpoints of the study: PP NRS responder and IGA success. If needed, specific PK/PD analyses might be conducted for safety.

Results of PopPK and PK/PD analyses will not be included in the CSR final TFLs. PopPK and PK/PD analyses will be described in an ad hoc Modeling & Simulation Plan. PopPK and PK/PD analyses results will be described in ad hoc Modeling & Simulation Report.

### 11.3. Biomarkers

Blood and stratum corneum (D-Squames) samples will be collected from approximately 100 subjects at selected sites to investigate the effect of Nemolizumab (CD14152) on selected RNA and protein biomarkers, including but not limited to IL-31. Optional skin biopsies for RNA and immunohistochemistry analyses will be collected from approximately 30 subjects at selected sites who sign the additional consent form. Samples will be collected at Baseline and Week 16.

These biomarker data will be analyzed according to a separate Analysis Plan and presented in a separate biomarkers report.

Filing requirements: TMF

# 12. Immunogenicity

Blood samples to assess anti-Nemolizumab ADA will be collected at Baseline, Week 8, Week 16, and Early Termination. Immunogenicity analyses will be summarized on the PK analysis population.

Details related to the processing of serum samples and the assessments of ADA will be described in the bioanalytical plan, which will be finalized before the beginning of sample analysis. Results will be described in the bioanalytical report, which will be included as an appendix in the final clinical study report.

Incidence of ADA results will be summarized (absolute occurrence and percent of subjects) by treatment group at each visit. The concentration of ADA titer (ng/mL) and neutralizing antibodies (ng/mL) will be summarized depending on the data requirement.

The number and percentage of subjects with treatment related ADA will be summarized. A treatment-related ADA is defined when the Baseline screening or confirmatory ADA result is negative and the post-baseline confirmatory ADA result is positive in the Nemolizumab treated group only.

# 13. Safety

All safety data will be summarized and listed on the SAF population.

Safety assessments will be conducted for all subjects at the screening visit (upon signing of the ICF) and at every subsequent visit. Safety will be assessed on the basis of AEs (including TEAEs, AESIs, SAEs and adjudicated AEs), physical examination and vital signs, clinical laboratory tests, electrocardiogram (ECG), respiratory examination and assessments. Summary of all safety endpoints will be presented for each treatment group.

#### 13.1. Adverse Events

AEs will be coded using MedDRA Version 25.0.

Treatment-emergent AEs (TEAEs), defined as those AEs occurring after the first administration of study treatment until the last study visit, will be tabulated in frequency tables by System Organ Class (SOC) and Preferred Term (PT) based on the Medical Dictionary for Regulatory Activities for treatment and follow-up periods. Missing date information will be handled using the algorithm described in Section 8.3.

TEAEs during treatment period are defined as AEs with onset date on or after the first dose date till 4 weeks after the last treatment or early discontinuation date whichever is earlier. TEAEs during follow-up period are defined as AEs with onset date post treatment period (4 weeks after the last treatment or early discontinuation date, whichever is earlier) to follow-up visit date.

AEs will be summarized using the number and percent of subjects reporting each SOC and PT and sorted alphabetically by SOC and by descending frequency of PT within SOC.

Subjects who experienced multiple events within the same SOC will be counted once in the SOC summary. Subjects who experienced multiple occurrences of events with the same PT will be counted once in the PT summary.

When summarizing by causality or maximum severity, if a subject experiences more than 1 occurrence of the same AE, the occurrence with the greatest severity and the closest association with the study drug will be used in summary tables. TEAEs related to study drug/study procedure are those that are identified as reasonable possibility. If relationship or severity are missing, the event will be considered as AE related to study drug/study procedure or severe AE.

An AESI is a noteworthy treatment-emergent event for the study drug that should be monitored closely and reported promptly. An AESI can be either serious or non-serious. Based on the potential risks of Nemolizumab and the risks associated with biologics in general (i.e., class effects), the following AEs will be considered as AESIs:

- Injection-related reactions,
- Newly diagnosed asthma or worsening of asthma,
- Infections.
- · Peripheral oedema: limbs, bilateral,
- Facial oedema
- Elevated ALT or AST (> 3 x ULN) in combination with elevated bilirubin (> 2 x ULN).

The following summary tables for TEAEs will be presented for all TEAEs (i.e., TEAE all causalities) and study drug related TEAEs separately by treatment period and follow-up period.

## Overall Summary of TEAEs :

- Overall summary table includes summary of subjects reporting TEAEs,
- Overall summary table includes summary of subjects reporting TEAEs by Country,
- TEAE by maximum severity [Mild, Moderate, Severe],
- TEAE related to study drug,
- TEAE related to study drug by maximum severity [Mild, Moderate, Severe],
- TEAE related to protocol procedure,
- Serious TEAE,
- Serious TEAE related to study drug,
- Severe TEAE,
- TEAE of special interest,
- TEAE leading to study drug interruption,
- TEAE leading to study drug withdrawal,
- TEAE leading to study discontinuation,
- TEAE leading to death,
- TEAE related to study drug leading to death
- TEAEs by SOC and PT
- TEAEs by SOC and PT and by Country
- Serious TEAEs by SOC and PT
- TEAEs by SOC, PT and maximum severity
- Severe TEAEs by SOC and PT
- TEAEs leading to study drug withdrawal by SOC and PT
- TEAEs leading to study discontinuation by SOC and PT
- TEAEs of special interest by category by SOC and PT
- TEAEs occurred in > 5% of subjects by SOC and PT
- TEAEs occurred in > 5% of subjects by Preferred Term
- Adjudicated TEAEs by SOC and PT
- TEAEs of Asthma and AESI reported by investigator with adjudication outcome by IAC
- Confirmed adjudicated TEAEs by SOC, PT and maximum severity
- TEAEs of special interest by category, SOC, PT and maximum severity

For overall study period which includes all periods (treatment and follow-up), the following summary tables will also be presented and repeated for all TEAEs (all causalities) and study drug related TEAEs.

• Overall Summary of TEAEs

This document is confidential.

Filing requirements: TMF

TEAEs by SOC and PT

For the subset of subjects with COVID-19 infection, the following summary tables will be provided additionally for all TEAEs and study drug related TEAEs, separately.

- Overall summary of TEAEs
- TEAEs by SOC and PT
- Serious TEAEs, by SOC and PT
- TEAEs of Special Interest by category by SOC and PT

In addition, the exposure-adjusted incidence rate (i.e., number of subjects per 100 patient-years) will be summarized for all TEAEs (all causalities) and study drug related TEAEs during treatment period.

Exposure-adjusted incidence rates of TEAEs is defined as the number of subjects exposed to treatment and experiencing a certain event divided by the total time of all subjects who are at risk for the event. Specially, for subjects with no event the exposure time is the time from the first drug intake to the end of treatment period. Exposure years is calculated as last study drug exposure date minus first study drug exposure date plus one, divided by 365.25 which is the number of days count in a year. This exposure year calculated for each subject is then added cumulatively and is derived for each treatment arm. So each treatment arm will have one value for exposure years (also known as "patient years"). The exposure year calculation is different in case of subjects who have completed the study or discontinued from the study or having withdrawn from the study due to any reason. Only the event occurred during the treatment period will account for calculation.

Subject listings will be presented for all

- TEAEs.
- TEAEs of special interest,
- Serious TEAEs.
- Severe TEAEs.
- TEAE leading to permanent discontinuation of study drug,
- TEAEs leading to deaths,
- Pre-treatment AEs,
- Adjudicated Asthma AEs,
- TEAE comments,
- Adjudicated Asthma AE comments by Independent Adjudication Committee.

Subject listings of TEAEs for subjects with COVID-19 infection will also be generated.

# 13.2. Laboratory Evaluations

### 13.2.1. Clinical Laboratory Evaluations

The hematology laboratory analyses, clinical chemistry laboratory analyses, and urinalyses will be performed at a central laboratory. Reference ranges will be supplied by the central laboratory and used by the investigator to assess the laboratory data for clinical significance and pathological changes. Reference ranges will be provided in the laboratory manual.

The following parameters will be reported for laboratory data.

- **Hematology:** Hemoglobin, hematocrit, white blood cell (WBC) count (with differential including eosinophils), red blood cell (RBC) count, platelet count, and mean cell volume (MCV).
- Chemistry: Creatinine, aspartate aminotransferase (AST), alanine aminotransferase (ALT), gamma glutamyltransferase (GGT), alkaline phosphatase, lactate dehydrogenase (LDH), total bilirubin, direct bilirubin, creatinine phosphokinase ([CPK], CPK isoenzyme test will be performed only if CPK is elevated to > 2.5 × ULN), albumin, total protein, uric acid, sodium, potassium, calcium, chloride, glucose, urea, total cholesterol, triglycerides, low-density lipoprotein (LDL), and high-density lipoprotein (HDL). Follicle-stimulating hormone (FSH) will be collected for postmenopausal subjects.
- Urinalysis: pH, glucose, ketones, blood, protein, leukocytes, nitrites, bilirubin, urobilinogen, and specific gravity.

Laboratory assessments are performed at Screening, Baseline/Day 1, Week 4, Week 8, Week 16, Early Termination and Week 24/Follow-up.

Hematology and chemistry laboratory data (absolute values and change from Baseline) will be summarized as continuous variables by visit (Baseline and scheduled visits only). Urinalysis laboratory data will be summarized by visit (Baseline and scheduled visits only). Last post-baseline, worst post-baseline and maximum post-baseline results will also be included in the summaries and will include unscheduled visits in the derivation. Worst post-baseline value will be defined as the highest or lowest value relative to the reference range. Parameters will be presented in alphabetically order.

Shift tables will be generated using the reference ranges (Low, Normal, High and Missing) for hematology and chemistry laboratory data. The number and percentage of subjects shifting from reference ranges between Baseline and each visit (scheduled visits only) will be summarized. Last, worst and maximum post baseline values will also be included in the shift tables and will include unscheduled visits in the derivation.

Summary of the number and percentage of subjects who met criteria of potential clinically significant (CS) value will be summarized (Baseline and scheduled visits only) for hematology and chemistry laboratory data. Last, worst and maximum post-baseline results will also be included in the summaries. Potentially CS ranges are listed in Section 21.4.

For statistical and graphical summaries of the laboratory tests, values below or above the limit of detection (e.g. '< 3' or '> 500') are substituted with the lower limit of detection minus 1% for values below the lower limit and are substituted with the upper limit of detection plus 1% for values above the upper limit (e.g. '< 3' is substituted by '2.97', '> 500' is substituted by '505'). In data listings, the values are shown including the < or > sign.

Distribution of continuous hematology and chemistry laboratory data (in particular, Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT), Alkaline Phosphatase (ALP), Total Bilirubin (BILI), Creatinine Kinase (CK) and Leukocytes (WBC)) will be displayed graphically as boxplot by treatment group for baseline and for each scheduled visits and the maximum post-Baseline (including unscheduled visits in the derivation) values.

Individual subject plots will be generated for all subjects with at least one abnormal result (outside of reference range). These plots will be provided for the chemistry laboratory parameters.


By-subject listing will be presented for all laboratory data. By-subject listing for subjects with at least one abnormal result will be provided for hematology and clinical chemistry. By-subject listing for subjects with at least one potentially CS result will be provided for hematology, clinical chemistry and urinalysis.

All laboratory data will be listed for the Safety population.

#### 13.2.2. Pregnancy Testing

All women of childbearing potential will have a serum pregnancy test at the screening visit and urine pregnancy tests (UPTs) at Baseline, Week 4, Week 8, Week 12 and Week 16, Early Termination visit, and Week 24/Follow-up. Pregnancy test results must be available prior to the administration of the study drug.

All test results including Tests not done will be summarized by visit on the Safety population.

All confirmed pregnancy test results together with the premenses status and childbearing potential assessment results will be listed on the Safety population.

## 13.2.3. Virology and TB Testing

Virology including HBsAg, HBcAb, hepatitis C, human immunodeficiency virus 1, and human immunodeficiency virus 2 antibodies will be assessed at the screening visit. Subjects with a positive HBcAb and a negative HBsAg will also be assessed for hepatitis B surface antibody. Subjects with positive HCV antibodies will have a confirmatory test for HCV (e.g., PCR). All virology and genomics results will be listed on the Safety population. All Immunoglobulin E results will also be listed on the Safety population.

Subjects will be assessed for TB infection with a QuantiFERON-TB Gold test at the screening visit. All TB test results will be listed on the Safety population.

### 13.3. Vital Signs

Vital signs will include pulse rate, systolic and diastolic blood pressure (after the subject has been sitting for at least 5 minutes) and body temperature.

Vital signs will be collected at the Screening visit and at Baseline/Day 1, Week 4, Week 8, Week 12 and Week 16, Early Termination visit, and at Week 24/Follow-up.

Height and weight will be measured at Screening for all subjects. Weight assessments will be conducted at Baseline/Day 1, and Week 16 and Early Termination.

All vital signs including height and weight (absolute values and change from Baseline) will be summarized as continuous (Baseline and scheduled visits only). Last post-Baseline results (including unscheduled visits in the derivation) will also be included.

The number and percentage of subjects who met criteria of potential CS value (Section 21.4) for vital signs and weight will be summarized (Baseline and scheduled visits only). Last post-Baseline results (including unscheduled visits in the derivation) will also be included.

Distribution of pulse rate, systolic and diastolic blood pressure will be displayed graphically as boxplot by treatment group for Baseline and each scheduled visit and maximum post-Baseline (including unscheduled visits in the derivation) values.

By-subject listing of subjects with potentially CS vital signs and weight will be provided.

All vital signs results will be listed on the Safety population.

### 13.4. ECG

A 12-lead electrocardiogram (ECG) will be performed and read centrally at Screening, Baseline/Day 1, Week 16 and Early Termination visit.

All ECG data (absolute values and change from Baseline) will be summarized as continuous variables by visit (Baseline and scheduled visits only). All parameters will be presented in alphabetically order.

The overall results of the ECGs recorded as 'Normal', 'Abnormal, NCS' or 'Abnormal, CS' will be summarized by treatment group and visit (scheduled visits only). Clinical significance will be determined by the investigator.

Additionally all ECG findings will be summarized with numbers and percentages by visit (Baseline and scheduled visits only.

All ECG results will be listed on the Safety population.

# 13.5. Physical Examination

Following body system assessments will be performed at Screening, Baseline/Day 1, Week 8, Week 16, Early Termination, and Week 24/Follow-up:

- Head, ears, eyes, nose, throat, neck (including thyroid),
- · Skin/integumentary system,
- Cardiovascular system,
- Respiratory system,
- · Gastrointestinal system,
- Musculoskeletal system,
- Lymph nodes,
- · Nervous system, and
- Extremities.

The number and percentage of subjects with physical examination results by body system classified as 'Normal', 'Abnormal, NCS' or 'Abnormal, CS' will be summarized (Baseline and scheduled visits only).

Shift from Baseline of the physical examination category will also be summarized by body system and by visit.

By-subject listing will be provided for subjects who have at least one abnormal result from any body system or who missed the assessment due to any reason.

All physical examination results will be listed on the Safety population.

# Sponsor: Galderma S.A./Galderma R&D, LLC; Protocol No.: RD.06.SPR.203065

#### 13.6. **Respiratory Assessments**

#### 13.6.1. Respiratory Examination

A respiratory examination consists of medical interview. Questions regarding medical history of asthma, wheeze, dyspnea, and cough, will be performed for all subjects at Screening. At Baseline/Day 1, Week 4, Week 8, Week 12, Week 16, Early Termination and Week 24/Follow-up questions are asked regarding:

- newly diagnosed (de novo) with Asthma / experience a worsening of Asthma since last visit
- newly diagnosed with Wheeze since last visit / experience a worsening of Wheeze since last visit
- newly diagnosed with Dyspnea since last visit / experience a worsening of Dyspnea since last visit
- newly diagnosed with Cough since last visit / experience a worsening of Cough since last visit

Newly diagnosed asthma or unexpected worsening of asthma are also reported as AESI. All Respiratory examination questionnaire results will be summarized with numbers and percentages by visit and listed on the Safety population.

#### 13.6.2. Peak Expiratory Flow

Peak expiratory flow (PEF) testing during the clinical study will be performed under the supervision of qualified study personnel. Peak expiratory flow measurements should consist of 3 good efforts, with the best result documented. Obtained PEF values will be compared to predicted values based on the subject's age, sex and height.

PEF testing will be performed for all subjects at screening, Baseline/Day 1, Week 8, Week 16, Early Termination, and Week 24/Follow-up visits. For subjects reporting a medical history of asthma, PEF testing will be performed at all visits during the clinical study. For subjects diagnosed with de novo asthma, PEF testing will be performed at all visits, starting with the visit in which the diagnosis was confirmed.

Following PEF parameters will be summarized as a continuous variable (Baseline and scheduled visits only):

- Actual peak expiratory flow rate
- Predicted peak expiratory flow rate
- Actual PEF of predicted value (%).

These PEF parameters will be summarized separately for the subset of subjects with and without history of asthma.

The number and percentage of subjects with PEF < 80% of predicted value will be summarized by treatment group, visit (baseline and scheduled visits only), and medical history of asthma (with and without history of asthma).

All PEF results will be listed on the Safety population.

#### 13.6.3. Asthma Control Test

Subjects with a medical history of asthma will take an Asthma Control Test (ACT) at Screening, Baseline/Day 1, Week 4, Week 8, Week 12 and Week 16, Early Termination visit, and Week 24/Follow-up.


Subjects with de novo asthma will complete the ACT testing beginning from de novo diagnosis and at all subsequent scheduled visits.

The ACT is composed of 5 questions. For each question, the subject will choose the best answer out of 5 possible answers. The test provides a numerical score ranging from 5 to 25 to assess asthma control; a higher score indicates better asthma control while a score of 19 or less indicates the subject's asthma may not be under control.

ACT total score (absolute values and change from Baseline) will be summarized as a continuous variable (Baseline and scheduled visits only).

The number and percentage of subjects with an ACT score ≤ 19 will be summarized (scheduled visits only).

The ACT results and the ACT score will be listed on the Safety population.

# 14. Changes from Analysis Planned in Protocol

In Sections 5.3 and 10.3, "Proportion of subjects with PP NRS improvement ≥ 4 from baseline and IGA success at Week 16" was added as endpoint.

In protocol Section 9.10 (Prior and Concomitant Therapy), concomitant medications/therapies are defined as any therapies taken during the study (i.e., from the screening visit to the end of study).

However, for the analysis purpose, concomitant medications/therapies are defined as medications/therapies which start or stop or ongoing on or after the 1st injection of study drug.

In protocol stratification variable weight is named 'body weight at baseline'. This wording is corrected to 'weight at randomization', to clarify that this is the body weight at the time of randomization and how this information is provided by the investigator.

#### 15. **Reference List**

1. Liublinska V., Rubin DB. Sensitivity analysis for a partially missing binary outcome in a two-arm randomized clinical trial. Stat Med. 2014 October 30; 33(24): 4170-4185. doi:10.1002/sim.6197.

# 16. Programming Considerations

All TFLs and statistical analyses will be generated using SAS® 9.4 or higher (SAS® Institute Inc., Cary, NC, USA) on a SAS Server. Changes to the software version (e.g. upgrades), or use of additional software consistent with the SAP will not be considered a violation of the SAP.

#### 16.1. General Considerations

All TFLs will be produced in accordance to Syneos Health QC Processes (see Section 17).

- A separate SAS program will be created for each output.
- Each output will be stored in a separate file.
- Output files will be provided in separate Word rtf and as combined PDF format including all outputs in one PDF file.
- Numbering of TFLs will follow International Conference on Harmonization (ICH) E3 Guidance.

# 16.2. Table, Figure, and Listing Format

#### 16.2.1. General

- All TFLs will be produced in landscape format, unless otherwise specified.
- All TFLs will be produced on paper size A4 using the Courier New font, size 8.
- The data displays for all TFLs will have a 1 inch binding margin on top and bottom of a landscape oriented page and a minimum 1.25 inch margin on the left side and a minimum of 0.75 inch right side.
- Headers and footers for figures will be in Courier New font, size 8.
- Legends will be used for all figures with more than 1 variable, group, or item displayed.
- TFLs will be in black and white (no color), unless otherwise specified.
- Specialized text styles, such as bolding, italics, borders, shading, and superscripted and subscripted text, will not be used in the TFLs, unless otherwise specified. On some occasions, superscripts 1, 2, or 3 may be used (see below).
- Only standard keyboard characters will be used in the TFLs. Special characters, such as non-printable control characters, printer-specific, or font-specific characters, will not be used. Hexadecimal-derived characters will be used, where possible, if they are appropriate to help display math symbols (e.g., μ). Certain subscripts and superscripts (e.g., cm2, Cmax) will be employed on a case-by-case basis.
- Mixed case will be used for all titles, footnotes, column headers, and programmer-supplied formats, as appropriate.

## 16.2.2. Headers

• All output should have the following header at the top left of each page:

```
Galderma Protocol RD.06.SPR.203065
Dry-run/Draft/Final
```

- All output should have Page n of N at the top corner of each page. TFLs are internally paginated in relation to the total length (i.e., the page number should appear sequentially as page n of N, where N is the total number of pages in the table).
- The date output was generated should appear along with the program name as a footer on each page.

# 16.2.3. Display Titles

- Each TFL are identified by the designation and a numeral. (i.e., Table 14.1.1.1). ICH E3 numbering is used. A decimal system (x.y and x.y.z) are used to identify TFLs with related contents. The title is centered. The analysis population are identified on the line immediately following the title. The title and table designation are single spaced. A solid line spanning the margins will separate the display titles from the table.
- Column headers. There will be 1 blank line between the last title and the solid line.

Table 14.1.1.1
Subject Disposition
Screened Population

## 16.2.4. Column Headers

- Column headings are displayed immediately below the solid line described above in Initial uppercase characters.
- In the case of efficacy tables, the variable (or characteristic) column will be on the far left followed by the treatment group column.
- For numeric variables, include "unit" in column or row heading when appropriate.
- Analysis population sizes will be presented for dose group in the column heading as "N=XX" (or in the row headings, if applicable). This is distinct from the 'n' used for the descriptive statistics representing the number of subjects in the analysis population.

## 16.2.5. Body of the Data Display

#### 16.2.5.1. General Conventions

Data in columns of a table or listing are formatted as follows:

- Alphanumeric values will be left-justified;
- Whole numbers (e.g., counts) will be right-justified; and
- Numbers containing fractional portions will be decimal aligned. The "%" is not presented for example "5 (0.6)"

#### **16.2.5.2.** Table Conventions

- Units will be included where available.
- If the categories of a parameter are ordered, then all categories between the maximum and minimum category are presented in the table, even if n=0 for all treatment groups in a given category that is between the minimum and maximum level for that parameter. For example, the frequency distribution for symptom severity would appear as:

| Severity | N |
|----------|---|
| Rating | |
| severe | 0 |
| moderate | 8 |
| mild | 3 |

Where percentages are presented in these tables, zero percentages will not be presented and so counts of 0 will be presented as 0 and not as 0 (0).

- If the categories are not ordered (e.g., Medical History, Reasons for Discontinuation from the Study, etc.), then only those categories for which there is at least 1 subject represented are included.
- An Unknown or Missing category will be added to each parameter for which information is not available for 1 or more subjects.
- Unless otherwise specified, the estimated mean, median, Q1 and Q3 for a set of values are printed
  out to 1 more significant digit than the original values, and standard deviations are printed out to 2
  more significant digits than the original values. The minimum and maximum should report the same
  significant digits as the original values. Missing descriptive statistics or p-values which cannot be
  estimated are reported as "-".
- Percentage values will be printed to one decimal place without the "%", with the "." in alignment, one space after the count (e.g., 7 (12.8), 13 (5.4)). Unless otherwise noted, for all percentages, the number of subjects in the analysis set for the treatment group who have an observation will be the denominator. Percentages after zero counts will not be displayed and percentages equating to 100% will be presented as 100, without decimal places.
- Tabular display of data for medical history, prior/concomitant medications, and all tabular displays of
  adverse event data are presented by the body system, treatment class, or SOC. The body system,
  drug class and SOC are displayed in alphabetically order. Within body system, drug class and SOC,
  preferred term will be display in descending frequency. If incidence for more than 1 preferred term is
  identical, they should then be sorted alphabetically.
- P-values will be output in the format: '0.xxxx', where xxx is the value rounded to 4 decimal places. Every p-value less than 0.0001 will be presented as "<0.0001". If the p-value is returned as >0.9999, then present as ">0.9999".
- The percentage of subjects is normally calculated as a proportion of the number of subjects assessed in the relevant treatment group (or overall) for the analysis population presented. However, careful consideration is required in many instances due to the complicated nature of selecting the denominator, usually the appropriate number of subjects exposed. These details are described in footnotes or programming notes.

- For categorical summaries (number and percentage of subjects) where a subject can be included in
  more than one category, it is described in a footnote or programming note as needed if the subject
  are included in the summary statistics for all relevant categories or just 1 category and the criteria for
  selecting the criteria.
- Where a category with a subheading (such as system organ class) has to be split over more than
  one page, output the subheading followed by "(continued)" at the top of each subsequent page. The
  overall summary statistics for the subheading should only be output on the first relevant page.

# 16.2.5.3. Listing Conventions

- Listings will be sorted for presentation in order of subject number, visit/collection day, and visit/collection time.
- Missing data will be represented on subject listings as either a hyphen ('-') with a corresponding footnote ('- = unknown or not evaluated'), or as 'N/A', with the footnote 'N/A = not applicable', whichever is appropriate.
- Dates will be printed in SAS DATE9.format ('DD\_MMM\_YYYY': 01JUL2000). Missing portions of
  dates will be represented on subject listings as dashes (--JUL2000). Dates that are missing because
  they are not applicable for the subject will be output as 'N/A', unless otherwise specified.
- All observed time values will be presented using a 24-hour clock HH:MM or HH:MM:SS format (e.g., 11:26:45, or 11:26). Time will only be reported if it was measured as part of the study.
- Units will be included where available.

### **16.2.5.4.** Figure Conventions

• Unless otherwise specified, for all figures, study visits will be displayed on the X-axis and endpoint (e.g., treatment mean change from Baseline) values will be displayed on the Y-axis.

# 16.2.6. Footnotes

- A solid line spanning the margins will separate the body of the data display from the footnotes.
- All footnotes will be left justified with single-line spacing immediately below the solid line underneath
  the data display.
- Footnotes will always begin with 'Notes:' if an informational footnote, or 1, 2, 3, etc. if a reference footnote. Each new footnote will start on a new line, where possible.
- Subject specific footnotes are avoided, where possible.
- Footnotes will be used sparingly and add value to the TFL. If more than 10 lines of footnotes are
  planned, then a cover page is strongly recommended to be used to display footnotes, and only those
  essential to comprehension of the data will be repeated on each page.
- The last line of the footnote section will be a standard source line that indicates the name of the program used to produce the data display, date the program was run, the date of extraction indicated

```
with "Data Cut-off: DDMMMYYYY" and the listing source (i.e., 'Program: t-14-01-03-02-01.sas, Run date: 16MAR2021 12:57', date cut-off: DDMMMYYYY, Listing Source(s): 16.x.y.z).
```

 Sources and/or cross-references in footnotes will use the keyword prefix (in singular form) for each reference and will be separated by a comma when multiple cross-references are displayed. Example

Listing source: 16.2.1.1

# 17. Quality Control

SAS programs are developed to produce output such as analysis data sets, summary tables, data listings, figures or statistical analyses. An overview of the development of programs is detailed in Syneos Health Developing Statistical Programs Standard Operation Procedure (SOP) (3907).

Syneos Health SOPs Developing Statistical Programs (3907) and Conducting the Transfer of Biostatistical Deliverables (SDTM, ADaM, TFL) (3908) describes the quality control procedures that are performed for all SAS programs and output. Quality control is defined here as the operational techniques and activities undertaken to verify that the SAS programs produce the output by checking for their logic, efficiency and commenting and by review of the produced output. A detailed description of project specific QC procedure can be found in the document "SAS Programming and Validation Plan" (version 1.0, dated 18-May-2020).

#### **Index of Tables** 18.

This section contains lists of the tables tentatively planned for this study. Changes in the number or content of planned listings are not considered deviations from this SAP.

| Header | Table<br>Number | Name | Analysis Set |
|---|---|---|---|
| 14. | | TABLES AND FIGURES | |
| 14.1 | 1 | Demographic Data Summary Tables | |
| 14.1.1 | 1 | Subject Disposition | |
| | 14.1.1.1 | Subject Accounting by Overall, Country and Site | Screened Subjects |
| | 14.1.1.2 | Subject Accounting by Visit | ITT Population |
| | 14.1.1.3 | Summary of Subject Disposition | ITT Population |
| | 14.1.1.4 | Summary of Subject Disposition by Site | ITT Population |
| | 14.1.1.5 | Summary of Screen Failure | Screened Subjects |
| | 14.1.1.6 | Summary of Analysis Populations | ITT Population |
| 14.1.2 | | Protocol Deviations | |
| | 14.1.2.1 | Summary of Major Protocol Deviations | ITT Population |
| | 14.1.2.2 | Summary of Major Protocol Deviations by Site | ITT Population |
| 14.1.3 | | Demographic and Baseline Characteristics | |
| 14.1.3.1 | | Subject Demographic and Baseline Characteristics | |
| | 14.1.3.1.1 | Subject Demographic and Baseline Characteristics | ITT Population |
| W | 14.1.3.1.2 | Subject Demographic and Baseline Characteristics | Safety Population |
| | 14.1.3.1.3 | Subject Demographic and Baseline Characteristics | PP Population |
| | 14.1.3.1.4 | Subject Demographic and Baseline Characteristics | PK Analysis |
| | 111101111 | Cabjeet Bernegrapine and Baconine Characteriones | Population |
| 14.1.3.2 | | Baseline Disease Characteristics | |
| 1111012 | 14.1.3.2.1 | Summary of Baseline Disease Characteristics | ITT Population |
| | 14.1.3.2.2 | Summary of Baseline Disease Characteristics | Safety Population |
| | 14.1.3.2.3 | Summary of Baseline Disease Characteristics | PP Population |
| | 14.1.3.2.4 | Summary of Baseline Disease Characteristics | PK Analysis |
| | 11.1.0.2.1 | Culturally of Buscimic Biocust Characterious | Population |
| | 14.1.3.2.5 | Summary of Proportion of Subjects with Differences between Randomization Stratification and Actual Stratification | ITT Population |
| 14.1.3.3 | 9 | Medical History, Medical and Surgical Procedures | |
| , | 14.1.3.3.1 | Summary of Previous and Ongoing Medical History | ITT Population |
| ). | 14.1.3.3.2 | Summary of Prior Medical and Surgical Procedures before Informed Consent Signed | ITT Population |
| × | 14.1.3.3.3 | Summary of Prior Medical and Surgical Procedures during Screening Period | ITT Population |
| | 14.1.3.3.4 | Summary of Concomitant Medical and Surgical<br>Procedures during Treatment Period | ITT Population |
| | 14.1.3.3.5 | Summary of Concomitant Medical and Surgical<br>Procedures during Follow-up Period | ITT Population |
| | 14.1.3.3.6 | Summary of Rescue Medical and Surgical<br>Procedures during Treatment Period | ITT Population |
| | 14.1.3.3.7 | Summary of Rescue Medical and Surgical<br>Procedures during Follow-up Period | ITT Population |
| 14.1.4 | | Medications | |
| | 14.1.4.1 | Summary of Prior Medications before Informed Consent Signed by ATC level and Preferred Term | ITT Population |

| Header | Table<br>Number | Name | Analysis Set |
|---|---|---|---|
| | 14.1.4.2 | Summary of Prior Medications during Screening<br>Period by ATC level and Preferred Term | ITT Population |
| | 14.1.4.3 | Summary of Concomitant Medications during Treatment Period by ATC level and Preferred Term | ITT Population |
| | 14.1.4.4 | Summary of Concomitant Medications during Follow-<br>up Period by ATC level and Preferred Term | ITT Population |
| | 14.1.4.5 | Summary of Rescue Medications during Treatment Period by ATC level and Preferred Term | ITT Population |
| | 14.1.4.6 | Summary of Rescue Medications during Follow-up<br>Period by ATC level and Preferred Term | ITT Population |
| 14.1.5 | | Extent of Exposure and Treatment Compliance | |
| | 14.1.5.1 | Summary of Exposure to Study Drug | Safety Population |
| 14.2 | 1 | Efficacy Data Summary Tables | & 8 |
| 14.2.1 | | Primary Efficacy Parameters | |
| 14.2.1.1 | | Analysis of Primary Efficacy Endpoint: Improvement of >= 4 from Baseline in Peak Pruritus Numeric Rating Scale at Week 16 | |
| | 14.2.1.1.1 | Analysis of Proportion of Subjects with an<br>Improvement of >= 4 from Baseline in Weekly<br>Average PP NRS at Week 16 - Missing as Non-<br>Responder | ITT Population |
| | 14.2.1.1.3 | Sensitivity Analysis of Proportion of Subjects with an<br>Improvement of >= 4 from Baseline in Weekly<br>Average PP NRS at Week 16 - Missing as Non-<br>Responder | PP Population |
| | 14.2.1.1.5 | Sensitivity Analysis of Proportion of Subjects with an<br>Improvement of >= 4 from Baseline in Weekly<br>Average PP NRS at Week 16 - Tipping Point<br>Analysis | ITT Population |
| | 14.2.1.1.7 | Sensitivity Analysis of Proportion of Subjects with an Improvement of >= 4 from Baseline in Weekly Average PP NRS at Week 16 - Multiple Imputation (MI) Method with Missing at Random (MAR) Assumption | ITT Population |
| | 14.2.1.1.8 | Sensitivity Analysis of Proportion of Subjects with an Improvement of >= 4 from Baseline in Weekly Average PP NRS at Week 16 - Multiple Imputation (MI) Method with Missing Not at Random (MNAR) Assumption | ITT Population |
| | 14.2.1.1.9 | Sensitivity Analysis of Proportion of Subjects with an<br>Improvement of >= 4 from Baseline in Weekly<br>Average PP NRS at Week 16 – LOCF | ITT Population |
| | 14.2.1.1.10 | Sensitivity Analysis of Proportion of Subjects with an<br>Improvement of >= 4 from Baseline in Weekly<br>Average PP NRS at Week 16 – OC | ITT Population |
| | 14.2.1.1.11 | Sensitivity Analysis of Proportion of Subjects with an<br>Improvement of >= 4 from Baseline in Weekly<br>Average PP NRS at Week 16 using Actual<br>Stratifications - Missing as Non-Responder | ITT Population |
| Header | Table<br>Number | Name | Analysis Set |
|---|---|---|---|
| | 14.2.1.1.13 | Sensitivity Analysis of Proportion of Subjects with an<br>Improvement of >= 4 from Baseline in Weekly<br>Average PP NRS at Week 16 - Missing as Non-<br>Responder | ITT Population –<br>Removal of<br>COVID-19 affected<br>Visits |
| | 14.2.1.1.14 | Sensitivity Analysis of Proportion of Subjects with an Improvement of >= 4 from Baseline in Weekly Average PP NRS by Visit using at least 2 Assessments - Missing as Non-Responder | ITT Population |
| | 14.2.1.1.15 | Sensitivity Analysis of Proportion of Subjects with an Improvement of >= 4 from Baseline in Weekly Average PP NRS by Visit using at least 3 Assessments - Missing as Non-Responder | ITT Population |
| | 14.2.1.2.1 | Analysis of Proportion of Subjects with an IGA Success at Week 16 - Missing as Non-Responder | ITT Population |
| | 14.2.1.2.3 | Sensitivity Analysis of Proportion of Subjects with an IGA Success at Week 16 - Missing as Non-Responder | PP Population |
| | 14.2.1.2.5 | Sensitivity Analysis of Proportion of Subjects with an IGA Success at Week 16 - Tipping Point Analysis | ITT Population |
| | 14.2.1.2.7 | Sensitivity Analysis of Proportion of Subjects with an IGA Success at Week 16 - Multiple Imputation (MI) Method with Missing at Random (MAR) Assumption | ITT Population |
| | 14.2.1.2.8 | Sensitivity Analysis of Proportion of Subjects with an IGA Success at Week 16 - Multiple Imputation (MI) Method with Missing Not at Random (MNAR) Assumption | ITT Population |
| | 14.2.1.2.9 | Sensitivity Analysis of Proportion of Subjects with an IGA Success at Week 16 – LOCF | ITT Population |
| | 14.2.1.2.10 | Sensitivity Analysis of Proportion of Subjects with an IGA Success at Week 16 – OC | ITT Population |
| | 14.2.1.2.11 | Sensitivity Analysis of Proportion of Subjects with an IGA Success at Week 16 using Actual Stratifications - Missing as Non-Responder | ITT Population |
| | 14.2.1.2.13 | Sensitivity Analysis of Proportion of Subjects with an IGA Success at Week 16 - Missing as Non-Responder | ITT Population –<br>Removal of<br>COVID-19 affected<br>Visits |
| 14.2.2 | | Key Secondary Efficacy Parameters Analysis of Key Secondary Efficacy Parameters: Improvement of >= 4 from Baseline in Peak Pruritus Numeric Rating Scale at Week 4 | |
| | 14.2.2.1.1 | Analysis of Proportion of Subjects with an Improvement of >= 4 from Baseline in Weekly Average PP NRS at Week 4 - Missing as Non-Responder | ITT Population |
| | 14.2.2.1.3 | Sensitivity Analysis of Proportion of Subjects with an Improvement of >= 4 from Baseline in Weekly Average PP NRS at Week 4 - Missing as Non-Responder | PP Population |
| | 14.2.2.1.5 | Sensitivity Analysis of Proportion of Subjects with an Improvement of >= 4 from Baseline in Weekly Average PP NRS at Week 4 - Tipping Point Analysis | ITT Population |

| Header | Table<br>Number | Name | Analysis Set |
|---|---|---|---|
| | 14.2.2.1.7 | Sensitivity Analysis of Proportion of Subjects with an Improvement of >= 4 from Baseline in Weekly Average PP NRS at Week 4 - Multiple Imputation (MI) Method with Missing at Random (MAR) Assumption | ITT Population |
| | 14.2.2.1.8 | Sensitivity Analysis of Proportion of Subjects with an Improvement of >= 4 from Baseline in Weekly Average PP NRS at Week 4 - Multiple Imputation (MI) Method with Missing Not at Random (MNAR) Assumption | ITT Population |
| | 14.2.2.1.9 | Sensitivity Analysis of Proportion of Subjects with an<br>Improvement of >= 4 from Baseline in Weekly<br>Average PP NRS at Week 4 – LOCF | ITT Population |
| | 14.2.2.1.10 | Sensitivity Analysis of Proportion of Subjects with an<br>Improvement of >= 4 from Baseline in Weekly<br>Average PP NRS at Week 4 – OC | ITT Population |
| | 14.2.2.1.11 | Sensitivity Analysis of Proportion of Subjects with an<br>Improvement of >= 4 from Baseline in Weekly<br>Average PP NRS at Week 4 using Actual<br>Stratifications - Missing as Non-Responder | ITT Population |
| | 14.2.2.1.13 | Sensitivity Analysis of Proportion of Subjects with an<br>Improvement of >= 4 from Baseline in Weekly<br>Average PP NRS at Week 4 - Missing as Non-<br>Responder | ITT Population –<br>Removal of<br>COVID-19 affected<br>Visits |
| 14.2.2.2 | | Analysis of Key Secondary Efficacy Parameters: Peak Pruritus Numeric Rating Scale < 2 at Week 4 and 16 | |
| | 14.2.2.2.1 | Analysis of Proportion of Subjects with Weekly<br>Average PP NRS < 2 at Weeks 4 and 16 - Missing<br>as Non-Responder | ITT Population |
| | 14.2.2.2.3 | Sensitivity Analysis of Proportion of Subjects with Weekly Average PP NRS < 2 at Weeks 4 and 16 - Missing as Non-Responder | PP Population |
| | 14.2.2.2.5 | Sensitivity Analysis of Proportion of Subjects with Weekly Average PP NRS < 2 at Weeks 4 and 16 - Tipping Point Analysis | ITT Population |
| | 14.2.2.2.7 | Sensitivity Analysis of Proportion of Subjects with Weekly Average PP NRS < 2 at Weeks 4 and 16 - Multiple Imputation (MI) Method with Missing at Random (MAR) Assumption | ITT Population |
| | 14.2.2.2.8 | Sensitivity Analysis of Proportion of Subjects with Weekly Average PP NRS < 2 at Weeks 4 and 16 - Multiple Imputation (MI) Method with Missing Not at Random (MNAR) Assumption | ITT Population |
| | 14.2.2.2.9 | Sensitivity Analysis of Proportion of Subjects with Weekly Average PP NRS < 2 at Weeks 4 and 16 – LOCF | ITT Population |
| | 14.2.2.2.10 | Sensitivity Analysis of Proportion of Subjects with Weekly Average PP NRS < 2 at Weeks 4 and 16 – OC | ITT Population |

| Header | Table<br>Number | Name | Analysis Set |
|---|---|---|---|
| | 14.2.2.2.11 | Sensitivity Analysis of Proportion of Subjects with Weekly Average PP NRS < 2 at Weeks 4 and 16 using Actual Stratifications - Missing as Non-Responder | ITT Population |
| | 14.2.2.2.13 | Sensitivity Analysis of Proportion of Subjects with Weekly Average PP NRS < 2 at Weeks 4 and 16 - Missing as Non-Responder | ITT Population –<br>Removal of<br>COVID-19 affected<br>Visits |
| | 14.2.2.2.14 | Sensitivity Analysis of Proportion of Subjects with Weekly Average PP NRS < 2 by visit using at least 2 Assessments - Missing as Non-Responder | ITT Population |
| | 14.2.2.2.15 | Sensitivity Analysis of Proportion of Subjects with Weekly Average PP NRS < 2 by visit using at least 3 Assessments - Missing as Non-Responder | ITT Population |
| 14.2.2.3 | | Analysis of Key Secondary Efficacy Parameters:<br>Sleep Disturbance Numeric Rating Scale<br>Improvement >= 4 at Week 4 and Week 16 | |
| | 14.2.2.3.1 | Analysis of Proportion of Subjects with an<br>Improvement >= 4 from Baseline in Weekly Average<br>SD NRS at Week 4 and Week 16 - Missing as Non-<br>Responder | ITT Population |
| | 14.2.2.3.3 | Sensitivity Analysis of Proportion of Subjects with an Improvement >= 4 from Baseline in Weekly Average SD NRS at Week 4 and Week 16 - Missing as Non-Responder | PP Population |
| | 14.2.2.3.5 | Sensitivity Analysis of Proportion of Subjects with an<br>Improvement >= 4 from Baseline in Weekly Average<br>SD NRS at Week 4 and Week 16 - Tipping Point<br>Analysis | ITT Population |
| | 14.2.2.3.7 | Sensitivity Analysis of Proportion of Subjects with an Improvement >= 4 from Baseline in Weekly Average SD NRS at Week 4 and Week 16 - Multiple Imputation (MI) Method with Missing at Random (MAR) Assumption | ITT Population |
| | 14.2.2.3.8 | Sensitivity Analysis of Proportion of Subjects with an Improvement >= 4 from Baseline in Weekly Average SD NRS at Week 4 and Week 16 - Multiple Imputation (MI) Method with Missing Not at Random (MNAR) Assumption | ITT Population |
| | 14.2.2.3.9 | Sensitivity Analysis of Proportion of Subjects with an<br>Improvement >= 4 from Baseline in Weekly Average<br>SD NRS at Week 4 and Week 16 – LOCF | ITT Population |
| | 14.2.2.3.10 | Sensitivity Analysis of Proportion of Subjects with an<br>Improvement >= 4 from Baseline in Weekly Average<br>SD NRS at Week 4 and Week 16 – OC | ITT Population |
| | 14.2.2.3.11 | Sensitivity Analysis of Proportion of Subjects with an Improvement >= 4 from Baseline in Weekly Average SD NRS at Week 4 and Week 16 using Actual Stratifications - Missing as Non-Responder | ITT Population |

| Header | Table<br>Number | Name | Analysis Set |
|---|---|---|---|
| | 14.2.2.3.13 | Sensitivity Analysis of Proportion of Subjects with an Improvement >= 4 from Baseline in Weekly Average SD NRS at Week 4 and Week 16 - Missing as Non-Responder | ITT Population –<br>Removal of<br>COVID-19 affected<br>Visits |
| | 14.2.2.3.14 | Sensitivity Analysis of Proportion of Subjects with an Improvement >= 4 from Baseline in Weekly Average SD NRS by visit using at least 2 Assessments - Missing as Non-Responder | ITT Population |
| | 14.2.2.3.15 | Sensitivity Analysis of Proportion of Subjects with an Improvement >= 4 from Baseline in Weekly Average SD NRS by visit using at least 3 Assessments - Missing as Non-Responder | ITT Population |
| 14.2.3 | | Secondary Efficacy Parameters | |
| 14.2.3.1 | | Secondary Efficacy Parameter: IGA | |
| w. | 14.2.3.1.1 | Summary of IGA - OC | ITT Population |
| (30) | 14.2.3.1.2 | Summary of IGA - OC | PP Population |
| | 14.2.3.1.3 | Summary of Proportion of Subjects with IGA Success | ITT Population |
| | 14.2.3.1.4 | Analysis of Proportion of Subjects with an IGA Success - Missing as Non-Responder | ITT Population |
| | 14.2.3.1.6 | Analysis of Proportion of Subjects with an IGA<br>Success - Missing as Non-Responder | PP Population |
| 14.2.3.2 | | Secondary Efficacy Parameter: Prurigo Activity Score | |
| | 14.2.3.2.1 | Summary of Categorical Parameter of Prurigo<br>Activity Score - OC | ITT Population |
| 5 | 14.2.3.2.2 | Summary of Continuous Parameter of Prurigo<br>Activity Score - OC | ITT Population |
| 15 m | 14.2.3.2.3 | Summary of Categorical Parameter of Prurigo<br>Activity Score - OC | PP Population |
| | 14.2.3.2.4 | Summary of Continuous Parameter of Prurigo<br>Activity Score - OC | PP Population |
| | 14.2.3.2.5 | Analysis of Proportion of Subjects with Prurigo<br>Activity Score Items 5a at all scheduled visits -<br>Missing as Non-Responder | ITT Population |
| | 14.2.3.2.6 | Analysis of Proportion of Subjects with Prurigo<br>Activity Score Items 5a at all scheduled visits -<br>Missing as Non-Responder | PP Population |
| | 14.2.3.2.7 | Analysis of Proportion of Subjects with Prurigo<br>Activity Score Items 5b at all scheduled visits -<br>Missing as Non-Responder | ITT Population |
| | 14.2.3.2.8 | Analysis of Proportion of Subjects with Prurigo<br>Activity Score Items 5b at all scheduled visits -<br>Missing as Non-Responder | PP Population |
| | 14.2.3.2.9 | Analysis of Change from Baseline in Prurigo Activity<br>Score Item 4 – ANCOVA using MI-MAR | ITT Population |
| | 14.2.3.2.10 | Analysis of Change from Baseline in Prurigo Activity<br>Score Item 4 – ANCOVA using MI-MAR | PP Population |
| 14.2.3.3 | | Secondary Efficacy Parameter: Peak Pruritus<br>Numeric Rating Scale | |
| | 14.2.3.3.1 | Summary of Weekly Average PP NRS – OC | ITT Population |
| 10 | 14.2.3.3.2 | Summary of Weekly Average PP NRS – OC | PP Population |

| Header | Table<br>Number | Name | Analysis Set |
|---|---|---|---|
| S | 14.2.3.3.3 | Summary of Proportion of Subjects with Weekly Average PP NRS Improvement >= 4 | ITT Population |
| | 14.2.3.3.4 | Analysis of Proportion of Subjects with Weekly Average PP NRS Improvement >= 4 from Baseline at Weeks 8 and 12 - Missing as Non-Responder | ITT Population |
| | 14.2.3.3.7 | Analysis of Proportion of Subjects with Weekly<br>Average PP NRS < 2 at Weeks 4, 8, 12 and 16 -<br>Missing as Non-Responder | ITT Population |
| | 14.2.3.3.10 | Analysis of Proportion of Subjects with Weekly<br>Average PP NRS < 3 at Weeks 4, 8, 12 and 16 -<br>Missing as Non-Responder | ITT Population |
| | 14.2.3.3.11 | Analysis of Change from Baseline in Weekly<br>Average PP NRS at Weeks 4, 8, 12 and 16 –<br>ANCOVA using MI-MAR | ITT Population |
| | 14.2.3.3.12 | Analysis of Change from Baseline for Weekly<br>Average PP NRS at Weeks 4, 8, 12 and 16 – MMRM<br>Analysis | ITT Population |
| | 14.2.3.3.13 | Analysis of Percentage Change from Baseline in Weekly Average PP NRS – ANCOVA using MI-MAR | PP Population |
| | 14.2.3.3.14 | Analysis of Percentage Change from Baseline for Weekly Average PP NRS – MMRM Analysis | PP Population |
| | 14.2.3.3.15 | Summary of Proportion of Subjects with Weekly<br>Average PP NRS Improvement >= 4 from Baseline<br>and IGA Success at Week 16 | ITT Population |
| | 14.2.3.3.16 | Summary of Proportion of Subjects with Weekly Average PP NRS Improvement >= 4 from Baseline and IGA Success at Week 16 | PP Population |
| | 14.2.3.3.17 | Analysis of Proportion of Subjects with Weekly Average PP NRS Improvement >= 4 from Baseline and IGA Success at Week 16 - Missing as Non- Responder | ITT Population |
| | 14.2.3.3.18 | Analysis of Proportion of Subjects with Weekly Average PP NRS Improvement >= 4 from Baseline and IGA Success at Week 16 - Missing as Non- Responder | PP Population |
| 14.2.3.4 | | Secondary Efficacy Parameter: Average Pruritus<br>Numeric Rating Scale | |
| | 14.2.3.4.1 | Summary of Weekly Average AP NRS – OC | ITT Population |
| × | 14.2.3.4.2 | Summary of Proportion of Subjects with Weekly Average AP NRS Improvement >= 4 from Baseline | ITT Population |
| | 14.2.3.4.3 | Analysis of Proportion of Subjects with Weekly Average AP NRS Improvement >= 4 from Baseline - Missing as Non-Responder | ITT Population |
| | 14.2.3.4.4 | Analysis of Proportion of Subjects with Weekly<br>Average AP NRS < 2 - Missing as Non-Responder | ITT Population |
| | 14.2.3.4.5 | Analysis of Change from Baseline in Weekly<br>Average AP NRS – ANCOVA using MI-MAR | ITT Population |
| | 14.2.3.4.6 | Analysis of Change from Baseline for Weekly<br>Average AP NRS – MMRM Analysis | ITT Population |
| | 14.2.3.4.7 | Analysis of Percentage Change from Baseline in Weekly Average AP NRS – ANCOVA using MI-MAR | PP Population |

| Header | Table<br>Number | Name | Analysis Set |
|---|---|---|---|
| | 14.2.3.4.8 | Analysis of Percentage Change from Baseline for Weekly Average AP NRS – MMRM Analysis | ITT Population |
| 14.2.3.5 | | Secondary Efficacy Parameter: Sleep Disturbance<br>Numeric Rating Scale | |
| | 14.2.3.5.1 | Summary of Weekly Average SD NRS - OC | ITT Population |
| | 14.2.3.5.2 | Summary of Proportion of Subjects with Weekly Average SD NRS Improvement >= 4 | ITT Population |
| | 14.2.3.5.3 | Analysis of Proportion of Subjects with Weekly Average SD NRS Improvement >= 4 from Baseline at all scheduled visits – Missing as Non-Responder | ITT Population |
| | 14.2.3.5.5 | Analysis of Change from Baseline in Weekly<br>Average SD NRS – ANCOVA using MI-MAR | ITT Population |
| | 14.2.3.5.6 | Analysis of Change from Baseline for Weekly<br>Average SD NRS – MMRM Analysis | ITT Population |
| | 14.2.3.5.7 | Analysis of Percentage Change from Baseline in Weekly Average SD NRS – ANCOVA using MI-MAR | PP Population |
| | 14.2.3.5.8 | Analysis of Percentage Change from Baseline for Weekly Average SD NRS – MMRM Analysis | PP Population |
| 14.2.3.6 | 14.2.3.6.1 | Secondary Efficacy Parameter: Subject Sleep Diary Summary of Weekly Average Sleep Diary Metrics – OC | ITT Population |
| 14.2.3.7 | | Secondary Efficacy Parameter: PN Associated Pain Intensity and Frequency | |
| | 14.2.3.7.1 | Summary of PN Associated Pain Intensity – OC | ITT Population |
| | 14.2.3.7.2 | Summary of PN Associated Pain Frequency - OC | ITT Population |
| 14.2.3.8 | | Secondary Efficacy Parameter: Patient Global<br>Assessment of Disease | |
| | 14.2.3.8.1 | Summary of PGAD – OC | ITT Population |
| | 14.2.3.8.2 | Analysis of Proportion of Subjects with Reporting<br>Low Disease Activity Based on PGAD - OC | ITT Population |
| 14.2.3.9 | | Secondary Efficacy Parameter: Patient Global Assessment of Treatment | |
| | 14.2.3.9.1 | Summary of PGAT – OC | ITT Population |
| | 14.2.3.9.2 | Analysis ITT Population of Proportion of Subjects<br>Satisfied with Study Treatment Based on PGAT –<br>OC | ITT Population |
| 14.2.3.10 | | Secondary Efficacy Parameter: Dermatology Life Quality Index | |
| | 14.2.3.10.1 | Summary of DLQI – OC | ITT Population |
| | 14.2.3.10.2 | Summary of Proportion of Subjects with DLQI<br>Improvement >= 4 | ITT Population |
| | 14.2.3.10.3 | Analysis of Proportion of Subjects with DLQI<br>Improvement >= 4 from Baseline at all scheduled<br>visits – Missing as Non-Responder | ITT Population |
| | 14.2.3.10.5 | Analysis of Change from Baseline in DLQI – ANCOVA using MI-MAR | ITT Population |
| | 14.2.3.10.6 | Analysis of Change from Baseline for DLQI – MMRM Analysis | ITT Population |
| 14.2.3.11 | | Secondary Efficacy Parameter: Hospital Anxiety and Depression Scale | |
| | 14.2.3.11.1 | Summary of HADS Total Scores – OC | ITT Population |

| Header | Table<br>Number | Name | Analysis Set |
|---|---|---|---|
| | 14.2.3.11.2 | Analysis of Change from Baseline in HADS Total<br>Scores – ANCOVA using OC | ITT Population |
| 14.2.3.12 | | Secondary Efficacy Parameter: EuroQoL 5 Dimension Instrument | |
| | 14.2.3.12.1 | Summary of EQ-5D Parameters- OC | ITT Population |
| | 14.2.3.12.2 | Summary of EQ-5D VAS – OC | ITT Population |
| | 14.2.3.12.3 | Analysis of Change from Baseline in EQ-5D VAS – ANCOVA using OC | ITT Population |
| 14.2.3.13 | | Rescue Therapy | |
| | 14.2.3.13.1.1 | Incidence of Medication of Rescue Therapy | ITT Population |
| | 14.2.3.13.1.2 | Incidence of Procedure of Rescue Therapy | ITT Population |
| | 14.2.3.13.1.3 | Time to First Rescue Therapy | ITT Population |
| | 14.2.3.13.1.5 | Incidence of Selected Prior Prurigo Nodularis<br>Medications | ITT Population |
| | 14.2.3.13.1.6 | Incidence of Selected Prior Prurigo Nodularis Procedures | ITT Population |
| 14.2.4 | | Pharmacokinetics | |
| | 14.2.4.1 | Summary of Nemolizumab Serum Concentrations | PK Analysis<br>Population |
| 14.2.5 | | Immunogenicity | |
| × | 14.2.5.1 | Summary of Immunogenicity - Anti-drug Antibody (ADA) and Neutralizing Antibody | PK Analysis<br>Population |
| 14.3 | | Safety Data Summary Tables | |
| 14.3.1 | | Adverse Events | |
| | 14.3.1.1.1 | Overall Summary of Treatment Emergent Adverse<br>Events (TEAEs) during Treatment Period, All<br>Causalities | Safety Population |
| 50 | 14.3.1.1.2 | Overall Summary of Treatment Emergent Adverse<br>Events (TEAEs) during Follow-up Period, All<br>Causalities | Safety Population |
| | 14.3.1.1.3 | Overall Summary of Treatment Emergent Adverse<br>Events (TEAEs) during Overall Study Period, All<br>Causalities | Safety Population |
| | 14.3.1.1.4 | Overall Summary of Treatment Emergent Adverse<br>Events (TEAEs) during Treatment Period, Study<br>Drug Related | Safety Population |
| | 14.3.1.1.5 | Overall Summary of Treatment Emergent Adverse<br>Events (TEAEs) during Follow-up Period, Study Drug<br>Related | Safety Population |
| 3 | 14.3.1.1.6 | Overall Summary of Treatment Emergent Adverse<br>Events (TEAEs) during Overall Study Period, Study<br>Drug Related | Safety Population |
| | 14.3.1.1.7 | Overall Summary of Treatment Emergent Adverse<br>Events (TEAEs) during Treatment Period, All<br>Causalities | Safety Population – Subjects with COVID-19 Infection |

| Header | Table<br>Number | Name | Analysis Set |
|---|---|---|---|
| | 14.3.1.1.8 | Overall Summary of Treatment Emergent Adverse<br>Events (TEAEs) during Follow-up Period, All<br>Causalities | Safety Population – Subjects with COVID-19 Infection |
| | 14.3.1.1.9 | Overall Summary of Treatment Emergent Adverse<br>Events (TEAEs) during Treatment Period, Study<br>Drug Related | Safety Population – Subjects with COVID-19 Infection |
| | 14.3.1.1.10 | Overall Summary of Treatment Emergent Adverse<br>Events (TEAEs) during Follow-up Period, Study Drug<br>Related | Safety Population – Subjects with COVID-19 Infection |
| | 14.3.1.1.11 | Overall Summary of Treatment Emergent Adverse<br>Events (TEAEs) during Overall Study Period by<br>Country, All Causalities | Safety Population |
| | 14.3.1.1.12 | Overall Summary of Treatment Emergent Adverse<br>Events (TEAEs) of Special Interest during Treatment<br>Period, All Causalities | Safety Population |
| | 14.3.1.1.13 | Overall Summary of Treatment Emergent Adverse<br>Events (TEAEs) of Special Interest during Follow-up<br>Period, All Causalities | Safety Population |
| | 14.3.1.1.14 | Overall Summary of Treatment Emergent Adverse<br>Events (TEAEs) of Special Interest during Treatment<br>Period, Study Drug Related | Safety Population |
| | 14.3.1.1.15 | Overall Summary of Treatment Emergent Adverse<br>Events (TEAEs) of Special Interest during Follow-up<br>Period, Study Drug Related | Safety Population |
| | 14.3.1.2.1 | Treatment Emergent Adverse Events (TEAEs) during Treatment Period by SOC and PT, All Causalities | Safety Population |
| | 14.3.1.2.2 | Treatment Emergent Adverse Events (TEAEs) during Follow-up Period by SOC and PT, All Causalities | Safety Population |
| | 14.3.1.2.3 | Treatment Emergent Adverse Events (TEAEs) during<br>Overall Study Period by SOC and PT, All Causalities | Safety Population |
| | 14.3.1.2.4 | Treatment Emergent Adverse Events (TEAEs) during<br>Treatment Period by SOC and PT, All Causalities | Safety Population – Subjects with COVID-19 Infection |
| | 14.3.1.2.5 | Treatment Emergent Adverse Events (TEAEs) during Follow-up Period by SOC and PT, All Causalities | Safety Population – Subjects with COVID-19 Infection |
| | 14.3.1.2.6 | Treatment Emergent Adverse Events (TEAEs) during<br>Overall Study Period by SOC and PT and by<br>Country, All Causalities | |
| (3)<br>(5) | 14.3.1.3.1 | Treatment Emergent Adverse Events (TEAEs) during<br>Treatment Period by SOC and PT, Study Drug<br>Related | Safety Population |
| | 14.3.1.3.2 | Treatment Emergent Adverse Events (TEAEs) during Follow-up Period by SOC and PT, Study Drug Related | Safety Population |

| Header | Table<br>Number | Name | Analysis Set |
|---|---|---|---|
| | 14.3.1.3.3 | Treatment Emergent Adverse Events (TEAEs) during<br>Overall Study Period by SOC and PT, Study Drug<br>Related | Safety Population |
| | 14.3.1.3.4 | Treatment Emergent Adverse Events (TEAEs) during Treatment Period by SOC and PT, Study Drug Related | Safety Population – Subjects with COVID-19 Infection |
| | 14.3.1.3.5 | Treatment Emergent Adverse Events (TEAEs) during Follow-up Period by SOC and PT, Study Drug Related | Safety Population – Subjects with COVID-19 Infection |
| | 14.3.1.4.1 | Exposure-Adjusted Incidence Rate for Treatment Emergent Adverse Events (TEAEs) during Treatment Period by SOC and PT, All Causalities | Safety Population |
| | 14.3.1.5.1 | Exposure-Adjusted Incidence Rate of Treatment<br>Emergent Adverse Events (TEAEs) during Treatment<br>Period by SOC and PT, Study Drug Related | Safety Population |
| | 14.3.1.6.1 | Serious Treatment Emergent Adverse Events<br>(TEAEs) during Treatment Period by SOC and PT,<br>All Causalities | Safety Population |
| | 14.3.1.6.2 | Serious Treatment Emergent Adverse Events<br>(TEAEs) during Follow-up Period by SOC and PT, All<br>Causalities | Safety Population |
| | 14.3.1.6.3 | Serious Treatment Emergent Adverse Events<br>(TEAEs) during Treatment Period by SOC and PT,<br>All Causalities | Safety Population – Subjects with COVID-19 Infection |
| | 14.3.1.6.4 | Serious Treatment Emergent Adverse Events<br>(TEAEs) during Follow-up Period by SOC and PT, All<br>Causalities | Safety Population – Subjects with COVID-19 Infection |
| | 14.3.1.7.1 | Serious Treatment Emergent Adverse Events<br>(TEAEs) during Treatment Period by SOC and PT,<br>Study Drug Related | Safety Population |
| | 14.3.1.7.2 | Serious Treatment Emergent Adverse Events<br>(TEAEs) during Follow-up Period by SOC and PT,<br>Study Drug Related | Safety Population |
| | 14.3.1.7.3 | Serious Treatment Emergent Adverse Events<br>(TEAEs) during Treatment Period by SOC and PT,<br>Study Drug Related | Safety Population – Subjects with COVID-19 Infection |
| | 14.3.1.7.4 | Serious Treatment Emergent Adverse Events<br>(TEAEs) during Follow-up Period by SOC and PT,<br>Study Drug Related | Safety Population – Subjects with COVID-19 Infection |
| | 14.3.1.8.1 | Treatment Emergent Adverse Events (TEAEs) during Treatment Period by SOC, PT and Maximum Severity, All Causalities | Safety Population |
| | 14.3.1.8.2 | Treatment Emergent Adverse Events (TEAEs) during Follow-up Period by SOC, PT and Maximum Severity, All Causalities | Safety Population |

| Header | Table<br>Number | Name | Analysis Set |
|---|---|---|---|
| | 14.3.1.9.1 | Treatment Emergent Adverse Events (TEAEs) during<br>Treatment Period by SOC, PT and Maximum<br>Severity, Study Drug Related | Safety Population |
| | 14.3.1.9.2 | Treatment Emergent Adverse Events (TEAEs) during Follow-up Period by SOC, PT and Maximum Severity, Study Drug Related | Safety Population |
| | 14.3.1.10.1 | Severe Treatment Emergent Adverse Events (TEAEs) during Treatment Period by SOC and PT, All Causalities | Safety Population |
| | 14.3.1.10.2 | Severe Treatment Emergent Adverse Events<br>(TEAEs) during Follow-up Period by SOC and PT, All<br>Causalities | Safety Population |
| | 14.3.1.11.1 | Severe Treatment Emergent Adverse Events<br>(TEAEs) during Treatment Period by SOC and PT,<br>Study Drug Related | Safety Population |
| | 14.3.1.11.2 | Severe Treatment Emergent Adverse Events<br>(TEAEs) during Follow-up Period by SOC and PT,<br>Study Drug Related | Safety Population |
| | 14.3.1.12.1 | Treatment Emergent Adverse Events (TEAEs) Leading to Study Drug Withdrawal during Treatment Period by SOC and PT, All Causalities | Safety Population |
| 25 | 14.3.1.13.1 | Treatment Emergent Adverse Events (TEAEs) Leading to Study Drug Withdrawal during Treatment Period by SOC and PT, Study Drug Related | Safety Population |
| | 14.3.1.14.1 | Treatment Emergent Adverse Events (TEAEs) Leading to Study Discontinuation during Treatment Period by SOC and PT, All Causalities | Safety Population |
| | 14.3.1.14.2 | Treatment Emergent Adverse Events (TEAEs) Leading to Study Discontinuation during Follow-up Period by SOC and PT, All Causalities | Safety Population |
| | 14.3.1.15.1 | Treatment Emergent Adverse Events (TEAEs) Leading to Study Discontinuation during Treatment Period by SOC and PT, Study Drug Related | Safety Population |
| e e | 14.3.1.15.2 | Treatment Emergent Adverse Events (TEAEs) Leading to Study Discontinuation during Follow-up Period by SOC and PT, Study Drug Related | Safety Population |
| | 14.3.1.16.1 | Treatment Emergent Adverse Events (TEAEs) of<br>Special Interest during Treatment Period by<br>Category, SOC and PT, All Causalities | Safety Population |
| | 14.3.1.16.2 | Treatment Emergent Adverse Events (TEAEs) of<br>Special Interest during Follow-up Period by<br>Category, SOC and PT, All Causalities | Safety Population |
| | 14.3.1.16.3 | Treatment Emergent Adverse Events (TEAEs) of<br>Special Interest during Treatment Period by<br>Category, SOC and PT | Safety Population – Subjects with COVID-19 Infection |
| | 14.3.1.16.4 | Treatment Emergent Adverse Events (TEAEs) of Special Interest during Follow-up Period by Category, SOC and PT | Safety Population – Subjects with COVID-19 Infection |

| Header | Table<br>Number | Name | Analysis Set |
|---|---|---|---|
| | 14.3.1.17.1 | Treatment Emergent Adverse Events (TEAEs) of<br>Special Interest during Treatment Period by<br>Category, SOC and PT, Study Drug Related | Safety Population |
| | 14.3.1.17.2 | Treatment Emergent Adverse Events (TEAEs) of<br>Special Interest during Follow-up Period by<br>Category, SOC and PT, Study Drug Related | Safety Population |
| | 14.3.1.17.3 | Treatment Emergent Adverse Events (TEAEs) of<br>Special Interest during Treatment Period by<br>Category, SOC and PT, Study Drug Related | Safety Population – Subjects with COVID-19 Infection |
| | 14.3.1.17.4 | Treatment Emergent Adverse Events (TEAEs) of Special Interest during Follow-up Period by Category, SOC and PT, Study Drug Related | Safety Population – Subjects with COVID-19 Infection |
| | 14.3.1.18.1 | Treatment Emergent Adverse Events (TEAEs) Occurred in PT > 5% of Subjects during Treatment Period by SOC and PT, All Causalities | Safety Population |
| | 14.3.1.18.2 | Treatment Emergent Adverse Events (TEAEs) Occurred in PT > 5% of Subjects during Follow-up Period by SOC and PT, All Causalities | Safety Population |
| 38<br>50 | 14.3.1.18.3 | Treatment Emergent Adverse Events (TEAEs) Occurred in PT > 5% of Subjects during Treatment Period by PT, All Causalities | Safety Population |
| | 14.3.1.18.4 | Treatment Emergent Adverse Events (TEAEs) Occurred in PT > 5% of Subjects during Follow-up Period by PT, All Causalities | Safety Population |
| 58 | 14.3.1.19.1 | Treatment Emergent Adverse Events (TEAEs) Occurred in PT > 5% of Subjects during Treatment Period by SOC and PT, Study Drug Related | Safety Population |
| | 14.3.1.19.2 | Treatment Emergent Adverse Events (TEAEs) Occurred in PT > 5% of Subjects during Follow-up Period by SOC and PT, Study Drug Related | Safety Population |
| | 14.3.1.19.3 | Treatment Emergent Adverse Events (TEAEs) Occurred in PT > 5% of Subjects during Treatment Period by PT, Study Drug Related | Safety Population |
| | 14.3.1.19.4 | Treatment Emergent Adverse Events (TEAEs) Occurred in PT > 5% of Subjects during Follow-up Period by PT, Study Drug Related | Safety Population |
| | 14.3.1.20.1 | Adjudicated Treatment Emergent Adverse Events (TEAEs) during Treatment Period by SOC and PT, All Causalities | Safety Population |
| | 14.3.1.20.2 | Adjudicated Treatment Emergent Adverse Events (TEAEs) during Follow-up Period by SOC and PT, All Causalities | Safety Population |
| | 14.3.1.21.1 | Adjudicated Treatment Emergent Adverse Events (TEAEs) during Treatment Period by SOC and PT, Study Drug Related | Safety Population |
| | 14.3.1.21.2 | Adjudicated Treatment Emergent Adverse Events (TEAEs) during Follow-up Period by SOC and PT, Study Drug Related | Safety Population |

| Header | Table<br>Number | Name | Analysis Set |
|---|---|---|---|
| | 14.3.1.22.1 | Treatment Emergent Adverse Events (TEAEs) of<br>Asthma and AESI reported by Investigator with<br>Adjudication Outcome during Treatment Period by<br>IAC, All Causalities | Safety Population |
| | 14.3.1.22.2 | Treatment Emergent Adverse Events (TEAEs) of<br>Asthma and AESI reported by Investigator with<br>Adjudication Outcome during Follow-up Period by<br>IAC, All Caualities | Safety Population |
| | 14.3.1.23.1 | Treatment Emergent Adverse Events (TEAEs) of<br>Asthma and AESI reported by Investigator with<br>Adjudication Outcome during Treatment Period by<br>IAC, Study Drug Related | Safety Population |
| | 14.3.1.23.2 | Treatment Emergent Adverse Events (TEAEs) of<br>Asthma and AESI reported by Investigator with<br>Adjudication Outcome during Treatment Period by<br>IAC, Study Drug Related | Safety Population |
| | 14.3.1.24.1 | Confirmed Adjudicated Treatment Emergent Adverse<br>Events (TEAEs) during Treatment Period by SOC,<br>PT and Maximum Severity, All Causalities | Safety Population |
| 10 | 14.3.1.24.2 | Confirmed Adjudicated Treatment Emergent Adverse<br>Events (TEAEs) during Follow-up Period by SOC, PT<br>and Maximum Severity, All Causalities | Safety Population |
| | 14.3.1.25.1 | Confirmed Adjudicated Treatment Emergent Adverse Events (TEAEs) during Treatment Period by SOC, PT and Maximum Severity, Study Drug Related | Safety Population |
| | 14.3.1.25.2 | Confirmed Adjudicated Treatment Emergent Adverse<br>Events (TEAEs) during Follow-up Period by SOC, PT<br>and Maximum Severity, Study Drug Related | Safety Population |
| | 14.3.1.26.1 | Treatment Emergent Adverse Events (TEAEs) of<br>Special Interest during Treatment Period by<br>Category, SOC, PT and Maximum Severity, All<br>Causalities | Safety Population |
| | 14.3.1.26.2 | Treatment Emergent Adverse Events (TEAEs) of<br>Special Interest during Follow-up Period by<br>Category, SOC, PT and Maximum Severity, All<br>Causalities | Safety Population |
| | 14.3.1.27.1 | Treatment Emergent Adverse Events (TEAEs) of<br>Special Interest during Treatment Period by<br>Category, SOC, PT and Maximum Severity, Study<br>Drug Related | Safety Population |
| | 14.3.1.27.2 | Treatment Emergent Adverse Events (TEAEs) of<br>Special Interest during Follow-up Period by<br>Category, SOC, PT and Maximum Severity, Study<br>Drug Related | Safety Population |
| 14.3.2 | | Listings of Deaths, Other Serious and Significant Adverse Events | |
| | 14.3.2.1 | Listing of Serious Treatment Emergent Adverse Events (TEAEs) | Safety Population |
| | 14.3.2.2 | Listing of Severe Treatment Emergent Adverse Events (TEAEs) | Safety Population |
| | 14.3.2.3 | Listing of Treatment Emergent Adverse Events (TEAEs) Leading to Study Discontinuation | Safety Population |

| Header | Table<br>Number | Name | Analysis Set |
|---|---|---|---|
| | 14.3.2.4 | Listing of Treatment Emergent Adverse Events (TEAEs) of Special Interest | Safety Population |
| | 14.3.2.5 | Listing of Treatment Emergent Adverse Events (TEAEs) Leading to Death | Safety Population |
| 14.3.3 | | Narratives of Deaths, Other Serious and Certain<br>Other Significant Adverse Events | |
| 14.3.4 | | Laboratory Value | |
| 14.3.4.1 | | Clinical Laboratory Data | |
| 14.3.4.1.1 | | Hematology Data | |
| | 14.3.4.1.1.1 | Summary of Laboratory Data for Hematology | Safety Population |
| | 14.3.4.1.1.2 | Shift from Baseline for Hematology by Reference Ranges | Safety Population |
| | 14.3.4.1.1.3 | Summary of Potentially Clinically Significant<br>Hematology | Safety Population |
| | 14.3.4.1.1.4 | Listing of Subjects with Abnormal Hematology<br>Results | Safety Population |
| | 14.3.4.1.1.5 | Listing of Subjects with Potentially Clinically Significant Hematology Results | Safety Population |
| 14.3.4.1.2 | | Blood Chemistry Data | |
| | 14.3.4.1.2.1 | Summary of Laboratory Data for Clinical Chemistry | Safety Population |
| | 14.3.4.1.2.2 | Shift from Baseline for Clinical Chemistry by Reference Range | Safety Population |
| | 14.3.4.1.2.3 | Summary of Potentially Clinically Significant Clinical Chemistry | Safety Population |
| | 14.3.4.1.2.4 | Listing of Subjects with Abnormal Clinical Chemistry Results | Safety Population |
| | 14.3.4.1.2.5 | Listing of Subjects with Potentially Clinically Significant Clinical Chemistry Results | Safety Population |
| 14.3.4.1.3 | | Urinalysis Data | |
| | 14.3.4.1.3.1 | Summary of Laboratory Data for Urinalysis | Safety Population |
| 14.3.4.1.4 | | Pregnancy Test | |
| | 14.3.4.1.4.1 | Summary of Pregnancy Test Results by Visit | Safety Population |
| 14.3.4.2 | | Vital Signs | , |
| | 14.3.4.2.1 | Summary of Vital Signs, Height and Weight | Safety Population |
| | 14.3.4.2.2 | Proportions of Subjects with Potentially Clinically Significant Vital Signs and Weight | Safety Population |
| | 14.3.4.2.3 | Listing of Subjects with Potentially Clinically Significant Vital Signs and Weight | Safety Population |
| 14.3.4.3 | | Electrocardiogram (ECG) Data | |
| | 14.3.4.3.1 | Summary of Observed Values and Changes from Baseline for Electrocardiogram (ECG) Parameters by Visit | Safety Population |
| 33 | 14.3.4.3.2 | Summary of Electrocardiogram (ECG) Interpretation | Safety Population |
| | 14.3.4.3.3 | Summary of Electrocardiogram (ECG) Findings by Visit | Safety Population |
| 14.3.4.4 | | Other Safety | |
| | 14.3.4.4.1 | Summary of Physical Examination | Safety Population |
| | 14.3.4.4.2 | Shift from Baseline in Physical Examination | Safety Population |
| | 14.3.4.4.3 | Listing of Subjects with Abnormal Results in Physical Examination | Safety Population |

| Header | Table<br>Number | Name | Analysis Set |
|---|---|---|---|
| 10 | 14.3.4.4.4 | Summary of Respiratory Assessments – Peak<br>Expiratory Flow (PEF) | Safety Population |
| | 14.3.4.4.5 | Summary of Respiratory Assessments – Peak<br>Expiratory Flow (PEF) for Subjects with Asthma<br>History | Safety Population |
| | 14.3.4.4.6 | Summary of Respiratory Assessments – Peak<br>Expiratory Flow (PEF) for Subjects without Asthma<br>History | Safety Population |
| | 14.3.4.4.7 | Summary of Peak Expiratory Flow (PEF) < 80% of<br>Predicted Value | Safety Population |
| | 14.3.4.4.8 | Summary of Peak Expiratory Flow (PEF) < 80% of<br>Predicted Value for Subjects with Asthma History | Safety Population |
| 38 | 14.3.4.4.9 | Summary of Peak Expiratory Flow (PEF) < 80% of<br>Predicted Value for Subjects without Asthma History | Safety Population |
| 18 | 14.3.4.4.10 | Safety Population | |
| | 14.3.4.4.11 | Safety Population | |
| | 14.3.4.4.12 | Summary of Respiratory Examination | Safety Population |

#### **Index of Figures** 19.

This section contains lists of the figures tentatively planned for this study. Changes in the number or content of planned listings are not considered deviations from this SAP.

| Figure<br>Number | Name | Analysis Set (Examples) |
|---|---|---|
| 14.1.1.7 | Time (days) to Permanent Discontinuation of Study Drug by Reason for Discontinuation | ITT Population |
| 14.2.1.1.2 | Bar Chart of Proportion of Subjects with an Improvement of >= 4 from Baseline in Weekly Average PP NRS at Week 16 - Missing as Non-Responder | ITT Population |
| 14.2.1.1.4 | Bar Chart of Proportion of Subjects with an Improvement of >= 4 from Baseline in Weekly Average PP NRS at Week 16 - Missing as Non-Responder | PP Population |
| 14.2.1.1.6 | Sensitivity Analysis of Proportion of Subjects with an Improvement of >= 4 from Baseline in Weekly Average PP NRS at Week 16 - Tipping Point Analysis | ITT Population |
| 14.2.1.1.12 | Subgroup Analysis of Proportion of Subjects with an Improvement of >= 4 from Baseline in Weekly Average PP NRS at Week 16 with Forest Plot – Missing as Non-Responder | ITT Population |
| 14.2.1.2.2 | Bar Chart of Proportion of Subjects with an IGA Success at Week 16 - Missing as Non-Responder | ITT Population |
| 14.2.1.2.4 | Bar Chart of Proportion of Subjects with an IGA Success at Week 16 - Missing as Non-Responder | PP Population |
| 14.2.1.2.6 | Sensitivity Analysis of Proportion of Subjects with an IGA Success at Week 16 - Tipping Point Analysis | ITT Population |
| 14.2.1.2.12 | Subgroup Analysis of Proportion of Subjects with an IGA Success at Week 16 with Forest Plot – Missing as Non-Responder | ITT Population |
| 14.2.2.1.2 | Bar Chart of Proportion of Subjects with an Improvement of >= 4 from Baseline in Weekly Average PP NRS at Week 4 - Missing as Non-Responder | ITT Population |
| 14.2.2.1.4 | Bar Chart of Proportion of Subjects with an Improvement of >= 4 from Baseline in Weekly Average PP NRS at Week 4 - Missing as Non-Responder | PP Population |
| 14.2.2.1.6 | Sensitivity Analysis of Proportion of Subjects with an Improvement of >= 4 from Baseline in Weekly Average PP NRS at Week 4 - Tipping Point Analysis | ITT Population |
| 14.2.2.1.12 | Subgroup Analysis of Proportion of Subjects with an Improvement of >= 4 from Baseline in Weekly Average PP NRS at Week 4 with Forest Plot – Missing as Non-Responder | ITT Population |
| 14.2.2.2.2 | Bar Chart of Proportion of Subjects with Weekly Average PP NRS < 2 at Weeks 4 and 16 - Missing as Non-Responder | ITT Population |
| 14.2.2.2.4 | Bar Chart of Proportion of Subjects with Weekly Average PP NRS < PP Population 2 at Weeks 4 and 16 - Missing as Non-Responder | |
| 14.2.2.2.6 | Sensitivity Analysis of Proportion of Subjects with Weekly Average PP NRS < 2 at Weeks 4 and 16 - Tipping Point Analysis | |
| 14.2.2.2.12 | Subgroup Analysis of Proportion of Subjects with Weekly Average PP NRS < 2 at Weeks 4 and 16 with Forest Plot – Missing as Non-Responder | ITT Population |
| 14.2.2.3.2 | Bar Chart of Proportion of Subjects with an Improvement >= 4 from Baseline in Weekly Average SD NRS at Week 4 and Week 16 - Missing as Non-Responder | ITT Population |

| Figure<br>Number | Name | Analysis Set (Examples) |
|---|---|---|
| 14.2.2.3.4 | Bar Chart of Proportion of Subjects with an Improvement >= 4 from Baseline in Weekly Average SD NRS at Week 4 and Week 16 - Missing as Non-Responder | PP Population |
| 14.2.2.3.6 | Sensitivity Analysis of Proportion of Subjects with an Improvement >= 4 from Baseline in Weekly Average SD NRS at Week 4 and Week 16 - Tipping Point Analysis | ITT Population |
| 14.2.2.3.12 | Subgroup Analysis of Proportion of Subjects with an Improvement >= 4 from Baseline in Weekly Average SD NRS at Week 4 and Week 16 with Forest Plot – Missing as Non-Responder | ITT Population |
| 14.2.3.1.5 | Line Plot of Proportion of Subjects with IGA Success – Missing as Non-Responder | ITT Population |
| 14.2.3.1.7 | Line Plot of Proportion of Subjects with IGA Success – Missing as Non-Responder | PP Population |
| 14.2.3.3.5 | Line Plot of Proportion of Subjects with Weekly Average PP NRS Improvement >= 4 - Missing as Non-Responder | ITT Population |
| 14.2.3.3.6 | Line Plot of Proportion of Subjects with Weekly Average PP NRS<br>Improvement >= 4 - Missing as Non-Responder | PP Population |
| 14.2.3.3.8 | Line Plot of Proportion of Subjects with Weekly Average PP NRS < 2 - Missing as Non-Responder | ITT Population |
| 14.2.3.3.9 | Line Plot of Proportion of Subjects with Weekly Average PP NRS < 2 - Missing as Non-Responder | PP Population |
| 14.2.3.3.19 | Line Plot of Change from Baseline in PP NRS - OC | PP Population |
| 14.2.3.3.20 | Line Plot of Percentage Change from Baseline in Weekly Average PP NRS by Visit - OC | ITT Population |
| 14.2.3.5.4 | Line Plot of Proportion of Subjects with Weekly Average SD NRS Improvement >= 4 - Missing as Non-Responder | ITT Population |
| 14.2.3.10.4 | Line Plot of Proportion of Subjects with DLQI Improvement >= 4 - Missing as Non-Responder | ITT Population |
| 14.2.3.13.1.4 | Kaplan Meier Curve for Time to First Rescue Therapy | ITT Population |
| 14.2.4.2 | Mean Nemolizumab Time-Concentration Profiles | PK Analysis Population |
| 14.2.4.3 | Individual Time-Concentration Profiles | PK Analysis<br>Population |
| 14.3.4.1.1.6 | Distribution of Hematology Laboratory Parameters by Visit with Maximum Post-Baseline Values Safety Population | |
| 14.3.4.1.2.6 | Distribution of Chemistry Laboratory Parameters by Visit with Maximum Post-Baseline Values Po | |
| 14.3.4.1.2.7 | Individual Subject Plots of Abnormal Chemistry Laboratory Parameters of Special Interest by Visit | Safety<br>Population |
| 14.3.4.2.4 | Distribution of Vital Signs by Visit with Maximum Post-baseline Values | Safety<br>Population |

#### **Index of Listings** 20.

This section contains lists of the listings tentatively planned for this study. Changes in the number or content of planned listings are not considered deviations from this SAP.

| Header Listing Number | | | |
|---|---|---|---|
| 16.2 | | Subject Data Listings | |
| 16.2.1 | | Discontinued Subjects | |
| | 16.2.1.1 | Randomization | ITT Population |
| | 16.2.1.2 | Study Completion Status | ITT Population |
| | 16.2.1.3 | Screen Failures | Screened Subjects |
| | 16.2.1.4 | Study Drug Completion Status | ITT Population |
| | 16.2.1.5 | Visit Dates | ITT Population |
| | 16.2.1.6 | Missing Assessment due to COVID-19 | ITT Population |
| 16.2.2 | | Protocol Deviations | |
| | 16.2.2.1 | Protocol Deviations | ITT Population |
| | 16.2.2.2 | Protocol Deviations Related to COVID-19 | ITT Population |
| 16.2.3 | | Subjects Excluded from Analysis Populations | |
| | 16.2.3.1 | Subjects in Analysis Populations | ITT Population |
| | 16.2.3.2 | Inclusion and Exclusion Criteria Not Met | Screened Subjects |
| 16.2.4 | 0.0000000000000000000000000000000000000 | Demographic Data | |
| | 16.2.4.1 | Demographics and Baseline Characteristics | ITT Population |
| | 16.2.4.2 | Baseline Disease Characteristics | |
| | 16.2.4.3 | Medical History | ITT Population |
| | 16.2.4.4 | Medical and Surgical Procedures | ITT Population |
| | 16.2.4.5 | Rescue Medical and Surgical Procedures | ITT Population |
| | 16.2.4.6 | Prior and Concomitant Medications | ITT Population |
| | 16.2.4.7 | Rescue Medications | ITT Population |
| | 16.2.4.8 | Subjects with Difference between<br>Randomization Stratification and Actual<br>Stratification | ITT Population |
| 16.2.5 | Î | Compliance and Exposure Information | |
| 8 | 16.2.5.1 | Study Drug Dispensation | Safety Population |
| 8 | 16.2.5.2 | Study Drug Administration | Safety Population |
| 8 | 16.2.5.3 | Study Drug Compliance | Safety Population |
| 16.2.6 | Î | Individual Efficacy Response Data | |
| 18 | 16.2.6.1 | Pruritus Numeric Rating Scale | ITT Population |
| 18 | 16.2.6.2 | Investigator's Global Assessment (IGA) | ITT Population |
| js. | 16.2.6.3 | Prurigo Activity Score (PAS) | ITT Population |
| js. | 16.2.6.4 | Sleep Disturbance NRS | ITT Population |
| is . | 16.2.6.5.1 | Subject Sleep Diary | ITT Population |
| 8 | 16.2.6.5.2 | Weekly Average Sleep Diary Metrics | ITT Population |
| | 16.2.6.6 | PN Associated Pain Intensity and Frequency | ITT Population |
| | 16.2.6.7 | Patient Global Assessment of Disease (PGAD) | ITT Population |
| | 16.2.6.8 | Patient Global Assessment of Treatment (PGAT) | ITT Population |
| | 16.2.6.9 | Dermatology Life Quality Index (DLQI) | ITT Population |

| Header | Listing<br>Number | Name | Analysis Set |
|---|---|---|---|
| 2 | 16.2.6.10 | Hospital Anxiety and Depression Scale (HADS) | ITT Population |
| | 16.2.6.11 | EuroQoL 5 Dimension Instrument (EQ5D) | ITT Population |
| | 16.2.6.12 | Nemolizumab Serum Concentrations Population | PK Analysis |
| | 16.2.6.13 | Immunogenicity - Anti-drug Antibody (ADA) and Neutralizing Antibodies | PK Analysis |
| 16.2.7 | | Adverse Event Listings | |
| | 16.2.7.1 | Treatment Emergent Adverse Events (TEAE) | Safety Population |
| | 16.2.7.2 | Pre-Treatment Adverse Events | Safety Population |
| | 16.2.7.3 | Treatment Emergent Adverse Events (TEAE) | Safety Population –<br>Subjects with COVID-<br>19 Infection |
| 55<br>56 | 16.2.7.4 | Treatment Emergent Adverse Events (TEAE) Comments | Safety Population |
| | 16.2.7.5 | Adjudicated Asthma Adverse Events | Safety Population |
| | 16.2.7.6 | Adjudicate Asthma Adverse Events Comments by Independent Adjudication Committee | Safety Population |
| 16.2.8 | | Listing of Individual Laboratory<br>Measurements by Subject | |
| 16.2.8.1 | | Clinical Laboratory Data | |
| | 16.2.8.1.1 | Laboratory Data - Hematology | Safety Population |
| | 16.2.8.1.2 | Laboratory Data – Clinical Chemistry | Safety Population |
| | 16.2.8.1.3 | Laboratory Data - Urinalysis | Safety Population |
| | 16.2.8.1.4 | Childbearing Potential and Premenses<br>Status | Safety Population |
| | 16.2.8.1.5 | Pregnancy Test Results | Safety Population |
| | 16.2.8.1.6 | Tuberculosis Test Results | Safety Population |
| | 16.2.8.1.7 | Virology and Genomics | Safety Population |
| | 16.2.8.1.8 | Immunoglobulin E | Safety Population |
| 16.2.8.2 | | Other Safety Data | MO 446 |
| | 16.2.8.2.1 | Vital Signs, Height and Weight | Safety Population |
| | 16.2.8.2.2 | Electrocardiogram (ECG) | Safety Population |
| | 16.2.8.2.3 | Physical Examination | Safety Population |
| | 16.2.8.2.4 | Respiratory Assessement – Medical<br>Interview | Safety Population |
| | 16.2.8.2.5 | Respiratory Assessment – Peak Expiratory Flow (PEF) | Safety Population |
| d. | 16.2.8.2.6 | Known Asthma, Wheeze, Dyspnea and Cough Triggers | Safety Population |
| 4 | 16.2.8.2.7 | Asthma Control Test (ACT) | Safety Population |
| 74 | 16.2.8.2.8 | Subjects with a drop by >= 15% from<br>Baseline for either PEF or ACT | Safety Population |

### 21. Appendices

#### 21.1. Tipping Point Analysis

Tipping point analysis will be performed by converting non-responders due to missing data to responders in successive increments ( $\Delta$ ) for both treatment groups to assess the robustness of analysis (Liublinska, 2015, see Section 15). The value of  $\Delta$  that overturns (i.e. non-significant) the primary results will represent the tipping point. A graphic display of all possible combination of the number of responders among both treatment groups will be presented.

#### 21.2. Multiple Imputation

Multiple imputation (MI) methods will be done for monotone missing data. The MI imputation will be carried out as follows.

#### 21.2.1. Imputation Phase

50 imputed datasets with a monotone missing pattern will be created using SAS MI procedure based on the observed data (Markov-Chain-Monte-Carlo method, MCMC). The seed to be used is 203065 (the Protocol number). Pattern of missing data will be evaluated and it is expected that the pattern of missing data will be monotonic. For non-monotone missing data patterns, MCMC method of MI procedure will be used to impute enough data so that the remaining missing data is monotone.

Each of the imputed datasets will be used to generate 50 complete datasets, using following approaches:

- Binary endpoint: A logistic regression method to impute the ordinal missing data, including treatment, randomization strata, and assessments from earlier time points as covariates. Response or total score of the subjects will be derived using these imputed data.
- Continuous endpoint: A linear regression model including treatment, randomization strata, and
  assessments from earlier time points as covariates will be used to impute the score. Response or
  total score of the subjects will be derived using these imputed data.

#### 21.2.2. Analysis Phase

The analysis will be conducted using the complete datasets.

- Binary endpoint: The complete datasets will be modelled for the endpoint using CMH method. Proportion of responders in each treatment arm, difference and standard error will be calculated.
- Continuous endpoint: The complete datasets will be analyzed using ANCOVA including treatment group and randomization stratification factors as factors and appropriate Baseline values as a covariate, if applicable. LSMeans in each treatment arm, difference and standard errors will be calculated.

#### 21.2.3. Pooling Phase

The results from the analysis phase will be combined as follows.

 Binary endpoint: The results from the CMH analysis of the multiple imputed datasets will be combined to produce pooled CMH statistics and p-value. Proportion of responders in each treatment arm, difference and standard error will be combined using the MIANALYZE procedure in SAS.  Continuous endpoint: The LSMeans in each treatment arm, difference and standard errors from the ANCOVA of the multiple imputed datasets will be combined using the MIANALYZE procedure in SAS.

#### 21.3. Example SAS Code

```
1. The example SAS code for CMH model is listed as below:
proc freq data=analysis data;
  tables stratum*trt*resp/ cmh alpha=0.1;
run;
2. The example SAS code for MMRM model is listed as below:
proc mixed data = analysis_data;
  class stratum trtp avisit subjid;
 model chg = base stratum trtp avisit trtp*avisit/ ddfm=kr;
  repeated avisit / subject=subjid(trtp) type=un;
 Ismeans trtp/ cl diff;
 Ismeans trtp*avisit/ slice=avisit cl diff;
run;
3. The example SAS code for ANCOVA model is listed as below:
proc mixed data = analysis data;
  class stratum trtp;
 model chg = base stratum trtp;
 Ismeans trtp/ cl diff;
run;
4. The example SAS code for imputation phase by PROC MI:
proc mi data=analysis data seed=203065 minimum=xx maximum=xx nimpute=50 out=out data;
  mcmc impute=monotone chain = multiple;
  var base stratum y4 y8 y12 y16;
run;
proc mi data = analysis data seed=203065 minimum=xx maximum=xx nimpute=number of imputations
out=out data;
  by imputation;
  class trtp stratum;
  monotone reg (/details); [OR montone logistic;]
 mnar model (y4 / modelobs = (trtp = 'Placebo'));
 mnar model (y8 / modelobs = (trtp = 'Placebo'));
 mnar model (y12 / modelobs = (trtp = 'Placebo'));
 mnar model (y16 / modelobs = (trtp = 'Placebo'));
  var base stratum y4 y8 y12 y16;
```

5. The example SAS code for pooling phase for ANCOVA model by PROC MIANALYZE:

This document is confidential.

run;


```
proc sort data=diff;
  by avisitn trtp;
run;
proc sort data=Ism;
  by avisitn trtp;
run;
proc mianalyze data=diff;
  by avisitn trtp;
  modeleffects estimate;
  stderr stderr;
ods output ParameterEstimates=estdiff; run;
proc mianalyze data=lsm;
  by avisitn trtp;
  modeleffects estimate;
  stderr stderr;
ods output ParameterEstimates=estlsm; run;
```

Filing requirements: TMF

## 21.4. Potentially Clinically Significant Ranges

Potentially clinically significant ranges for Hematology parameters are defined in Table 21-1.

Table 21-1: Potentially Clinically Significant Ranges for Hematology Parameters

| Test Parameter | Test<br>Parameter<br>Code | Normal Range Lower<br>Limit (LLN) | Normal Range Upper<br>Limit (ULN) | Potentially Clinically Significant Ranges |
|---|---|---|---|---|
| Basophils (x10 <sup>9</sup> /L) | BASO | 0.00 | 0.20 | > 0.2 at post-baseline, if baseline value ≤ 0.2 |
| Eosinophils (x10^9/L) | EOS | 0.00 | 0.57 | > 0.7 at post-baseline, if baseline value ≤ 0.7 |
| | | 80 (≥59 years old) | 100 (≥59 years old) | > 105 at post-baseline, if baseline value ≤ 105 |
| Hematocrit (L/L) | HCT | 0.39 (12-<59 years old, Male) | 0.54 (12-<59 years old, Male) | < 0.30 at post-baseline, if baseline value ≥ 0.30 |
| | | 0.37 (≥ 59 years old,<br>Male) | 0.51 (≥ 59 years old, Male) | > 0.6 at post-baseline, if baseline value ≤ 0.6 |
| | | 0.34 (Female) | 158.00 (Female) | |
| Hemoglobin (g/L) | HGB | 127 (12-<59 years old, Male) | 181 (12-<59 years old, Male) | Male < 100 at post-baseline, if baseline value ≥ 100 |
| | | 116 (12-<59 years old, Female) | 164 (12-<59 years old, Female) | Male ≥ 200 at post-baseline, if baseline value < 200 |
| | | 125 (≥ 59 years old,<br>Male) | 170 (≥ 59 years old,<br>Male) | Female <90 g/L at post-baseline and ≥ 90 g/L at baseline |
| | | 115 (≥ 59 years old,<br>Female) | 158 (≥ 59 years old,<br>Female) | Female ≥180 g/L at post-baseline and < 180 g/L at baseline |
| Leukocytes (x10^9/L) | WBC | 3.80 | 10.70 | < 3.0 at post-baseline, if baseline value ≥ 3.0 |
| | | | | > 15.0 at post-baseline, if baseline value ≤ 15.0 |
| Lymphocytes (x10^9/L) | LYM | 0.91 (18 – <59 years old) | 4.28 (18 – <59 years old) | < 0.8 at post-baseline, if baseline value ≥ 0.8 |
| | | 0.80 (≥ 59 years old) | 3 (≥ 59 years old) | > 4.28 at post-baseline, if baseline value ≤ 4.28 (age 18 - < 59); > 3.00 at post-baseline, if baseline value ≤ 3.00 (age ≥ 59) |
| Monocytes (x10^9/L) | MONO | 0.12 | 0.92 | > 0.92 at post-baseline, if baseline value ≤ 0.92 |
| Neutrophils,<br>Segmented (GI/L) | NEUTSG | 1.96 | 7.23 | < 1.5 at post-baseline, if baseline value is ≥ 1.5 |
| | | | | > 9 at post-baseline, if baseline value is ≤ 9 |
| Platelets (x10^9/L) | PLAT | 140 (18 - <60 years old) | 400 (18 - <60 years old) | < 100 at post-baseline, if baseline value ≥ 100 |

| 130 (≥ 60 years old) | 394 (≥ 60 years old) | > 700 at post-baseline, if baseline value ≤ 700 |
|---|---|---|

Potentially clinically significant ranges for Blood Chemistry parameters are defined in Table 21-2.

Table 21-2: Potentially Clinically Significant Ranges for Blood Chemistry Parameters

| Test Parameter | Test<br>Parameter<br>Code | Normal Range Lower<br>Limit (LLN) | Normal Range Upper<br>Limit (ULN) | Potentially Clinically Significant Ranges |
|---|---|---|---|---|
| Aspartate Aminotransferase (U/L) | AST | 8.00 | 40.00 | > 3 x ULN at post-baseline, if baseline value ≤ 3 x ULN |
| Alkaline Phosphatase (U/L) | ALP | 55 (< 19 years old,<br>Male) | 149 (< 19 years old,<br>Male) | > 2.5 x ULN at post-baseline, if baseline value ≤ 2.5 x ULN |
| | | 45 (< 19 years old,<br>Female) | 87 (< 19 years old, Female) | |
| | | 40 (≥ 19 years old,<br>Male) | 129(≥ 19 years old,<br>Male) | |
| | | 35 (≥ 19 years old,<br>Female) | 104 (≥ 19 years old,<br>Female) | |
| Alanine<br>Aminotransferase (U/L) | ALT | 5 (Male) | 48 (Male) | > 3 x ULN at post-baseline, if baseline value ≤ 3 x ULN |
| | | 4 (Female) | 43 (Female) | |
| Bilirubin (umol/L) | BILI | 3.00 | 21.00 | > 1.5 x ULN at post-baseline, if baseline value ≤ 1.5 * ULN |
| Calcium (mmol/L) | CA | 2.07 | 2.64 | < 2 at post-baseline, if baseline value ≥ 2 |
| | | | | > 2.9 at post-baseline, if baseline value ≤ 2.9 |
| Chloride (mmol/L) | CL | 94.00 | 112.00 | < 94 at post-baseline, if baseline value ≥ 94 |
| | | | | > 115 at post-baseline, if baseline value ≤ 115 |
| Cholesterol (mmol/L) | CHOL | 2.95 (< 20 years old,<br>Male) | 5.12 (< 20 years old,<br>Male) | > 7.75 at post-baseline, if baseline value ≤ 7.75 (Female ≤ 60 years old, Male ≤ 70 years old); > 8.28 at post-baseline, if baseline value ≤ 8.28 (Female < 60 - 70 years old); > 7.76 at post-baseline, if baseline value ≤ 7.76 (Male > 70 years old); > 9.10 at post-baseline, if baseline value ≤ 9.10 (Female > 70 years old) |

| Test Parameter | Test<br>Parameter<br>Code | Normal Range Lower<br>Limit (LLN) | Normal Range Upper<br>Limit (ULN) | Potentially Clinically Significant Ranges |
|---|---|---|---|---|
| | | 3.23 (< 20 years old, | 5.48 (< 20 years old, | |
| | | Female) | Female) | |
| | | 3.31 (20 - < 30 years | 6.10 (20 - < 30 years | |
| | | old, Male) | old, Male) | |
| | | 3.31 (20 - < 30 years | 5.64 (20 - < 30 years | |
| | | old, Female) | old, Female) | |
| | | 3.88 (30 - < 40 years | 6.83 (30 - < 40 years | |
| | | old, Male) | old, Male) | |
| | | 3.65 (30 - < 40 years | 6.21 (30 - < 40 years | |
| | | old, Female) | old, Female) | |
| | | 4.19 (40 - < 50 years | 7.24 (40 - < 50 years | |
| | | old, Male) | old, Male) | |
| | | 4.01 (40 - < 50 years | 6.85 (40 - < 50 years | |
| | | old, Female) | old, Female) | |
| | | 4.40 (50 - < 60 years | 7.53 (50 - < 60 years | |
| | | old, Male) | old, Male) | |
| | | 4.42 (50 - < 60 years | 7.53 (50 - < 60 years | |
| | | old, Female) | old, Female) | |
| | | 4.53 (60 - < 70 years | 7.71 (60 - < 70 years | |
| | | old, Male) | old, Male) | |
| | | 4.86 (60 - < 70 years | 8.28 (60 - < 70 years | |
| | | old, Female) | old, Female) | |
| | | 4.58 (≥ 70 years old, | 7.76 (≥ 70 years old, | |
| | | Male) | Male) | |
| | | 5.35 (≥ 70 years old, | 9.10 (≥ 70 years old, | |
| | | Female) | Female) | |
| Creatinine (umol/L) | CREAT | 40 (18 - < 50 years | 110 (18 - < 50 years | > 1.5 x ULN at post-baseline, if baseline value ≤ 1.5 |
| | | old, Male) | old, Male) | x ULN |
| | | 31 (18 - < 50 years | 101 (18 - < 50 years | |
| | | old, Female) | old, Female) | |
| | | 40 (50 - < 70 years | 119 (50 - < 70 years | |
| | | old, Male) | old, Male) | |
| | | 31 (50 - < 70 years | 101 (50 - < 70 years | |
| | | old, Female) | old, Female) | |

| Test Parameter | Test<br>Parameter<br>Code | Normal Range Lower<br>Limit (LLN) | Normal Range Upper<br>Limit (ULN) | Potentially Clinically Significant Ranges |
|---|---|---|---|---|
| | | 40 (70 - < 80 years | 137 (70 - < 80 years | |
| | | old, Male) | old, Male) | |
| | | 31 (70 - < 80 years | 110 (70 - < 80 years | |
| | | old, Female) | old, Female) | |
| | | 40 (≥ 80 years old, | 145 (≥ 80 years old, | |
| | | Male) | Male) | |
| | | 31 (≥ 80 years old, | 128 (≥ 80 years old, | |
| | | Female) | Female) | |
| Creatine Kinase (U/L) | CK | 39 (Male) | 308 (Male) | > 2.5 x ULN at post-baseline, if baseline value ≤ 2.5 x ULN |
| | | 26 (Female) | 192 (Female) | |
| Direct Bilirubin (umol/L) | BILDIR | <2.00 | 7.00 | > 1.5 x ULN at post-baseline, if baseline value ≤ 1.5 x ULN |
| Gamma Glutamyl | GGT | 10 (< 59 years old, | 61 (< 59 years old, | > 2.5 x ULN at post-baseline, if baseline value ≤ 2.5 |
| Transferase (U/L) | | Male) | Male) | x ULN |
| | | 4 (< 59 years old, | 49 (< 59 years old, | |
| | | Female) | Female) | |
| | | 10 (≥ 59 years old, | 50 (≥ 59 years old, | |
| | | Male) | Male) | |
| | | 5 (≥ 59 years old, | 50 (≥ 59 years old, | |
| | | Female) | Female) | |
| Glucose (mmol/L) | GLUC | 3.90 | 5.60 | < 3 at post-baseline, if baseline value ≥ 3 |
| | | | | > 13.9 at post-baseline, if baseline value ≤ 13.9 |
| Potassium (mmol/L) | K | 3.5 | 5.2 | < 3.5 at post-baseline, if baseline value ≥ 3.5 |
| , | | | | > 5.5 at post-baseline, if baseline value ≤ 5.5 |
| Sodium (mmol/L) | SODIUM | 132 (18 – < 59 years | 147 (18 – < 59 years | < 129 at post-baseline, if baseline value ≥ 129 |
| , | | old) | old) | , |
| | | 135 (≥ 59 years old) | 145 (≥ 59 years old) | > 150 at post-baseline, if baseline value ≤ 150 |
| Triglycerides (mmol/L) | TRIG | 0.42 (< 20 years old, | 1.67 (< 20 years old, | > 3.69 at post-baseline, if baseline value ≤ 3.69 |
| | | Male) | Male) | |
| | | 0.44 (< 20 years old, | 1.40 (< 20 years old, | |
| | | Female) | Female) | |
| | | 0.50 (20 – < 30 years | 2.81 (20 – < 30 years | |
| | | old, Male) | old, Male) | |

SAP Version: Final Version 1.0, 20-May-2022 Controlled Document ID: **3903A.02**, Effective Date 31-Aug-2020 Filing requirements: TMF

| Test Parameter | Test<br>Parameter<br>Code | Normal Range Lower<br>Limit (LLN) | Normal Range Upper<br>Limit (ULN) | Potentially Clinically Significant Ranges |
|---|---|---|---|---|
| | | 0.41 (20 – < 30 years | 1.63 (20 - < 30 years | |
| | | old, Female) | old, Female) | |
| | | 0.56 (30 – < 40 years | 3.62 (30 – < 40 years | |
| | | old, Male) | old, Male) | |
| | | 0.44 (30 – < 40 years | 1.99 (30 – < 40 years | |
| | | old, Female) | old, Female) | |
| | | 0.62 (40 – < 50 years | 3.69 (40 – < 50 years | |
| | | old, Male) | old, Male) | |
| | | 0.51 (40 – < 50 years | 2.42 (40 – < 50 years | |
| | | old, Female) | old, Female) | |
| | | 0.65 (50 – < 60 years | 3.61 (50 – < 60 years | |
| | | old, Male) | old, Male) | |
| | | 0.59 (50 – < 60 years | 2.96 (50 – < 60 years | |
| | | old, Female) | old, Female) | |
| | | 0.65 (≥ 60 years old, | 2.94 (≥ 60 years old, | |
| | | Male) | Male) | |
| | | 0.63 (≥ 60 years old, | 2.71 (≥ 60 years old, | |
| | | Female) | Female) | |
| Urate (mmol/L) | URATE | 125 (< 50 years old, | 488 (< 50 years old, | > 494 at post-baseline, if baseline value ≤ 494 |
| | | Male) | Male) | (Male); |
| | | | | > 446 at post-baseline, if baseline value ≤ 446 (Female) |
| | | 125 (< 50 years old, | 428 (< 50 years old, | |
| | | Female) | Female) | |
| | | 149 (50 - < 70 years | 494 (50 - < 70 years | |
| | | old, Male) | old, Male) | |
| | | 149 (50 - <70 years | 446 (50 - < 70 years | |
| | | old, Female) | old, Female) | |
| | | 149 (≥ 70 years old, | 494 (≥ 70 years old, | |
| | | Male) | Male) | |
| | | 149 (≥ 70 years old, | 446 (≥ 70 years old, | |
| | | Female) | Female) | |
| Urea Nitrogen (mmol/L) | UREAN | 1.40 (< 70 years old) | 8.60 (< 70 years old) | > 8.6 at post-baseline, if baseline value ≤ 8.6 (<70 years old); > 10.4 at post-baseline, if baseline value |

| Test Parameter | Test<br>Parameter<br>Code | Normal Range Lower<br>Limit (LLN) | Normal Range Upper<br>Limit (ULN) | Potentially Clinically Significant Ranges |
|---|---|---|---|---|
| | | | | ≤ 10.4 (70 - <80 years old); > 12.1 at post-baseline, if baseline value ≤ 12.1 (≥ 80 years old) |
| | | 1.40 (70 - < 80 years old) | 10.40 (70 - < 80 years old) | |
| | | 1.40 (≥ 80 years old) | 12.10 (≥ 80 years old) | |

Potentially clinically significant ranges for vital signs parameters are defined in Table 21-3.

Table 21-3: Potentially Clinically Significant Ranges for Vital Signs Parameters

| Test Parameter | Test Parameter Code | Potentially Clinically Significant Ranges |
|---|---|---|
| Pulse rate (beats/min) | PULSE | ≥120 bpm and increase from baseline ≥20 bpm |
| | | ≤50 bpm and decrease from baseline ≥20 bpm |
| Diastolic blood pressure (mmHg) | DIABP | ≥110 mmHg and increase from baseline ≥10 mmHg |
| | | ≤45 mmHg and decrease from baseline ≥10 mmHg |
| Systolic blood pressure (mmHg) | SYSBP | ≥160 mmHg and increase from baseline ≥20 mmHg |
| | | ≤95 mmHg and decrease from baseline ≥20 mmHg |
| Weight | WEIGHT | ≥5% increase from baseline |
| | | ≥5% decrease from baseline |

# Olympia - PIV 2 - SAP body text

Final Audit Report 2022-05-20

Created: 2022-05-20

By: Natalie Steigerwald (natalie.steigerwald@syneoshealth.com)

Status: Signed

Transaction ID: CBJCHBCAABAAhjTv9fEy5U4rzbypaLEKtFj0QsGGulE6

# "Olympia - PIV 2 - SAP body text" History

- Document created by Natalie Steigerwald (natalie.steigerwald@syneoshealth.com) 2022-05-20 11:44:57 AM GMT- IP address: 147.161.171.13
- Document emailed to Birgit Strobl (birgit.strobl@syneoshealth.com) for signature 2022-05-20 11:46:52 AM GMT
- Document emailed to Natalie Steigerwald (natalie.steigerwald@syneoshealth.com) for signature 2022-05-20 11:46:52 AM GMT
- Document emailed to Xiaoyu Lu (xiaoyu.lu@galderma.com) for signature 2022-05-20 11:46:52 AM GMT
- Natalie Steigerwald (natalie.steigerwald@syneoshealth.com) verified identity with Adobe Acrobat Sign authentication

2022-05-20 - 11:47:34 AM GMT

- Document e-signed by Natalie Steigerwald (natalie.steigerwald@syneoshealth.com)
  Signature Date: 2022-05-20 11:47:34 AM GMT Time Source: server- IP address: 147.161.171.13
- Email viewed by Birgit Strobl (birgit.strobl@syneoshealth.com)
  2022-05-20 12:42:26 PM GMT- IP address: 147.161.169.29
- ☑ Birgit Strobl (birgit.strobl@syneoshealth.com) verified identity with Adobe Acrobat Sign authentication
  2022-05-20 12:43:34 PM GMT
- Document e-signed by Birgit Strobl (birgit.strobl@syneoshealth.com)

  Signature Date: 2022-05-20 12:43:34 PM GMT Time Source: server- IP address: 147.161.169.29
- Email viewed by Xiaoyu Lu (xiaoyu.lu@galderma.com) 2022-05-20 8:53:55 PM GMT- IP address: 104.47.6.254
- Xiaoyu Lu (xiaoyu.lu@galderma.com) verified identity with Adobe Acrobat Sign authentication 2022-05-20 - 8:55:08 PM GMT



Adobe
Acrobat Sign

Document e-signed by Xiaoyu Lu (xiaoyu.lu@galderma.com)

Signature Date: 2022-05-20 - 8:55:08 PM GMT - Time Source: server- IP address: 165.225.38.19

Agreement completed.

2022-05-20 - 8:55:08 PM GMT



Powered by Adobe Acrobat Sign